Protocol/Amendment No.: 029-05

THIS PROTOCOL AMENDMENT AND ALL OF THE INFORMATION RELATING TO IT ARE CONFIDENTIAL AND PROPRIETARY PROPERTY OF MERCK SHARP & DOHME CORP., A SUBSIDIARY OF MERCK & CO., INC., WHITEHOUSE STATION, NJ, U.S.A.

#### **SPONSOR:**

Merck Sharp & Dohme Corp., a subsidiary of Merck & Co., Inc. (hereafter referred to as the Sponsor or Merck) One Merck Drive P.O. Box 100 Whitehouse Station, NJ 08889-0100, U.S.A.

Protocol-specific Sponsor Contact information can be found in the Investigator Trial File Binder (or equivalent).

### TITLE:

A Phase 1/2 Clinical Trial to Study the Safety and Tolerability of MK-3475 + Pegylated Interferon alfa-2b (PEG-IFN) and MK-3475 + Ipilimumab (IPI) in Subjects With Advanced Melanoma (MEL) and Renal Cell Carcinoma (RCC) (KEYNOTE 029)

**IND NUMBER:** 110080

**EudraCT NUMBER: 2013-004072-36** 

**Protocol/Amendment No.:** 029-05

# **TABLE OF CONTENTS**

| SUMN | MARY ( | OF CHANGES | 11 |
|---|---|---|---|
| 1.0 | TRIAI | SUMMARY | 14 |
| 2.0 | TRIAI | DESIGN | 16 |
| 2.1 | Tria | l Design | 16 |
| 2.2 | Tria | l Diagram | 21 |
| 3.0 | OBJE | CTIVE(S) & HYPOTHESIS(ES) | 23 |
| 3.1 | Prin | nary Objective(s) & Hypothesis(es) | 23 |
| 3.2 | Seco | ndary Objective(s) & Hypothesis(es) | 24 |
| 3.3 | Exp | oratory Objectives | 24 |
| 4.0 | BACK | GROUND & RATIONALE | 25 |
| 4.1 | Bacl | ground | 25 |
| 4. | .1.1 Pł | armaceutical and Therapeutic Background | 25 |
| | 4.1.1.1 | Pembrolizumab | 25 |
| | 4.1.1.2 | Pegylated Interferon Alfa-2b (PEG-IFN) | 27 |
| | 4.1.1.3 | Ipilimumab (IPI) | 28 |
| 4. | .1.2 Pr | e-clinical Trial with Pembrolizumab | 29 |
| 4. | .1.3 O | ngoing Clinical Trials | 29 |
| 4.2 | Rati | onale | 29 |
| 4. | .2.1 Ra | tionale for the Trial and Selected Subject Population | 29 |
| | 4.2.1.1 | Rationale for Evaluating anti-PD-1 Therapy in Advanced Melanoma and Renal Cell Carcinoma | 31 |
| | 4.2.1 | .1.1 Rationale for Pembrolizumab | 31 |
| | 4.2.1 | .1.2 Rationale for PEG-IFN | 31 |
| | 4.2 | 2.1.1.2.1 Hypothesis for Pembrolizumab + PEG-IFN Combination Therapies | 31 |
| | 4.2.1 | .1.3 Rationale for IPI | 32 |
| | 4 | 2.1.1.3.1 Hypothesis for Pembrolizumab + IPI Combination Therapies | 32 |
| 4. | .2.2 Ra | tionale for Dose Selection/Regimen/Modification | 33 |
| 4. | .2.3 Ra | tionale for Endpoints | 36 |
| | 4.2.3.1 | Safety Endpoints | 36 |
| | 4.2.3.2 | Efficacy Endpoints | 36 |

**Protocol/Amendment No.:** 029-05

| | 4.2. | .3.3 Planned Exploratory Biomarker Research | 38 |
|---|---|---|---|
| | 4.2. | .3.4 Future Biomedical Research | 39 |
| 5.0 | ME | ETHODOLOGY | <b>40</b> |
| 5.1 | E | Entry Criteria | <b>40</b> |
| 5 | 5.1.1 | Diagnosis/Condition for Entry into the Trial | 40 |
| 5 | 5.1.2 | Subject Inclusion Criteria. | 40 |
| 5 | 5.1.3 | Subject Exclusion Criteria | 43 |
| 5.2 | T | Trial Treatment(s) | 45 |
| 5 | 5.2.1 | Dose Selection/Modification | 45 |
| | 5.2. | .1.1 Dose Selection (Preparation) | 45 |
| | 5.2. | .1.2 Rules for Dose Finding (Part 1A) | 46 |
| | 5 | 5.2.1.2.1 Definition of Dose-Limiting Toxicities | 48 |
| | 5 | 5.2.1.2.2 Replacement of Subjects in DLT Period (Part 1A) | 49 |
| | 5.2. | .1.3 Dose Modification (Escalation/Titration/Other) | 50 |
| | 5 | 5.2.1.3.1 Dose Modification Guidelines for pembrolizumab + PEG-IFN or pembrolizumab + IPI Combination Therapy | 52 |
| | | 5.2.1.3.1.1 Dose Modification Guidelines for Treatment Group A (Part 1A Only): pembrolizumab + PEG-IFN | 52 |
| | | 5.2.1.3.1.2 Dose Modification Guidelines for PEG-IFN | 54 |
| | | 5.2.1.3.1.2.1 Dose Modification for Management of Depression | 54 |
| | | 5.2.1.3.1.2.2 Interruption or Discontinuation of PEG-IFN | 55 |
| | 5 | 5.2.1.3.2 Dose Modification Guidelines for Treatment Group B: pembrolizumab + IPI | 56 |
| | | 5.2.1.3.2.1 Dose Modification Guidelines for IPI | 58 |
| | | 5.2.1.3.2.1.1 Interruption or Discontinuation of IPI | 58 |
| | 5 | 5.2.1.3.3 Dose Modification and Supportive Care Guidelines for DRAEs for Pembrolizumab Monotherapy and Part 1C | 58 |
| 5 | 5.2.2 | Timing of Dose Administration | 64 |
| 5 | 5.2.3 | Treatment after Initial Evidence of Radiologic Disease Progression | 65 |
| 5 | 5.2.4 | Trial Blinding/Masking | 66 |
| 5.3 | F | Randomization or Treatment Allocation | 66 |
| 5.4 | S | Stratification | <b>67</b> |
| 5.5 | ( | Concomitant Medications/Vaccinations (Allowed & Prohibited) | <b>67</b> |
| 5 | 5.5.1 | Acceptable Concomitant Medications | 67 |

| | 5.5.2 | 2 Prohib | oited Concomitant Medications | 67 |
|---|---|---|---|---|
| 5. | .6 | Rescue 1 | Medications & Supportive Care | 68 |
| | 5.6.1 | Suppo | rtive Care Guidelines | 68 |
| | 5.6.2 | 2 Guide | lines for Pembrolizumab/PEG-IFN Combination Therapy | 69 |
| | 5. | 6.2.1 P | EG-IFN Dosing Considerations | 69 |
| 5. | .7 | Diet/Act | tivity/Other Considerations | 69 |
| | 5.7.1 | Diet | | 69 |
| | 5.7.2 | 2 Contra | aception | 69 |
| | 5.7.3 | Use in | Pregnancy | 71 |
| | 5.7.4 | Use in | Nursing Women | 71 |
| 5. | .8 | Subject | Withdrawal/Discontinuation Criteria | <b>71</b> |
| | 5.8.1 | Disco | ntinuation of Study Treatment after CR | 72 |
| 5. | .9 | Subject | Replacement Strategy | 72 |
| 5. | .10 | Beginni | ng and End of the Trial | 73 |
| 5. | .11 | Clinical | Criteria for Early Trial Termination | 73 |
| 6.0 | T] | RIAL FI | LOW CHART | <b>74</b> |
| 6 | .1 | Treatmo | ent Phase | <b>74</b> |
| | 6.1.1 | Treatn | nent Phase: Part 1A (MEL and RCC) and Part 1B and 1C (MEL only) . | 74 |
| | 6. | | reatment Group A: pembrolizumab + PEG-IFN Combination Therapy<br>Part 1A only) | |
| | 6. | | eatment Group B: pembrolizumab + IPI Combination Therapy (Part A, Part 1B and Part 1C) | |
| 6. | .2 | Second | Course Phase: All Parts - All Treatment Groups (MEL and RCC). | 85 |
| 7.0 | T | RIAL PF | ROCEDURES | 89 |
| 7. | .1 | Trial Pr | ocedures | 89 |
| | 7.1.1 | Admii | nistrative Procedures | 89 |
| | 7. | 1.1.1 In | formed Consent | 89 |
| | | 7.1.1.1.1 | General Informed Consent | 89 |
| | | 7.1.1.2 | Consent and Collection of Specimens for Future Biomedical Research | 90 |
| | 7. | 1.1.2 In | clusion/Exclusion Criteria | 90 |
| | 7. | 1.1.3 St | ubject Identification Card | 90 |
| | 7. | 1.1.4 M | ledical History | 90 |

| 7.1.1.5 Prior and Concomitant Medications Review | 90 |
|---|---|
| 7.1.1.5.1 Prior Medications | 90 |
| 7.1.1.5.2 Concomitant Medications | 90 |
| 7.1.1.5.3 Disease Details | 91 |
| 7.1.1.5.4 Prior Treatment Details | 91 |
| 7.1.1.5.5 Subsequent Anti-Cancer Therapy Status | 91 |
| 7.1.1.6 Assignment of Screening Number | 91 |
| 7.1.1.7 Assignment of Randomization Number | 91 |
| 7.1.1.8 Trial Compliance (Medication/Diet/Activity/Other) | 91 |
| 7.1.2 Clinical Procedures/Assessments | 92 |
| 7.1.2.1 Adverse Event (AE) Monitoring | 92 |
| 7.1.2.2 Physical Exam | 92 |
| 7.1.2.2.1 Full Physical Exam | 92 |
| 7.1.2.2.2 Directed Physical Exam | 92 |
| 7.1.2.3 Vital Signs | 93 |
| 7.1.2.4 Electrocardiogram (ECG) | 93 |
| 7.1.2.5 Eastern Cooperative Oncology Group (ECOG) Performance Scale | 93 |
| 7.1.2.6 Tumor Tissue Collection | 93 |
| 7.1.2.7 Tumor Imaging and Assessment of Disease | 94 |
| 7.1.2.8 Assessment of Disease | 94 |
| 7.1.2.9 Ophthalmologic Examination | 95 |
| 7.1.3 Laboratory Procedures/Assessments | 95 |
| 7.1.3.1 Laboratory Safety Evaluations (Hematology, Chemistry and Urinalysis) | 95 |
| 7.1.3.1.1 Serum/Urine β-hCG | 97 |
| 7.1.3.2 Pharmacokinetic/Pharmacodynamic Evaluations | 97 |
| 7.1.3.2.1 Blood Collection for Serum MK-3475 | . 100 |
| 7.1.3.2.2 Blood Collection for Anti-MK-3475 Antibodies (ADA) | . 100 |
| 7.1.3.2.3 Blood Collection for total IgG | . 100 |
| 7.1.3.3 Future Biomedical Research | . 100 |
| 7.1.4 Other Procedures | . 100 |
| 7.1.4.1 Withdrawal/Discontinuation | . 100 |
| 7.1.4.1.1 Withdrawal From Future Biomedical Research | . 101 |
| 7.1.4.2 Blinding/Unblinding | . 101 |

| Prod | luct: | MK-34 | 75 |
|------|-------|-------|----|

| 7.1.4.3 | Calibration of Critical Equipment | 101 |
|---|---|---|
| 7.1.5 Vis | it Requirements | 102 |
| 7.1.5.1 | Screening | 102 |
| 7.1.5.2 | Treatment Period | 102 |
| 7.1.5.2 | 2.1 Second Course Phase | 103 |
| 7.1.5.3 | Post-Treatment Visits | 104 |
| 7.1.5. | 3.1 Safety Follow-up Visit | 104 |
| 7.1.5. | 3.2 Follow-up Visits | 105 |
| 7.1.5. | 3.3 Survival Follow-up (SFU) | 105 |
| 7.1.5.4 | Survival Status | 105 |
| 7.2 Asses | sing and Recording Adverse Events | 106 |
| | inition of an Overdose for This Protocol and Reporting of Overdose Sponsor | |
| | porting of Pregnancy and Lactation to the Sponsor | |
| | nediate Reporting of Adverse Events to the Sponsor | |
| 7.2.3.1 | Serious Adverse Events | |
| 7.2.3.2 | Events of Clinical Interest | 109 |
| 7.2.3.3 | Protocol-Specific Exceptions to Serious Adverse Event Reporting | 110 |
| 7.2.4 Eva | luating Adverse Events | 110 |
| 7.2.5 Spc | nsor Responsibility for Reporting Adverse Events | 113 |
| 8.0 STATIS | TICAL ANALYSIS PLAN | 113 |
| 8.1 Statis | tical Analysis Plan Summary | 113 |
| 8.1.1 Par | : 1 | 113 |
| 8.2 Statis | tical Analysis Plan | 114 |
| 8.2.1 Res | ponsibility for Analyses/In-House Blinding | 114 |
| 8.2.2 Hyp | ootheses/Estimation | 114 |
| 8.2.3 Ana | alysis Endpoints | 114 |
| 8.2.3.1 | Safety Endpoints | 114 |
| 8.2.3.2 | Efficacy Endpoints | 115 |
| 8.2.4 Ana | alysis Populations | 115 |
| 8.2.4.1 | Efficacy Analysis Populations | 115 |
| 8.2.4.2 | Safety Analysis Populations | 115 |
| 8.2.5 Stat | istical Methods | 116 |

| 8 | 3.2.5.1 Sta | atistical Methods for Efficacy Analyses | 116 |
|---|---|---|---|
| | 8.2.5.1.1 | Progression-free Survival (PFS) | . 116 |
| | 8.2.5.1.2 | Overall Survival (OS) | 116 |
| | 8.2.5.1.3 | Objective Response Rate (ORR) | . 116 |
| | 8.2.5.1.4 | Ordinal Response Score | 116 |
| | 8.2.5.1.5 | Duration of Response (DOR) | . 116 |
| | 8.2.5.1.6 | Pharmacokinetic Parameters | . 116 |
| 8 | 3.2.5.2 Sta | ntistical Methods for Safety Analyses | 117 |
| 8 | | mmaries of Baseline Characteristics, Demographics, and Other | |
| 8.2 | .6 Multipl | licity | 119 |
| 8.2 | .7 Sample | Size and Power Calculations | 119 |
| 8 | 3.2.7.1 Par | rt 1 | 119 |
| 8.2 | .8 Interim | Analyses | 120 |
| 8.2 | .9 Compli | iance (Medication Adherence) | . 120 |
| 8.2 | .10 Extent | of Exposure | . 121 |
| | | G, PACKAGING, STORAGE AND RETURN OF CLINICAL | |
| 9.1 | | tional Product | |
| 9.1 | | g and Labeling Information | |
| 9.3 | | Supplies Disclosure | |
| 9.4 | | and Handling Requirements | |
| 9.5 | | and Reconciliation | |
| 9.6 | | l Policies | |
| | | TRATIVE AND REGULATORY DETAILS | |
| 10.1 | | tiality | |
| | | entiality of Data | |
| | | entiality of Subject Records | |
| | | entiality of Investigator Information | |
| | | entiality of IRB/IEC Information | |
| 10.2 | | nce with Financial Disclosure Requirements | |
| 10.3 | _ | nce with Law, Audit and Debarment | |
| 10.4 | _ | nce with Trial Registration and Results Posting Requirements | |

| 10.5 | Quality Management System | 127 |
|---|---|---|
| 10.6 | Data Management | 127 |
| 10.7 | Publications | 127 |
| 11.0 l | LIST OF REFERENCES1 | 128 |
| <b>12.0</b> A | APPENDICES1 | 137 |
| 12.1 | Merck Code of Conduct for Clinical Trials | 137 |
| 12.2 | Collection and Management of Specimens for Future Biomedical Research | 139 |
| 12.3 | Understanding the Intent, Scope and Public Health Benefits of Exploratory Biomarker Research: A Guide for IRBs/IECs and Investigational Site Staff | 145 |
| 12.4 | ECOG Performance Status | 156 |
| 12.5 | Common Terminology Criteria for Adverse Events V4.0 (CTCAE)1 | 157 |
| 12.6 | Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | 158 |
| 12.7 | List of Abbreviations | 159 |
| 13.0 | SIGNATURES1 | 163 |
| 13.1 | Sponsor's Representative | 163 |
| 13.2 | Investigator | 163 |

**Protocol/Amendment No.:** 029-05

# LIST OF TABLES

| Table 1 | Dose Finding Scheme for Treatment Group A: pembrolizumab + PEG- | |
|---|---|---|
| | IFN (Part 1A only) | 17 |
| Table 2 | Dose for Treatment Group B: pembrolizumab + IPI (Part 1A and 1B) | 17 |
| Table 3 | Adequate Organ Function Laboratory Values | 42 |
| Table 4 | Trial Treatments | 45 |
| Table 5 | Dose Finding Rules | 47 |
| Table 6 | Dose Modification Guidelines for DRAEs for pembrolizumab + PEG-IFN | 52 |
| Table 7 | Recommended Dose Reduction for PEG-IFN | 54 |
| Table 8 | Dose Modification Guidelines for DRAEs for pembrolizumab + IPI (Part 1A and 1B) | 56 |
| Table 9 | Dose Modification and Toxicity Management Guidelines for Immune-<br>Related AEs for Pembrolizumab Monotherapy and Part 1C | 59 |
| Table 10 | Pembrolizumab Infusion Reaction Dose Modification and Treatment Guidelines | |
| Table 11 | Imaging and Treatment after 1st Radiologic Evidence of PD | 66 |
| Table 12 | Laboratory Tests | 96 |
| Table 13 | Pharmacokinetic, Total IgG, and ADA Assessments | 97 |
| Table 14 | Timing of PK and ADA Assessments, Parts 1A and 1B | 98 |
| Table 15 | Timing of PK and ADA Assessments, Part 1C | 99 |
| Table 16 | Evaluating Adverse Events | 111 |
| Table 17 | Summary of Analysis Strategy for Key Efficacy Endpoints | 117 |
| Table 18 | Analysis Strategy for Safety Parameters | 118 |
| Table 19 | Product Descriptions | 121 |

**Protocol/Amendment No.:** 029-05

# LIST OF FIGURES

| Figure 2 Pembrolizumab + IPI dose finding: Part 1A Safety run-in and Part 1B | |
|---|---|
| rigule 2 Femololizumao + IFI dose midnig. Fait IA Safety fun-in and Fait ID | |
| Expansion cohort in MEL subjects. | . 22 |
| Figure 3 Part 1C – Phase I/II portion of the trial | . 23 |
| Figure 4 Effect of IFNα and Anti-PD-1 in MC38 models | . 32 |

**Protocol/Amendment No.:** 029-05

## **SUMMARY OF CHANGES**

## PRIMARY REASON(S) FOR THIS AMENDMENT:

| Section Number (s) | Section Title(s) | Description of Change (s) | Rationale |
|---|---|---|---|
| 5.2.1.3.3 | Dose Modification and<br>Supportive Care<br>Guidelines for DRAEs for<br>Pembrolizumab<br>Monotherapy and Part 1C | Insertion of subheading "Dose modification and toxicity management for immune-related AEs associated with pembrolizumab" and associated program language. Revised dose modification table to include myocarditis-specific guidelines and actions in the event of myocarditis; revised action for all other immune-related Grade 3 AEs; and other clarifications. | Consistency and alignment with program-wide safety update to dose modification guidance |
| 6.0 | Trial Flow Chart | To all flow charts: amended survival status rows to allow assessment throughout the trial. Clarification of existing footnotes for survival status follow-up. | Clarification and alignment with program standards |
| 7.1.5.3.2 | Follow-up Visits | Addition of text: The Sponsor may request survival status to be assessed at additional time points during the course of the study (not to exceed approximately 12 weeks). | |
| 7.1.5.3.3 | Survival Follow-up (SFU) | Clarification that subjects should be contacted <i>approximately</i> every 12 weeks. Deletion of redundant text. | |
| 7.1.5.4 | New Section: Survival<br>Status | Addition of text to enable survival follow-up activities throughout the study. | |

**Protocol/Amendment No.:** 029-05

# ADDITIONAL CHANGE(S) FOR THIS AMENDMENT:

| Section Number (s) | Section Title (s) | Description of Change (s) | Rationale |
|---|---|---|---|
| 4.1 | Background | Insertion of latest program-aligned background information for pembrolizumab. | Alignment with program language |
| 4.1.1 | Pharmaceutical and<br>Therapeutic Background | Deletion of redundant text now inserted in Section 4.1. | Deletion of repetition |
| 4.2.3.2 | Efficacy Endpoints | Clarification of clinical stability to include: • Absence of signs and symptoms (including worsening of laboratory values) indicating clinically significant disease progression. | Improved clarity and consistency with program language |
| 5.2.3 | Treatment after Initial Evidence of Radiologic Disease Progression | For the definition of clinical stability – insertion of text "clinically significant" to the bullet: • Absence of signs and symptoms (including worsening of laboratory values) indicating clinically significant disease progression | Improved clarity and consistency with program language |
| | | Clarification of clinical stability to includeclinically significant disease progression | Clarification |
| | | Table 11 – insertion of abbreviations to footnote. | |
| 5.8 | Subject<br>Withdrawal/Discontinuation<br>Criteria | Cross-reference to Section 7.1.5 amended to Section 5.2.3 | Correction |

| Section Number (s) | Section Title (s) | Description of Change (s) | Rationale |
|---|---|---|---|
| 6.0 | Trial Flow Chart | "also" replaced with "not" in Section 6.1.1.1 footnote #21, Section 6.1.1.2 footnote #22, and Section 6.2 footnote #19: | Correction |
| | | "Copies of digital photographs should also not be submitted to the central imaging vendor unless otherwise noted by the Sponsor" | |
| 7.1.2.8 | Assessment of Disease | Insertion of program language. | Consistency with program |
| | | Amended the definition of clinical stability: | language |
| | | Absence of signs and symptoms indicating | Alignment with Section 5.2.3 |
| | | clinically significant disease progression, | and programe language |
| | | including worsening of laboratory values | |
| 7.1.3.1 | Laboratory Safety | To Table 12: | Clarification/correction |
| | Evaluations (Hematology, Chemistry and Urinalysis) | • Footnote c deleted and moved into a table note. | |
| | | Additional information added to footnote | |
| | | e regarding hepatitis B/C testing. | |
| | | Addition of footnote e to LDH. Addition of footnote e to LDH. | |
| 7 2 2 1 | C | Deletion of Anti-HDV. Construction of Anti-HDV. Construction of Anti-HDV. Construction of Anti-HDV. | Commention |
| 7.2.3.1 | Serious Adverse Events | Cross-reference to Table 14 amended to Table 16 | Correction |
| | | 18010 10 | |
| Throughout | | Minor typographical corrections. | Improved |
| | | | consistency/readability |

**Protocol/Amendment No.:** 029-05

# 1.0 TRIAL SUMMARY

| Abbreviated Title | Dhase 1/2 Study of Downhastinowsky (MV 2475) DEC IEN 6 |
|---|---|
| Troote valed True | Phase 1/2 Study of Pembrolizumab (MK-3475) + PEG-IFN & Pembrolizumab + IPI in Subjects with Advanced MEL & RCC (KEYNOTE 029) |
| Trial Phase | Phase 1/2 |
| Clinical Indication | Advanced or Metastatic Melanoma and Renal Cell Carcinoma |
| Trial Type | Interventional |
| Type of control | No treatment control |
| Route of administration | Intravenous (pembrolizumab and IPI) and subcutaneous (PEG-IFN) |
| Trial Blinding | Unblinded Open-label |
| Treatment Groups | Part 1A: Treatment Group A: Pembrolizumab 2 mg/kg (or 200 mg)* IV every 3 weeks (q3w) + PEG-IFN 0.5µg/kg weekly Pembrolizumab 2 mg/kg (or 200 mg)* IV q3w + PEG-IFN 1µg/kg weekly Pembrolizumab 2 mg/kg weekly Pembrolizumab 2 mg/kg weekly Pembrolizumab 2 mg/kg weekl |
| | PEG-IFN 2μg/kg weekly; Pembrolizumab 2 mg/kg (or 200 mg)* IV q3w + PEG-IFN 3μg/kg weekly |
| | Treatment Group B: Pembrolizumab 2 mg/kg (or 200 mg)* IV q3w + IPI 1 mg/kg q3w |
| | Part 1B: |
| | Treatment Group B: |
| | Pembrolizumab 2 mg/kg (or 200 mg)* IV q3w + IPI 1mg/kg q3w |
| | *With the approval of Amendment 03, subjects continuing pembrolizumab treatment in Parts 1A and 1B will switch to a fixed dose of 200 mg q3w (not weight-based). |
| | Prior to the approval of Amendment 03, the Sponsor notified sites and IRBs that Part 2 would not be initiated. Part 2 is deleted in Amendment 03. |
| | Part 1C:<br>Treatment Group B: |
| | Arm 1:<br>Pembrolizumab 200 mg q3w + IPI 50 mg every 6 weeks (q6w) |
| | Arm 2:<br>Pembrolizumab 200 mg q3w + IPI 100 mg every 12 weeks (q12w) |
| Number of trial subjects | Approximately 233 up to a maximum of approximately 293 (up to 43 in Part 1A, 90 to 150 in Part 1B and up to 100 in Part 1C) subjects will be enrolled. |
| Estimated duration of trial | The sponsor estimates that the trial will require approximately 32 months for Parts 1A and 1B, from the time the first subject signs the informed consent until the last subject's last visit. For Part 1C, the Sponsor also estimates that the trial will require approximately 32 months from the time the first subject signs the informed consent until the last subject's last visit. |

**Protocol/Amendment No.:** 029-05

#### **Duration of Participation**

Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final contact.

After a screening phase of up to 28 days, eligible subjects will receive assigned treatment on Day 1 of each dosing cycle and thereafter following a weekly (PEG-IFN) or q3w (IPI) schedule in Part 1A and 1B, and q6w or q12w schedule (IPI) in Part 1C. Pembrolizumab will be given q3w. A cycle is 6 weeks.

In Part 1A, RCC and MEL subjects will be randomly assigned to receive pembrolizumab + PEG-IFN or pembrolizumab + IPI.

Treatment with pembrolizumab + PEG-IFN doublet (Treatment Group A) will continue until up to two years of therapy have been administered. documented disease progression, unacceptable adverse events (AEs), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.

Treatment with pembrolizumab + IPI doublet (Treatment Group B) will continue for 2 cycles (12 weeks), followed by treatment with pembrolizumab single agent until up to 24 months of therapy have been administered, documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.

In Part 1B, MEL subjects will receive pembrolizumab + IPI (Treatment Group B). Treatment duration will follow the same schema as described in Part 1A. Subjects in Part 1B who attain an investigator-determined complete response (CR) may consider stopping trial treatment with pembrolizumab, after all 4 doses of IPI and at least 24 weeks of pembrolizumab have been administered. In addition, if a confirmed CR per modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 is attained, at least 2 additional doses of pembrolizumab must be received after CR is first documented.

In Part 1C, MEL subjects will be randomly assigned to pembrolizumab + 2 dose regimens of IPI (Treatment Group B). Treatment with pembrolizumab + IPI will continue for a maximum of 4 cycles (24 weeks) in Arm 1 or 8 cycles (48 weeks) in Arm 2, followed by treatment with pembrolizumab single agent until up to 24 months of pembrolizumab have been administered, documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons. Subjects in Part 1C who attain an investigator-determined CR may consider stopping trial treatment with pembrolizumab, after at least 24 weeks of pembrolizumab have been administered. In addition, if a confirmed CR per modified RECIST 1.1 is attained, at least 2 additional doses of pembrolizumab must be received after CR is first documented. In addition, and only in Part 1C, upon Sponsor consultation, subjects who attain an investigator-determined CR or a very good partial response [VGPR: partial response per RECIST 1.1 with Percent Change from Baseline (maximum reduction in tumor line length) >60%] may consider stopping treatment with IPI, after a minimum of one dose of IPI on either treatment arm.

Protocol/Amendment No.: 029-05

| | In Part 1A, 1B and 1C, upon Sponsor consultation, subjects who stop pembrolizumab with SD or better per modified RECIST 1.1 may be eligible for retreatment with pembrolizumab + IPI or pembrolizumab monotherapy if they progress after stopping pembrolizumab at the discretion of the Investigator if they meet the criteria for retreatment, as long as the Part to which the subject was initially enrolled remains open; this will be designated the Second Course Phase. Subjects in Part 1A who received PEG-IFN will not be allowed to restart Second Course Phase with pembrolizumab + PEG-IFN; these subjects can only receive pembrolizumab monotherapy in Second Course. The Second Course Phase will be administered for a maximum of 17 doses of pembrolizumab and 4 doses of IPI. After the end of treatment, each subject will be followed for a minimum of 30 days for AE monitoring [serious adverse events (SAEs) will be collected for up to 90 days after the end of treatment]. Subjects will go into survival follow-up (SFU) for disease status, including initiating a non-study cancer treatment and experiencing disease progression, until death, withdrawal of consent, or lost to follow-up. |
|---|---|
| Randomization Ratio | Part 1A (MEL and RCC): 1:1. Part 1B (MEL): Single Arm Expansion. Part 1C (MEL): 1:1 |

A list of abbreviations used in this document can be found in Section 12.7.

#### 2.0 TRIAL DESIGN

#### 2.1 **Trial Design**

This is a multi-center, open-label, 3-part Phase 1/2 trial of intravenous (IV) pembrolizumab in combination with subcutaneous (SC) Pegylated Interferon Alfa-2b (PEG-IFN) or IV ipilimumab (IPI) in subjects with advanced or metastatic melanoma (MEL) or renal cell carcinoma (RCC).

The trial consists of three parts:

Part 1A is the phase I portion of the trial to define the preliminary maximum-tolerated dose (MTD) or maximum administered dose (MAD) for the combination doublets listed below and confirm the tolerability of the dose combination.

Treatment Group A: pembrolizumab + PEG-IFN

Treatment Group B: pembrolizumab + IPI

Subjects will be treated with doublets administered as detailed in Table 1 and Table 2.

If dose levels are open in Part 1A in both PEG-IFN and IPI dose finding Arms, subjects will be randomly assigned between the two combinations. Intermediate dose levels may be pursued, depending on emerging data from the current and other pembrolizumab studies.

Protocol/Amendment No.: 029-05

Table 1 Dose Finding Scheme for Treatment Group A: pembrolizumab + PEG-IFN (Part 1A only)

| Dose Level | Pembrolizumab Dose | PEG-IFN Dose (μg/kg) |
|------------|---------------------------|----------------------|
| (DL) | (mg/kg) IV | SC Weekly |
| -1 | 2 mg/kg (or 200 mg)** q3w | 0.5 |
| 1* | 2 mg/kg (or 200 mg)** q3w | 1 |
| 2 | 2 mg/kg (or 200 mg)** q3w | 2 |
| 3 | 2 mg/kg (or 200 mg)** q3w | 3 |

<sup>\*</sup>Starting Dose

Table 2 Dose for Treatment Group B: pembrolizumab + IPI (Part 1A and 1B)

| Dose Level<br>(DL) | Pembrolizumab Dose<br>(mg/kg) IV | IPI Dose<br>(mg/kg) q3w x<br>4 doses |
|---|---|---|
| 1 | 2 mg/kg (or 200 mg)*<br>q3w | 1 |

<sup>\*</sup>With the approval of Amendment 03, subjects continuing pembrolizumab treatment will switch to a fixed dose of 200 mg (not weight-based).

Dose-limiting toxicities (DLTs) observed in Cycle 1 will be used to determine tolerability of the doublet and possible escalation to the next dose level (when applicable). A cycle is 6 weeks. The guidelines used for dose escalation and dose confirmation are shown in Table 5.

The rules applied for the dose finding algorithm are as follows:

In the pembrolizumab + PEG-IFN combination, an initial cohort of 3 subjects is enrolled. Subsequent dosing decisions within a dose combination will be based on the rules in Table 5. The dose confirmation part will continue until <4 of 14 subjects experience a DLT. subjects become evaluable for DLT assessment, the number of subjects who are evaluable for DLT versus the number of subjects who developed a DLT will be continuously assessed and de-escalation and re-escalation to eligible doses will occur as shown in Table 5. In the pembrolizumab + IPI combination, an open-label run-in period (Part 1A), will be used to assess the safety and tolerability of the doublet therapy during the first cycle of treatment. A total of up to 18 subjects will be enrolled at dose level 1 (DL1) of pembrolizumab administered at a dose of 2 mg/kg q3w in combination with IPI administered at dose of 1 mg/kg q3w (for a total of 4 doses).

If  $\leq 6$  DLTs are observed in the 18 subjects enrolled, this dose level will be considered tolerable, and Part 1B will be initiated. Should this dose level (DL1) not be proven tolerable (>6 DLTs), the combination with IPI will not be further developed.

Part 1B is a single arm expansion cohort, designed to better characterize the safety and tolerability, as well as to evaluate preliminary efficacy of the combination pembrolizumab + IPI in MEL subjects. Pembrolizumab will be administered at a dose of 2 mg/kg q3w (or

<sup>\*\*</sup>With the approval of Amendment 03, subjects continuing pembrolizumab treatment will switch to a fixed dose of 200 mg (not weight-based).

**Protocol/Amendment No.:** 029-05

200mg q3w) in combination with IPI administered at a dose of 1 mg/kg (for 4 doses). At least 90 and up to an additional 150 subjects with advanced or metastatic MEL will be enrolled in the expansion cohort at this dose level.

With the approval of Amendment 03, subjects continuing pembrolizumab treatment on Parts 1A and 1B will switch to a fixed dose of 200 mg q3w (not weight-based). The rationale for fixed dose regimen is outlined in Section 4.2.2.

Prior to the approval of Amendment 03, the Sponsor notified sites and IRBs that Part 2 would not be initiated. Part 2 is removed from the protocol in Amendment 03.

Part 1C is the phase I/II randomized portion of the trial and is to further evaluate safety and tolerability of pembrolizumab + IPI in advanced MEL subjects, as well as preliminary clinical efficacy of the combination. Part 1C will evaluate the below listed treatments.

Treatment Group B: pembrolizumab + IPI

Arm 1: pembrolizumab 200 mg q3w for a maximum of 24 months + IPI 50 mg q6w for a maximum of 4 doses.

Arm 2: pembrolizumab 200 mg q3w for a maximum of 24 months + IPI 100 mg q12w for a maximum of 4 doses. Part 1C subjects will be randomized to the treatment groups in a 1:1 ratio. There will be no stratification prior to the randomization of subjects.

Approximately 233 to a maximum of approximately 293 subjects (up to 43 in Part 1A, at least 90 and up to 150 in Part 1B, and up to approximately 100 in Part 1C) will be enrolled in this trial to examine the safety and efficacy of the combinations pembrolizumab + PEG-IFN and pembrolizumab + IPI. The Part 1B sample size is driven by the expected number of PD-L1 negative subjects. Assuming that the prevalence of PD-L1 negative subjects is ~25%, then 90 subjects would be expected to provide ~22 subjects with PD-L1 negative MEL. If less than 22 PD-L1 negative MEL were enrolled in the pembrolizumab + IPI Arm in Part 1A and 1B combined, enrollment will continue until at least 22 PD-L1 negative subjects are enrolled, up to a maximum of 150 subjects in Part 1B.

#### Parts 1A and 1B:

Subjects will undergo first imaging evaluation at week 12 (± 3 days). Subsequently, subjects will be evaluated every 6 weeks (42 days  $\pm$  3 days), independently of any treatment delays, with radiographic imaging to assess response to treatment, until week 30. Subjects will then undergo imaging evaluation every 12 weeks ( $84 \pm 7$  days). RECIST 1.1 will be used as the primary response rate efficacy endpoint. RECIST 1.1 will be adapted as described in Section 4.2.3.2 to adjust for the tumor response patterns seen with pembrolizumab treatment (e.g., tumor flare), and this adapted/modified RECIST 1.1 will be used by the sites for treatment decisions. The primary response rate efficacy endpoint will be based on independent central review using RECIST 1.1 [1]. Modified RECIST 1.1 will also be used by the local site to determine eligibility and make treatment decisions.

**Protocol/Amendment No.:** 029-05

AEs will be monitored throughout the trial and graded in severity according to the guidelines outlined in the National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) Version 4.0.

Treatment will continue as outlined in Table 1 and Table 2 until documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, completion of 24 months of treatment with pembrolizumab, or administrative reasons.

Subjects in the pembrolizumab + IPI Arm who initially attain clinical benefit (defined as modified RECIST 1.1 confirmed PR or SD  $\geq$ 6 months), and experience disease progression while receiving single agent pembrolizumab will be eligible for reinduction with a maximum of 4 doses of IPI q3w as long as Part 1A or 1B remains open.

Subjects who attain an investigator-determined confirmed CR may consider stopping trial treatment after receiving at least 6 weeks of PEG-IFN treatment/all 4 doses of IPI and at least 24 weeks of pembrolizumab. In addition, if a confirmed CR per modified RECIST 1.1 is attained, at least 2 additional treatments of pembrolizumab must be received prior to treatment discontinuation. Upon consultation with the Sponsor, subjects who stop pembrolizumab with SD or better per modified RECIST 1.1 may be eligible for retreatment with a maximum of 17 doses of pembrolizumab and 4 doses of IPI if they progress after stopping pembrolizumab at the discretion of the investigator according to the criteria in Section 7.1.5.2.1, as long as the trial part to which the subject was initially enrolled remains open; this retreatment will be the Second Course Phase. Subjects enrolled in Part 1A who received PEG-IFN who are eligible for Second Course Phase will only be allowed to receive pembrolizumab monotherapy in Second Course. Response or progression in the Second Course Phase will not count towards the overall response rate (ORR) and progression-free survival (PFS) of the primary endpoint in this trial. The decision to retreat will be at the discretion of the investigator only if no cancer treatment was administered since the last dose of pembrolizumab, the subject still meets the safety parameters listed in the Inclusion/Exclusion criteria and the trial remains open (refer to Section 7.1.5.2.1 for further details).

After the end of treatment, each subject will be followed for 30 days for AE monitoring (SAEs will be collected for 90 days after the end of treatment). Subjects who discontinue treatment for reasons other than disease progression will have SFU for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone contact for overall survival (OS) until death, withdrawal of consent or the end of the trial, whichever comes first.

All subjects will be required to submit a tumor tissue sample for biomarker analyses and PD-L1 expression evaluation. In Part 1B, PD-L1 status must be assessed during screening, and if the tumor biopsy submitted is inadequate for determination of PD-L1 status by immunohistochemistry (IHC) at a central pathology laboratory, the subject will not be randomized. Subjects with an inadequate archival sample may obtain a new biopsy and

**Protocol/Amendment No.:** 029-05

subjects with an inadequate newly obtained biopsy may undergo re-biopsy at the discretion of the investigator.

The primary safety objectives of the trial (Part 1A and Part 1B) are to determine the safety and tolerability of pembrolizumab in combination with PEG-IFN or IPI in subjects with advanced MEL and RCC. The primary efficacy objective of Part 1B of the trial is to evaluate the anti-tumor activity in PD-L1 negative MEL subjects treated with pembrolizumab in combination with IPI at DL1.

Part 1C: Part 1C of the trial will enroll approximately 100 subjects with advanced MEL.

The primary objectives for Part 1C are rate of drug-related adverse events (DRAEs) and ORR. Secondary objectives include PFS, OS and duration of response (DOR). The pharmacokinetic (PK) properties for pembrolizumab + IPI in each doublet setting will be investigated as an exploratory objective.

In Part 1C, subjects will undergo imaging evaluation every 6 weeks ( $\pm$  3 days), independent of any treatment delays, with radiographic imaging to assess response to treatment, until week 24. Subjects will then undergo imaging evaluation every 12 weeks ( $84 \pm 7$  days). RECIST 1.1 will be used as the primary response rate efficacy endpoint and adapted/modified RECIST 1.1 will be used by the investigative sites for treatment decisions. The primary response rate efficacy endpoint will be based on independent central review using RECIST 1.1 [1]. Modified RECIST 1.1 will also be used by the treating investigator local site to determine eligibility.

AEs will be monitored throughout the trial and in severity according to the guidelines outlined in the NCI CTCAE Version 4.0.

Treatment with pembrolizumab + IPI doublets (Treatment Group B) will continue for a maximum of 4 cycles (24 weeks) in Arm 1 and 8 cycles (48 weeks) in Arm 2, followed by treatment with pembrolizumab single agent for up to 24 months of therapy, documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.

Subjects in Part 1C who attain an investigator-determined confirmed CR may consider stopping trial treatment with pembrolizumab after receiving at least 24 weeks of pembrolizumab. In addition, if a confirmed CR per modified RECIST 1.1 is attained, at least two additional doses of pembrolizumab must be received prior to treatment discontinuation. Upon Sponsor consultation, subjects who attain an investigator-determined confirmed CR or a VGPR [partial response per RECIST 1.1 with Percent Change from Baseline (maximum reduction in tumor line length) >60%] may consider stopping treatment with IPI after a minimum of one dose of IPI on either Arm of treatment.

Upon Sponsor consultation, subjects who stop pembrolizumab with SD or better per modified RECIST 1.1 may be eligible for retreatment with pembrolizumab + IPI or pembrolizumab monotherapy if they progress after stopping pembrolizumab at the discretion

MK-3475-029-05 Final Protocol 7-Nov-2017


**Protocol/Amendment No.:** 029-05

of the investigator according to the criteria in Section 7.1.5.2.1 as long as Part 1C remains open. Second Course Phase will be administered for a maximum of 17 doses of pembrolizumab and 4 doses of IPI.

After the end of treatment, each subject will be followed for 30 days for AE monitoring (SAEs will be collected for 90 days after the end of treatment). Subjects who discontinue treatment for reasons other than disease progression will have SFU for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone contact for OS until death, withdrawal of consent or the end of the trial, whichever comes first.

All subjects will be required to submit a tumor tissue sample for biomarker analyses and PD-L1 expression evaluation. Confirmation of the tumor tissue sample adequacy for determination of PD-L1 status by IHC at a central pathology laboratory is not required prior to enrollment in Part 1C.

The trial will be conducted in conformance with Good Clinical Practices.

Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the Trial Flow Chart - Section 6.0. Details of each procedure are provided in Section 7.0 – Trial Procedures.

Based on the data from Part 1A, pembrolizumab + PEG-IFN combination will not be pursued any further due to lack of added efficacy with the combination compared with pembrolizumab monotherapy, as well as the added toxicities. Part 1B further supported the early efficacy of pembrolizumab + IPI seen in Part 1A and confirmed a DRAE rate of 42% (data cutoff date March 17, 2016). Based on the goal to further minimize the AE profile of pembrolizumab + IPI, Part 1C has been designed to investigate two different dosing regimens of pembrolizumab + IPI. The previously described Part 2 in this protocol has been deleted as it is no longer applicable based on now available data from Parts 1A and 1B.

Upon consultation with the Sponsor, subjects in Part 1A, 1B and 1C may be eligible for Second Course Phase if they progress after stopping pembrolizumab as long as the trial Part to which the subject was initially enrolled remains open as per Section 7.1.5.2.1. Subjects enrolled in Part 1A who received PEG-IFN who are eligible for Second Course Phase will only be allowed to receive pembrolizumab monotherapy.

Subjects may have the opportunity to transition to a pembrolizumab extension trial if available in the future after closure of this trial

#### 2.2 Trial Diagram

The trial design is depicted in Figure 1, Figure 2, and Figure 3 below.

Protocol/Amendment No.: 029-05



<sup>\*</sup>DL1 starting dose

Figure 1 Pembrolizumab + PEG-IFN Dose finding: Part 1A

Note that if dose levels are opened in both PEG-IFN and IPI Arms, subjects will be randomly assigned to the two combinations.



<sup>\*</sup>With the approval of Amendment 03, subjects continuing pembrolizumab treatment will switch to a fixed dose of 200 mg (not weight-based).

Figure 2 Pembrolizumab + IPI dose finding: Part 1A Safety run-in and Part 1B Expansion cohort in MEL subjects.

Expansion in MEL subjects will proceed once DL1 is declared safe on safety run-in (Part 1A).

MK-3475-029-05 Final Protocol

<sup>\*\*</sup>With the approval of Amendment 03, subjects continuing pembrolizumab treatment will switch to a fixed dose of 200 mg (not weight-based).

**Protocol/Amendment No.:** 029-05

With the approval of Amendment 03, subjects continuing pembrolizumab treatment on Parts 1A and 1B will switch to a fixed dose of 200mg q3w (not weight-based).



Figure 3 Part 1C – Phase I/II portion of the trial.

### 3.0 OBJECTIVE(S) & HYPOTHESIS(ES)

## 3.1 Primary Objective(s) & Hypothesis(es)

1. **Objective (Part 1A):** To establish a maximum tolerated dose (MTD) or a maximum administered dose (MAD) of pembrolizumab when given in combination with PEG-IFN to subjects with advanced MEL or RCC.

**Hypothesis:** The DLTs observed in subjects with advanced MEL or RCC after IV administration of pembrolizumab in each combination will allow for definition of an MTD or a MAD.

- 2. **Objective (Part 1A, 1B):** To establish the tolerability of pembrolizumab when given in combination with IPI at the DL1 (pembrolizumab 2 mg/kg or 200 mg IV q3w + IPI 1 mg/kg q3w) in subjects with advanced MEL or RCC.
- 3. **Objective (Part 1A, 1B):** To determine the safety and tolerability of pembrolizumab in combination with PEG-IFN or IPI in subjects with advanced MEL or RCC.

**Hypothesis:** IV administration of pembrolizumab in combination with PEG-IFN or IPI to subjects with advanced MEL or RCC is sufficiently well-tolerated to permit continued clinical investigation.

4. **Objective (Part 1C):** To establish the safety and tolerability of pembrolizumab in combination with either IPI 50 mg q6w or IPI 100 mg q12w in subjects with advanced MEL.

**Hypothesis:** IV administration of pembrolizumab in combination with IPI to subjects with advanced MEL is sufficiently well-tolerated to permit continued clinical investigation.

5. **Objective (Part 1C):** To determine the rate of Grade 3-5 DRAEs.

**Hypothesis:** IV administration of pembrolizumab in combination with either IPI 50 mg q6w or IPI 100 mg q12w will produce Grade 3-5 DRAEs that are <40-55% as

Protocol/Amendment No.: 029-05

observed with the combination of pembrolizumab + IPI 1 mg/kg in Part 1A and 1B. The criteria are described in section 8 – SAP.

6. Objective (Part 1C): To evaluate efficacy of pembrolizumab + IPI in subjects with advanced unresectable/metastatic MEL in Part 1C.

Hypothesis: IV administration of pembrolizumab in combination with either IPI 50 mg q6w or IPI 100 mg q12w will produce ORR rates similar to the 48% or higher observed with combinations of pembrolizumab + IPI 1 mg/kg in Part 1B.

#### 3.2 Secondary Objective(s) & Hypothesis(es)

1. Objective (Part 1B): To evaluate efficacy of pembrolizumab in combination with IPI in subjects with advanced unresectable/metastatic MEL.

**Hypothesis:** IV administration of pembrolizumab in combination with IPI to subjects with PD-L1 negative advanced MEL results in a clinically meaningful ORR through 24 weeks based on RECIST 1.1 by central independent review.

- 2. Objective (Part 1B, 1C): To evaluate the efficacy of pembrolizumab administered intravenously in combination with IPI with respect to ordinal response score [derived from RECIST 1.1 definitions, with PR being divided into Moderate Partial Response (MPR) and VGPR based on the degree of tumor shrinkage] in subjects with advanced MEL (more details in Section 8.2.5.1.4).
- 3. Objective (Part 1B, 1C): To evaluate the DOR in subjects with advanced MEL receiving pembrolizumab in combination with IPI.
- 4. **Objective (Part 1B, 1C):** To evaluate efficacy with respect to PFS of pembrolizumab in combination with IPI in subjects with advanced MEL.
- 5. Objective (Part 1B, 1C): To evaluate OS in subjects with advanced MEL receiving pembrolizumab in combination with IPI.
- **6.** Objective (Part 1A, 1B): To compare the rates of Grade  $\geq 3$  toxicities across all subjects treated with each doublet (pembrolizumab + PEG-IFN and pembrolizumab + IPI).

**Hypothesis**: Administration of pembrolizumab + PEG-IFN results in different rate of Grade 3-4 toxicity than pembrolizumab + IPI.

7. **Objective (Part 1B and 1C)**: To evaluate the relationship between PD-L1 expression on IHC to clinical outcomes (ORR, PFS and OS) in MEL subjects treated with pembrolizumab + IPI.

#### **Exploratory Objectives** 3.3

1. **Objective (Part 1A):** To evaluate efficacy with respect to PFS and ORR based on modified RECIST 1.1 by site investigator, ordinal response score, DOR and OS of pembrolizumab in combination with PEG-IFN or IPI in subjects with RCC.

**Protocol/Amendment No.:** 029-05

2. **Objective (Part 1A):** To evaluate the relationship between PD-L1 expression on IHC to clinical outcomes (ORR, PFS and OS) in Part 1A RCC subjects treated with pembrolizumab + IPI or pembrolizumab + PEG-IFN.

- 3. **Objective (Part 1A, 1B, 1C):** To investigate the relationship between candidate efficacy biomarkers and anti-tumor activity of pembrolizumab utilizing pre- and post-treatment biopsies and blood sampling using in vitro assays.
- 4. **Objective (Part 1A, 1B, 1C):** To evaluate ORR as determined by RECIST 1.1 criteria using line length compared to RECIST 1.1 criteria using tumor volumetric changes of subjects with MEL and RCC treated with pembrolizumab + IPI and pembrolizumab + PEG-IFN.
- 5. **Objective (Part 1A, 1B, 1C)**: To evaluate the rate of pembrolizumab anti-drug antibodies (ADA) and impact on PK when pembrolizumab is given in monotherapy and in combination with PEG-IFN or IPI.
- 6. **Objective (Part 1B):** To evaluate the best objective response rate (ORR) by RECIST 1.1 in subjects on pembrolizumab + IPI after re-induction with IPI.
- 7. **Objective (Part 1A, 1B, 1C):** To evaluate the ORR by RECIST 1.1 in subjects treated with pembrolizumab + IPI or pembrolizumab monotherapy as part of Second Course Phase.
- 8. **Objective (Part 1A, 1B, 1C):** To evaluate the use of time to growth (TTG) modeling and simulation and correlate with clinical outcomes in MEL and RCC subjects treated with pembrolizumab + PEG-IFN and pembrolizumab + IPI.

#### 4.0 BACKGROUND & RATIONALE

#### 4.1 Background

Pembrolizumab (previously known as SCH 900475 and MK-3475) is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2). Based on preclinical in vitro data, pembrolizumab has high affinity and potent receptor blocking activity for PD-1. Pembrolizumab has an acceptable preclinical safety profile and is in clinical development as an intravenous (IV) immunotherapy for advanced malignancies. Keytruda<sup>TM</sup> (pembrolizumab) is indicated for the treatment of patients across a number of indications. Refer to the Investigator's Brochure (IB)/approved labeling for detailed background information on PEG-IFN, IPI, and MK-3475.

#### 4.1.1 Pharmaceutical and Therapeutic Background

#### 4.1.1.1 Pembrolizumab

The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades [2]. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies [3] [4] [5] [6] [7]. In particular, the presence of CD8+ T-cells and the

MK-3475-029-05 Final Protocol 7-Nov-2017


Protocol/Amendment No.: 029-05

ratio of CD8+ effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in solid malignancies such as ovarian, colorectal and pancreatic cancer, hepatocellular carcinoma, malignant MEL and RCC. TILs can be expanded ex vivo and re-infused, inducing durable objective tumor responses in cancers such as MEL [8] [9].

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4 which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2) [10] [11]. The structure of murine PD-1 has been resolved [12]. PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail which is responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosinebased switch motif (ITSM). Following T-cell stimulation, PD-1 recruits the tyrosine phosphatases SHP-1 and SHP-2 to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ and ZAP70 which are involved in the CD3 T-cell signaling cascade [10] [13] [14] [15]. The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from that of CTLA-4 as both molecules regulate an overlapping set of signaling proteins [16] [17]. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, regulatory T cells (T regs) and Natural Killer cells [18] [19]. Expression has also been shown during thymic development on CD4-CD8- (double negative) T-cells as well as subsets of macrophages and dendritic cells [20]. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types, including non-hematopoietic tissues as well as in various tumors [1] [16] [21] [22] [23]. Both ligands are type I transmembrane receptors containing both IgV- and IgC-like domains in the extracellular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium, whereas PD-L2 protein is only detectably expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PD-L1 serves to dampen unwarranted T-cell function in peripheral tissues [16]. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. High expression of PD-L1 on tumor cells (and to a lesser extent of PD-L2) has been found to correlate with poor prognosis and survival in various cancer types, including RCC [24], pancreatic carcinoma [25], hepatocellular carcinoma [26], and ovarian carcinoma [27]. Furthermore, PD-1 has been suggested to regulate tumor-specific T-cell expansion in subjects with MEL [28]. This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

Protocol/Amendment No.: 029-05

Based on the preliminary clinical data, PD-1 inhibitors such as pembrolizumab appear to be attractive candidates for pursuing the above goal. Nivolumab has an observed ORR of 28% in MEL subjects; pembrolizumab has shown a promising response rate of 25% in MEL subjects who have received prior IPI treatment in KEYNOTE 002 [29]. Specifically, a response rate of 36% was observed with pembrolizumab in MEL subjects who have not received prior IPI treatment in KEYNOTE 006 [30]. This response rate is much higher than the 11-15% response rate observed with IPI in IPI registration trials.

On September 4, 2014, the Food and Drug Administration (FDA) granted accelerated approval for pembrolizumab 2mg/kg q3w in advanced MEL following disease progression with IPI and, if BRAF V600 mutation positive, a BRAF inhibitor [31]. The approval was based on a strong efficacy and safety profile demonstrated in 4 MEL expansion parts of the Phase I trial (KEYNOTE 001) [32]; the B2 IPI-refractory population was the subject population for the approval. On December 18, 2015, the FDA granted full approval of pembrolizumab for the treatment of subjects with unresectable or metastatic MEL with pembrolizumab based on KEYNOTE 002 and 006 [30] [33].

## 4.1.1.2 Pegylated Interferon Alfa-2b (PEG-IFN)

PEG-IFN is a pleiotropic cytokine with anti-viral, anti-proliferative, anti-angiogenic and immunomodulatory properties. PEG-IFN is a modified form of IFN  $\alpha$ -2b comprising a single molecule of polyethylene glycol (PEG) covalently linked to the IFN α-2b protein. PEG-IFN has shown good tolerability and similar efficacy to conventional interferon and dacarbazine single agent chemotherapy in stage IV MEL [34]. Based on the European Organization for Research and Treatment of Cancer (EORTC) 18991 trial, the United States (US) Food and Drug Administration (FDA) approved PEG-IFN for the adjuvant treatment of MEL subjects following definitive surgical resection, including complete lymphadenectomy [35] [36]. PEG-IFN α-2b was administered at 6 µg/kg/week subcutaneously for 8 weeks (induction phase) then at 3 µg/kg/week subcutaneously (maintenance phase) for an intended treatment duration of 5 years. There was an 18% reduction in the risk of relapse and death. PEG-IFN was safe and relatively well tolerated. The median length of therapy with PEG-IFN  $\alpha$ -2b was >12 months. The most commonly observed side-effects were fatigue, alanine and aspartate aminotransferase elevations and fever, myalgia, anorexia and nausea. A total of 525 deaths were reported during the trial (262 in the PEG-IFN group and 263 in the observation group). The most frequent causes of death were infection, malignant disease and cardiovascular disease. 31% of the 608 subjects who were treated with PEG IFNα-2b discontinued therapy due to Grade 3-4 AEs: fatigue (25%), anorexia (15%), depression (16%), liver function tests (13%), headache (12%), nausea (12%), and pyrexia (11%).

IFN- $\alpha$  used to be the mainstay of therapy for advanced RCC. ORRs ranged from 15-25%, with 5-10% of these subjects having durable responses. Targeted therapies with VEGF and mTOR inhibitors have largely replaced IFN-based regimens due to the ease of use and the higher efficacy, notably in term of PFS. Nevertheless, IFN- $\alpha$  remains an option in metastatic RCC. Furthermore, some front-line trials with an IFN- $\alpha$  comparator vs. a targeted therapy (sorafenib) did not show a PFS advantage [37], and the majority of trials did not show an OS advantage. The pegylated form of IFN- $\alpha$  is easier to use, may have less side effects [38] and

Protocol/Amendment No.: 029-05

it is not an unreasonable choice especially in subjects who failed prior standard targeted therapies.

Refer to the Investigator's Brochure (IB)/approved labeling for detailed background information on PEG-IFN.

#### 4.1.1.3 **Ipilimumab (IPI)**

Ipilimumab (Yervoy®) is an immunoregulatory agent that blocks CTLA-4 to promote anti-tumor immunity. In a Phase III study of 676 subjects with unresectable or metastatic MEL whose disease had progressed while receiving prior therapy for metastatic disease, IPI administered at 3 mg/kg q3w for up to 4 doses with or without a gp100 peptide vaccine was compared with gp100 alone [39]. The median OS was 10.1 months and 10.0 months for the IPI alone and IPI plus gp100 Arms respectively, while the median OS was 6.4 months for the gp100 alone Arm (p<0.001). An ORR of 10.9% was observed in IPI alone Arm, while the IPI plus gp100 Arm and gp100 alone Arm had lower response rates, 5.7% and 1.5%, respectively. The median duration of response was 11.5 months in the IPI plus gp100 Arm, and not reached in the IPI alone Arm with a median follow-up period of 27.8 months. The median time to progression was 2.86 months for the IPI alone Arm and 2.76 months for the other two Arms. In the IPI alone Arm, 97% of the subjects experienced an AE and Grade 3-4 AEs occurred in 46% of the subjects. The most common AEs related to IPI were immune-related events, which occurred in approximately 60% of the subjects treated with IPI and 32% of the subjects treated with gp100. The frequency of Grade 3-4 immune-related AEs was 15%. The immune-related AEs most often affected the skin and gastrointestinal tract, including pruritus, rash, vitiligo, diarrhea, and colitis.

Based on the above Phase III trial, IPI was approved by the FDA for treatment of subjects with unresectable or metastatic MEL and by the European Commission for treatment of subjects with previously-treated advanced MEL. The recommended regimen is 3 mg/kg administered q3w for a total of four doses.

A reduction of the risk of death (28%; p<0.001) was also demonstrated for IPI in the firstline setting when combined with dacarbazine in comparison with dacarbazine alone, and the ORRs were 15% and 10% (Investigator assessment per RECIST 1.1) in the IPI/dacarbazine Arm and dacarbazine alone Arm, respectively [40]. The IPI/dacarbazine Arm did show a statistically significant PFS improvement [hazard ratio (HR) 0.76; p=0.006] over the dacarbazine alone Arm. Median OS in the IPI/dacarbazine and dacarbazine Arms was 11.2 months and 9.1 months, respectively. The one-year OS rate for the IPI/dacarbazine Arm was 47.3%; the rate for the dacarbazine Arm was 36.3%.

In RCC, a Phase I/II trial by Yang revealed an ORR 9.8% [41], across different dose levels, in subject's treatment naïve and previously treated with interleukin-2. Given the greater response rates seen with tyrosine kinase inhibitors, IPI was not further developed as monotherapy in RCC.

Refer to the approved labeling for detailed background information on IPI.

**Protocol/Amendment No.:** 029-05

#### 4.1.2 Pre-clinical Trial with Pembrolizumab

Therapeutic studies in mouse models have shown that administration of antibodies blocking PD-1/PD-L1 interaction enhances infiltration of tumor-specific CD8+ T-cells and leads ultimately to tumor rejection, either as a mono-therapy or in combination with other treatment modalities. Anti-mouse PD-1 or anti-mouse PD-L1 antibodies have demonstrated anti-tumor responses as a monotherapy in models of squamous cell carcinoma, pancreatic carcinoma, MEL and colorectal carcinoma. Blockade of the PD-1 pathway effectively promoted CD8+ T-cell infiltration into the tumor and the presence of IFN-γ, granzyme B and perforin, indicating that the mechanism of action involved local infiltration and activation of effector T-cell function in vivo [28] [42] [43] [44] [25] [45]. Experiments have confirmed the in vivo efficacy of PD-1 blockade as a monotherapy as well as in combination with chemotherapy in syngeneic mouse tumor models (see the Investigator's Brochure [IB]).

## 4.1.3 Ongoing Clinical Trials

Ongoing clinical trials are being conducted in advanced MEL, non-small cell lung cancer (NSCLC), head and neck cancer, triple negative breast cancer, gastric cancer, bladder cancer and hematologic malignancies. For trial details please refer to the IB.

#### 4.2 Rationale

## 4.2.1 Rationale for the Trial and Selected Subject Population

MEL is the sixth most common malignancy in men and the seventh most common malignancy in women. The incidence of MEL is increasing worldwide, with a growing fraction of subjects with advanced disease for which prognosis remains poor. The median survival for subjects with metastatic MEL has been under 1 year. The 5-year survival rate of subjects with visceral involvement is under 10%. Treatment options for metastatic MEL have been limited to chemotherapeutic agents such as dacarbazine and high-dose interleukin-2 immunotherapy in a small percentage of subjects. In the past few years there has been steady progress in the development of targeted therapy and immunotherapy for metastatic MEL. Since 2011, three new agents were approved for the treatment of BRAF mutant MEL: vemurafenib, dabrafenib and trametinib, which produce response rates of 22-57% and have demonstrated a survival advantage relative to chemotherapy [46] [47] [48]. It is important to note these agents are not indicated for up to 60% of MEL subjects whose tumors do not contain a BRAF mutation [47] [46] [49] [50]. In addition, a major limitation with kinase inhibitors in the treatment of BRAF mutant MEL is a nearly universal development of resistance to these agents leading to the lack of response durability. Although high RRs offer benefits to the majority of subjects with BRAF mutant MEL, most subjects develop resistance rather quickly and experience progressive disease (PD).

IPI, an anti-CTLA4 monoclonal antibody, was also approved in 2011 for the treatment of subjects with unresectable or metastatic MEL based on the data described in Section 4.1.1.3. More recently, IPI has demonstrated increased efficacy in combination with nivolumab in 2 randomized phase III clinical trials. In CheckMate 069 [51], 142 patients with previously untreated metastatic MEL were randomly assigned to receive IPI 3 mg/kg combined with

04SGNN Confidential

Protocol/Amendment No.: 029-05

either nivolumab, 1 mg/kg, or placebo once q3w for 4 doses, followed by nivolumab 3 mg/kg every 2 weeks until disease progression or unacceptable toxic effects. ORR was 61% in the group that received both IPI and nivolumab versus 11% in the group that received IPI monotherapy (p<0.001). After a minimum follow-up of 18 months, median PFS was not reported with the combination therapy and was 4.3 months with IPI monotherapy [HR 0.34]: 95% confidence interval (CI): 0.2, 0.57; p<0.0001] [52]. The 12- and 18-month PFS rates were 55.1% and 53.4%, respectively, for the combination, and 16.2% and 8.1%, respectively, for IPI alone. At 18 months of follow-up, OS rates in BRAF wild-type patients were 73% for the combination versus 56% for IPI alone, and median OS had not been reached in either group (HR 0.56; 95% CI: 0.29, 1.10; p=0.089). Grade 3-4 DRAEs were reported more frequently with the combination than with IPI alone (55% vs. 22%) and led to discontinuation in 30% and 9% of patients, respectively [52]. In CheckMate 067, 945 subjects with unresectable stage III or IV MEL were randomly assigned in a 1:1:1 ratio to receive nivolumab 3 mg/kg every 2 weeks, nivolumab 1 mg/kg q3w plus IPI 3 mg/kg q3w for 4 doses followed by nivolumab 3 mg/kg every 2 weeks for Cycle 3 and beyond, or IPI 3 mg/kg q3w for 4 doses [53]. The median PFS was 11.5 months (95% CI: 8.9, 16.7) with nivolumab plus IPI, 2.9 months (95% CI: 2.8, 3.4) with IPI (HR 0.42; 99.5% CI: 0.31, 0.57; p < 0.001), and 6.9 months (95% CI: 4.3, 9.5) with nivolumab (HR for the comparison with IPI, 0.57; 99.5% CI: 0.43, 0.76; p<0.001). DRAEs of Grade  $\geq$  3 were reported in 16.3% of the subjects treated with nivolumab, 55.0% of the subjects treated with the combination, and 27.3% of those treated with IPI alone. On September 30, 2015, the FDA granted accelerated approval to nivolumab in combination with IPI for the treatment of subjects with BRAF V600 wild-type, unresectable or metastatic MEL. Approval was based on demonstration of an increase in the ORR, prolonged response durations, and improvement in PFS observed in CheckMate 069 trial.

RCC is the seventh most common cancer among US men and ninth among US women. Twenty percent of people present with advanced disease, and an additional 30% of those who present with localized disease will eventually develop distant metastases and become largely incurable. The targeted drugs, pazopanib, sunitinib, sorafenib, axitinib, bevacizumab, everolimus, and temsirolimus transformed the management of metastatic RCC after demonstration of superiority to cytokine therapy and placebo in pivotal phase III trials [54] [55] [56] [57]. Cytokine-based treatment with interleukin-2 (IL-2) or interferon-α (IFN-α) used to be the mainstay of therapy for RCC and can still benefit a small proportion of subjects.

More recently, nivolumab has been shown to improve OS in the second-line setting for subjects with previously treated advanced clear-cell RCC compared with everolimus; 25 months (95% CI: 21.8, not estimable) with nivolumab and 19.6 months (95% CI: 17.6, 23.1) with everolimus) [58]. The HR for death with nivolumab versus everolimus was 0.73 (98.5% CI: 0.57, 0.93; P=0.002). ORR was greater with nivolumab than with everolimus (25% vs. 5%; odds ratio, 5.98 (95% CI: 3.68, 9.72); P<0.001). The median PFS was 4.6 months (95% CI: 3.7, 5.4) with nivolumab and 4.4 months (95% CI: 3.7, 5.5) with everolimus (HR 0.88; 95% CI: 0.75, 1.03; P=0.11).

This is a multi-center, open-label, 3-part Phase I/II trial of pembrolizumab in combination with PEG-IFN or IPI in subjects with advanced or metastatic MEL and RCC. Subjects with

**Protocol/Amendment No.:** 029-05

advanced or metastatic MEL with any prior lines of therapy (Part 1A and 1B) and subjects with advanced or metastatic RCC with  $\geq 1$  line of therapy (Part 1A only) as well as subjects with advanced or metastatic MEL with no prior lines of therapy (Part 1C) will be enrolled in this trial.

Details regarding specific benefits and risks for subjects participating in this clinical trial may be found in the accompanying IB and Informed Consent documents.

### 4.2.1.1 Rationale for Evaluating anti-PD-1 Therapy in Advanced Melanoma and Renal Cell Carcinoma

#### 4.2.1.1.1 Rationale for Pembrolizumab

Pembrolizumab is a highly specific humanized anti-PD-1 antibody, which has shown to be very well-tolerated and lead to ORRs in MEL subjects of 36% [59]. KEYNOTE 006, a phase III trial, has demonstrated superior efficacy of pembrolizumab compared to IPI in PFS, OS and ORR, with an estimated 46.4% 6-month PFS rate versus 26.5% for IPI. The ORR was 32.9% for pembrolizumab versus 11.9% for IPI. Responses were ongoing in 96.7% of subjects after a median follow-up of 7.9 months. One-year estimates of survival for subjects receiving pembrolizumab q3w were 68.4% compared with IPI 58.2% (HR for death as compared with IPI 0.69; 95% CI: 0.52, 0.90; p=0.0036). Because the OS results were superior to IPI, the external Data Monitoring Committee (DMC) recommended stopping the study early to allow patients on IPI who progressed the option of receiving pembrolizumab [30].

Blockage of the PD-1/PD-L1 pathway also appears to be effective in a heavily pre-treated population with metastatic RCC [60] [61], leading to ORRs of up to approximately 29%.

## 4.2.1.1.2 Rationale for PEG-IFN

IFNα, the active component of PEG-IFN, is a pleiotropic cytokine, with anti-angiogenic and immunomodulatory properties. In MEL, IFN $\alpha$  is approved in the adjuvant setting. While IFN treatment as monotherapy has shown some clinical activity in metastatic MEL [62], IFN in metastatic MEL is only used as part of bio-chemotherapy combination regimens, albeit rarely [63] [64].

In RCC, IFNα has shown similar clinical activity as sorafenib, a tyrosine kinase inhibitor, in the first line setting [38]. Currently in metastatic RCC, IFNa is used in combination with bevacizumab [54], an anti-angiogenesis antibody targeting VEGF-A (vascular endothelial growth factor-A).

# 4.2.1.1.2.1 Hypothesis for Pembrolizumab + PEG-IFN Combination Therapies

Internal pre-clinical studies have shown that IFNα increases the expression of PD-L1 in RCC and MEL cell lines, as well as in breast cancer histoculture (data not published). In a pre-clinical study by Terawaki and others, IFNα increased PD-1 expression in tumor infiltrating lymphocytes (TILs) in MC38 (mouse colorectal) model [65].

Protocol/Amendment No.: 029-05

This study also evaluated the potential additive anti-tumor effect of the combination IFNα and anti-PD-1. In their experiment, mice received SC tumor implants in the flank, then received IFNα daily from Days 1–13. Anti-PD-1 (4H2) antibody was given at doses of 6 or 20 mg/kg on Days 0 and 3, or of 10 mg/kg three times with a 6-day interval. Figure 4A illustrates the mean tumor volumes in mice treated with IFN $\alpha$ , anti-PD-1 or the combination, showing a greater tumor control when both agents were given in combination. Figure 4B illustrates the individual tumor volumes in these mice. The median size of tumors was smaller in the animals treated with the combination IFNα+Anti-PD-1 and a greater number of mice had profound responses (tumors smaller than 100mm<sup>3</sup>, dashed line). None of the 15 animals treated with IFNα had profound responses, whereas a total of 9 out of 30 animals treated with 4H2 (at 3 and 10 mg/kg), and 12 out of 30 animals treated with IFNα+4H2 (at 3 and 10 mg/kg) were nearly disease free.



Figure 4 Effect of IFNα and Anti-PD-1 in MC38 models

#### 4.2.1.1.3 Rationale for IPI

IPI (Yervoy®) is approved for treatment of metastatic MEL, as it has shown OS advantage compared with peptide vaccine [66]. IPI monotherapy has shown modest activity in RCC [41]; however, it is not being further developed as a single agent.

## 4.2.1.1.3.1 Hypothesis for Pembrolizumab + IPI Combination Therapies

Pre-clinical studies have shown that concomitant CTLA-4 and PD-1 blockage elicited greater response rates than either single agent in MC38 mouse models [67]. Notably, while no mice treated with anti-CTLA-4 or anti-PD-1 were free of disease at the end of the experiment, 7-60% of mice treated with the combination at various dose levels were tumor free. This served as the foundation to explore anti-CTLA-4 in combination with anti-PD-1 in the clinical setting.

In a Phase 1 trial in subjects with MEL, IPI (anti-CTLA-4) combined with nivolumab (anti-PD-1) led to response rates ranging from 21-53%. These may represent greater responses than nivolumab monotherapy [68] [69] and historical responses to IPI in monotherapy (approximately 20-31% and 10%, respectively) [66]. As mentioned above, both anti-PD-1 antibodies nivolumab and pembrolizumab demonstrated superiority over single-agent IPI in

**Protocol/Amendment No.:** 029-05

previously untreated subjects (pembrolizumab), and over chemotherapy both in untreated subjects and after failure of IPI (nivolumab, pembrolizumab). The addition of IPI to nivolumab is associated with a higher response rate and a better PFS; however, it is associated with a high rate of Grade 3-4 DRAEs.

### Rationale for Dose Selection/Regimen/Modification

An open-label Phase I trial (KEYNOTE 001) was conducted to evaluate the safety and clinical activity of single agent pembrolizumab. The dose escalation portion of this trial evaluated three dose levels, 1 mg/kg, 3 mg/kg, and 10 mg/kg, administered every 2 weeks (q2w) in subjects with advanced solid tumors. All three dose levels were well-tolerated and no dose-limiting toxicities were observed. This first in human trial of pembrolizumab showed evidence of target engagement and objective evidence of tumor size reduction at all dose levels (1 mg/kg, 3 mg/kg and 10 mg/kg q2w). No MTD has been identified to date.

PK data analysis of pembrolizumab administered q3w showed slow systemic clearance, limited volume of distribution, and a long half-life (refer to IB). Pharmacodynamic data (IL-2 release assay) suggested that peripheral target engagement is durable (>21 days). This early PK and pharmacodynamic data provides scientific rationale for starting the dose escalation with a q3w dosing schedule for pembrolizumab.

The dose of pembrolizumab with Amendment 03 is 200 mg q3w. The dose recently approved in the United States and several other countries for treatment of MEL and NSCLC subjects is 2 mg/kg q3w. Information on the rationale for selecting 200 mg q3w is summarized below.

An integrated body of evidence suggests that 200 mg q3w is expected to provide similar response to 2 mg/kg q3w, 10 mg/kg q3w and 10 mg/kg q2w. A flat pembrolizumab exposure-response relationship for efficacy and safety has been found in subjects with MEL as well as NSCLC in the range of doses between 2 mg/kg and 10 mg/kg. Exposures for 200 mg q3w are expected to lie within this range and will be close to those obtained with 2 mg/kg q3w dose.

A population PK model, which characterized the influence of body weight and other patient covariates on exposure, has been developed. The PK profile of pembrolizumab is consistent with that of other humanized monoclonal antibodies, which typically have a low clearance and a limited volume of distribution. The distribution of exposures from the 200 mg fixed dose are predicted to (1) considerably overlap with those obtained from the 2 mg/kg dose and (2) maintain the individual patient exposures within the exposure range established in MEL to be associated with maximal clinical response. PK properties of pembrolizumab, and specifically the weight-dependency in clearance and volume of distribution are consistent with no meaningful advantage to weight-based dosing relative to fixed dosing.

In translating to other tumor types, similarly flat exposure-response relationships for efficacy and safety as observed in subjects with MEL can be expected, as the anti-tumor effect of pembrolizumab is driven through immune system activation rather than through a direct interaction with tumor cells, rendering it independent of the specific tumor type. In addition, available PK results in subjects with MEL, NSCLC, and other tumor types support a lack of

**Protocol/Amendment No.:** 029-05

meaningful difference in PK exposures obtained at tested doses among tumor types. Thus, the 200 mg q3w fixed dose regimen is considered an appropriate fixed dose for other tumor types as well.

A fixed dose regimen will simplify the dosing regimen to be more convenient for physicians and to reduce potential for dosing errors. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities and reduce wastage. Based on the existing data, 200 mg q3w is the appropriate dose for pembrolizumab.

In the pembrolizumab + PEG-IFN treatment Arms, the dose finding portion of this trial will evaluate up to four doses of PEG-IFN, 0.5  $\mu$ g/kg, 1  $\mu$ g/kg, 2 $\mu$ g/kg, and 3  $\mu$ g/kg, administered SC weekly. A lower dose of PEG-IFN, 0.5  $\mu$ g/kg/week, will be evaluated as DL-1, if needed.

As single agent, PEG-IFN is tolerated at doses higher than 3  $\mu$ g/kg weekly dose; the MTD was defined at 7.5-9  $\mu$ g/kg and 6  $\mu$ g/kg weekly, respectively, in subjects with CML and solid tumors [70] [71]. These studies showed a trend toward a dose-related increase of AEs. Lower rates of AEs were also seen when single agent non-pegylated IFN $\alpha$  was given at lower (5MU total/week) versus higher doses (25 MU total/week) in a randomized trial in RCC subjects [72]).

In combination with other immune-modulators, PEG-IFN 3  $\mu g/kg/week$  was found to be tolerable when given with IL-2 three times per week in subjects with RCC [73]. More recently, PEG-IFN was tolerated at 2  $\mu g/kg/week$  in combination with standard dose IPI, in subjects with MEL [74].

In addition to the greater tolerability, lower PEG-IFN doses  $(3\mu g/kg/week)$  and below, or the equivalent of non-pegylated IFN) have shown biological activity as single agent and in combinations. In RCC, a Phase I trial using PEG-IFN doses of 0.5- $2\mu g/kg$  revealed an ORR of 14% [75]. A previously mentioned RCC trial used low dose non-pegylated IFN $\alpha$ , 0.5 MU twice/day (5 MU total/week), versus higher doses of IFN $\alpha$ , 5 MU/day (25 MU total/week) showing the same ORR 6.7%, including a CR, and yielded a trend to better OS in the low dose IFN group, 25.5 months and 17.5 months, respectively [72]. These doses correspond to less than 0.25 $\mu$ g/kg to approximately  $1\mu$ g/kg weekly doses of PEG-IFN [70] In addition, larger trials used non-pegylated IFN $\alpha$  at 9 MIU/kg three times/week (27 MU/week corresponding approximately to PEG-IFN  $1\mu$ g/kg weekly), yielded an ORR of 13% [76] [77]. In MEL, low dose PEG-IFN $\alpha$ 2a (with same active principle, but a different PEG moiety) yielded an ORR of 6% in 48 subjects [36], including a CR.

In the combination setting, low dose IFN $\alpha$  (9 MU/week) with bevacizumab [78] appeared to have similar efficacy and a favorable side effect profile compared with historical data on standard dose IFN $\alpha$  (27 MU/week) plus bevacizumab [79]. Despite small numbers (3 PR/10 evaluable subjects), results of low dose PEG-IFN in combination with IPI also appear promising [74].

Given the toxicities associated with higher doses of IFN, this trial will investigate doses of up to 3  $\mu$ g/kg/week of PEG-IFN. These are biologically active doses, aiming at priming the immune system and increasing responses to anti-PD-1 therapy. The overall dosing strategy is

Protocol/Amendment No.: 029-05

intended to emphasize dose intensity with pembrolizumab rather than PEG-IFN, due to the known safety and efficacy of both agents.

In the pembrolizumab + IPI treatment Arms of Part 1A and 1B, pembrolizumab will be evaluated in combination with IPI 1 mg/kg. The schedule of IPI will follow the approved drug label of q3w. In a Phase I study by Sznol at ESMO 2013, efficacy of nivolumab 3 mg/kg + IPI 1 mg/kg (ORR 40% (95% CI 16-68%) and Aggregate Clinical Activity Rate (ACAR; defined as CR + PR + unconfirmed CR+ unconfirmed PR+ immune-related PR+ SD >24 week + irSD >24 week) 73%] appeared to have similar efficacy as nivolumab 1mg/kg + IPI 3 mg/kg (ORR 53% (95% CI 28-77%) and ACAR 65%) [68]. In addition, the combination of nivolumab 3 mg/kg + IPI 1 mg/kg showed lower rate of Grade 3-4 DRAEs compared with nivolumab 1 mg/kg + IPI 3 mg/kg (44% versus 65%, respectively). A total of 6/28 (21%) of patients experienced Grade 3-4 toxicities that were found to be dose-limiting.

The overall dosing strategy is intended to emphasize dose intensity with pembrolizumab rather than IPI; in addition, the dosing paradigm of anti-PD-1+ anti-CTLA4 combination will explore the lowest therapeutic dose of anti-PD-1 (pembrolizumab at 2 mg/kg q3w) and a lower dose than recommended monotherapy dose of anti-CTLA4 (IPI at 1 mg/kg q3w x 4 doses) in Part 1A as a safety run-in, due to known safety and efficacy profile of both agents. Up to 18 subjects will receive pembrolizumab 2 mg/kg q3w + IPI 1 mg/kg q3w x 4 doses. Once DL1 (pembrolizumab 2mg q3w + IPI 1mg/kg q3w x4 injections) is declared safe, dose expansion at DL1 in MEL subjects (Part 1B) will proceed.

In the pembrolizumab + IPI treatment Arms of Part 1C, the dose of pembrolizumab will be 200 mg q3w based on the rationale provided above. The dose of IPI will be 50 mg fixed dose g6w (Arm 1) and 100 mg IPI fixed dose g12w (Arm 2). The dose of IPI approved in the US and several other countries for treatment of MEL is 3 mg/kg q3w. Information on the rationale for selecting IPI 50 mg q6w and 100 mg q12 w is summarized below.

Results of 153 MEL patients in Part 1B show that lower doses of IPI (1 mg/kg q3w) in combination with pembrolizumab 2mg/kg q3w have a confirmed ORR of 57% by independent central review and a comparable rate of Grade 3-4 DRAEs to nivolumab 3 mg/kg + IPI 1 mg/kg (42 vs 44%) [53] or nivolumab 3 mg/kg + IPI 3mg/kg (55% and 54%) for CheckMate 067 and CheckMate 069, respectively) [53] [80]. In Part 1B, 72% of the subjects were able to complete all 4 planned doses of IPI, however, DRAEs were present in 42% of the subjects. To improve the safety and tolerability of the combination, pembrolizumab + IPI, lower doses as well as increased dosing interval of IPI will be explored in Part 1C.

An integrated body of evidence suggests that in combination with a PD-1 inhibitor, IPI 50 mg q6w and 100 mg q12w is expected to provide a similar response to IPI 1 mg/kg q6w and IPI 1 mg/kg g12w, respectively. Both IPI 1 mg/kg g6w and 1 mg/kg g12w have been shown to be effective when combined with nivolumab 3 mg/kg in subjects with NSCLC [81]. Simulations of PK profiles suggest that the systemic exposure and trough concentrations (Ctrough=pre-dose serum concentration of drug) for IPI 50 mg q6w are between those for IPI 1 mg/kg q12w and IPI 1 mg/kg q6w, and those for IPI 100 mg q12w overlap with IPI 1mg/kg g12w. The increased dosing interval (g6w or g12w) compared to the approved dosing

Protocol/Amendment No.: 029-05

interval for IPI monotherapy (q3w) may potentially increase the duration of time with IPI coverage and maintain IPI exposure for a longer time interval, while the lower Cmax (Cmax=maximum serum concentration of drug) may improve tolerability. The existing data suggest IPI 50 mg q6w and IPI 100 mg q12w are appropriate doses for IPI in combination with pembrolizumab 200 mg q3w.

The proposal to use fixed dose for IPI compared to weight-based dosing is supported by the published population PK analysis for IPI [82]. An allometric relationship is reported between IPI clearance and body weight, with estimated allometric coefficient of 0.642, which is consistent with no advantage for weight-based dosing compared to a fixed dose with respect to controlling exposure variability [83].

A fixed dose regimen is expected to simplify the dosing regimen (potentially reducing dosing errors), as well as be more convenient for physicians. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities, as well as reducing waste.

#### 4.2.3 Rationale for Endpoints

#### 4.2.3.1 Safety Endpoints

The primary safety objective of this trial is to characterize the safety and tolerability of pembrolizumab in combination with PEG-IFN or IPI in subjects with advanced MEL and RCC. The primary safety analysis will be based on subjects who experienced toxicities as defined by CTCAE criteria. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received pembrolizumab, including SAEs and events of clinical interest (ECIs).

Safety will be assessed by reported adverse experiences using CTCAE Version 4.0. The attribution to drug, time-of-onset, duration of the event, its resolution, and any concomitant medications administered will be recorded. AEs will be analyzed including but not limited to all AEs, SAEs, fatal AEs, and laboratory changes. Furthermore, potential immune-related adverse events (irAEs) will be collected and designated as immune-related ECIs as described in Section 7.2.3.2.

#### 4.2.3.2 Efficacy Endpoints

The primary efficacy objective of this trial is to evaluate the anti-tumor activity of pembrolizumab in subjects with advanced MEL treated with pembrolizumab in combination with PEG-IFN or IPI. Response rates per RECIST 1.1 and volumetric analysis will be evaluated.

The primary response rate efficacy endpoint will be based on independent central review using RECIST 1.1 (see Appendix 12.6) [1]. RECIST 1.1 will also be used by the local site to determine eligibility and make treatment decisions. For this later purpose, RECIST 1.1 will be adapted to account for the unique tumor response profile seen with treatment of pembrolizumab and this adapted/modified RECIST 1.1 will be used by the sites for treatment decisions. Modified RECIST 1.1 will also be used by the local site to determine eligibility. The primary efficacy endpoint is ORR, based on RECIST 1.1. Secondary endpoints are listed


07W8HB
**Protocol/Amendment No.:** 029-05

in section 3.2. As data permits, same efficacy endpoints will also be evaluated in Part 1A RCC subjects.

Immunotherapeutic agents such as pembrolizumab may produce antitumor effects by potentiating endogenous cancer-specific immune responses which may be functionally anergic. The response patterns seen with such an approach may extend beyond the typical time course of responses seen with cytotoxic agents, and can manifest a clinical response after an initial increase in tumor burden or even the appearance of new lesions. Standard RECIST criteria may not provide an accurate assessment of immunotherapeutic agents such as pembrolizumab. Therefore, RECIST 1.1 will be used with the following adaptation:

If radiologic imaging shows PD, tumor assessment should be repeated  $\geq 4$  weeks later in order to confirm PD with the option of continuing treatment per below while awaiting radiologic confirmation of progression. If repeat imaging shows a reduction in the tumor burden compared to the initial scan demonstrating PD, treatment may be continued as per treatment calendar. If repeat imaging confirms PD, subjects will be discontinued from trial therapy (exception noted in Section 7.1.2.8). In determining whether or not the tumor burden has increased or decreased, investigators should consider all target lesions as well as non-target lesions (please refer to the Site Imaging Manual).

In subjects who have initial evidence of radiological PD, it is at the discretion of the treating physician whether to continue a subject on study treatment until repeat imaging is obtained a minimum of 4 weeks later. This decision should be based on the clinical judgment of the subject's overall clinical condition, including performance status, clinical symptoms, and laboratory data. Subjects may receive treatment while waiting for confirmation of PD if they are clinically stable as defined by the following criteria:

- Absence of signs and symptoms (including worsening of laboratory values) indicating clinically significant disease progression
- No decline in Eastern Cooperative Oncology Group (ECOG) performance status
- Absence of rapid progression of disease
- Absence of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention

When feasible, subjects should not be discontinued until progression is confirmed. This allowance to continue treatment despite initial radiologic progression takes into account the observation that some subjects can have a transient tumor flare in the first few months after the start of immunotherapy, but with subsequent disease response. Subjects that are deemed clinically unstable or who have biopsy proven new metastatic lesions are not required to have repeat imaging for confirmation of PD.

Note: Treatment may be continued despite modified RECIST 1.1 defined progression if the subject is clinically stable and is considered to be deriving clinical benefit by the investigator. In these cases, subjects should continue to undergo imaging as outlined in the footnote in Table 11.

Protocol/Amendment No.: 029-05

Retrospective central review of all imaging time points may be performed for this study using volumetric analysis. Additional information is included in the Site Imaging Manual.

## 4.2.3.3 Planned Exploratory Biomarker Research

Tumor tissue for biomarker analysis from formalin fixed paraffin embedded tumor tissue sample or newly obtained formalin fixed biopsy of a tumor lesion not previously irradiated must be provided in the form of a tissue block or at least ten unstained slides and received by the central vendor before randomization.

Subjects must submit the tumor sample during screening. Subjects will be eligible to participate regardless of the level of PD-L1 expression. Subjects who do not submit a sample adequate for PD-L1 determination will not be enrolled in Part 1A or 1B. Subjects with an archival sample considered not acceptable may obtain a new biopsy. Subjects with a newly obtained biopsy considered not acceptable may undergo re-biopsy at the discretion of the investigator. Note for Part 1C: adequacy of the tumor sample for determination of PD-L1 status by IHC at the central pathology laboratory prior to enrollment is not required. Additional biopsy sample submission is encouraged but not mandatory for Part 1C when the sample is inadequate for PD-L1 testing.

Note: A fine needle aspirate, frozen sample, plastic embedded sample, bone, bone marrow, cell block, clot, or cytologic specimen will not be acceptable.

If new scientific data emerge that indicate that an existing biopsy or surgical specimen is suboptimal for identification of subjects, then only new biopsies will be acceptable for determination of PD-L1 status.

Biomarker research to identify factors important for pembrolizumab monotherapy or treatment doublets may also be pursued. For example, pre- and post-dose tumor (posttreatment tumor biopsies are optional at 12 weeks and upon progression) and blood samples from this study may undergo proteomic, genomic and transcriptional analyses. Additional research may evaluate factors important for predicting responsiveness or resistance to pembrolizumab monotherapy or doublets therapy and other immunologic targets.

Assays may include but are not be limited to:

## Multiparametric (Two-Color) IHC

Spatial association of PD-1+ tumor infiltrating lymphocytes (TILs) and PD-L1+ cells (tumor and myeloid cells) suggests "induction" of PD-L1. Interferon-gamma production by antigen-specific PD-1+ CD8+ T cells is hypothesized to drive local intratumoral upregulation of PD-L1 on adjacent tumor and myeloid cells, leading to a "stalled Cytotoxic T Lymphocyte (CTL)" response which may be predictive of response to pembrolizumab therapy. By assessing both of the required elements, i.e. PD-L1 positive cells and PD-1+ T cells, a two-color IHC assay may be a better predictor of response than PD-L1 positivity alone.

Protocol/Amendment No.: 029-05

### Transcriptional Analyses

Messenger RNA (mRNA) expression profiling will be completed to assess expression of approximately 600 genes and attempt to define a gene set critical for clinical response to pembrolizumab. The hypothesis to be tested is that pembrolizumab responders will exhibit a "stalled CTL" response within the tumor reflected in the physical proximity between PD-1 and PD-L1 expression and the presence of an aborted (e.g., weak but discernible) interferongamma transcriptional program will be detectable by profiling analyses. Global profiling will also be pursued.

Expression of individual genes related to the immune system may also be evaluated such as immune signatures and critical cytokines (e.g., IL-10).

### **Genetic Analysis**

New data are emerging that suggest we can define certain tumor types as being 'hypermutated'. There is a potential that this hypermutated state may correlate with response to pembrolizumab therapy, and/or that the converse, 'hypomutated' state may correlate with non-response.

DNA isolated from blood or tumor tissue will be analyzed in order to identify genetic alterations and to evaluate specific genetic alterations that may correlate with clinical response to pembrolizumab. These and other additional biomarker or genomic research to identify factors important for pembrolizumab therapy (for example, HLA genotype) may also be pursued.

### 4.2.3.4 Future Biomedical Research

The Sponsor will conduct Future Biomedical Research on blood and tumor tissue specimens collected during this clinical trial. This research may include genetic analyses (DNA), gene expression profiling (RNA), proteomics, metabolomics (serum, plasma) and/or the measurement of other analytes.

Such research is for biomarker testing to address emergent questions not described elsewhere in the protocol (as part of the main trial) and will only be conducted on specimens from appropriately consented subjects. The objective of collecting specimens for Future Biomedical Research is to explore and identify biomarkers that inform the scientific understanding of diseases and/or their therapeutic treatments. For instance, exploratory pharmacogenetic (PGt) studies may be performed Pharmacokinetic/Pharmacodynamic (PK/PD) relationships are observed or adverse events are identified. Genomic markers of disease may also be investigated. Such retrospective pharmacogenetic studies will be conducted with appropriate biostatistical design and analysis and compared to PK/PD results or clinical outcomes. Any significant PGt relationships to outcome would require validation in future clinical trials. The overarching goal is to use such information to develop safer, more effective drugs/vaccines, and/or to ensure that subjects receive the correct dose of the correct drug/vaccine at the correct time. The details of this Future Biomedical Research sub-trial are presented in Section 12.2 - Collection and Management of Specimens for Future Biomedical Research. Additional informational

MK-3475-029-05 Final Protocol 7-Nov-2017

Protocol/Amendment No.: 029-05

material for institutional review boards/ethics committees (IRBs/ERCs) and investigational site staff is provided in Section 12.3.

### 5.0 METHODOLOGY

#### 5.1 **Entry Criteria**

#### Diagnosis/Condition for Entry into the Trial 5.1.1

Male/Female subjects with advanced MEL (Part 1A, Part 1B and Part 1C) or RCC (Part 1A only) of at least 18 years of age will be enrolled in this trial.

# 5.1.2 Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

- 1. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent/assent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
- 2. Be  $\geq$  18 years of age on day of signing informed consent.
- 3. Have histologically or cytologically confirmed diagnosis of cancer that is recurrent, metastatic, or persistent and meet the following corresponding requirements for the cohort of the study they will enroll into.
  - a. MEL: histologically confirmed diagnosis of unresectable stage III or metastatic MEL not amenable to local therapy (Part 1A, Part 1B, and Part 1C).
    - i. Subject may not have a diagnosis of uveal or ocular MEL.
  - b. RCC: histologically confirmed diagnosis of advanced/unresectable or metastatic RCC with predominantly clear cell elements (Part 1A only).
- 4. MEL subjects may have received any number of prior lines of therapy for metastatic disease for Part 1A and 1B. RCC subjects must have received ≥1 prior line of therapy for metastatic disease

Note for Part 1C: Subjects must have previously untreated stage III-IV advanced or metastatic MEL.

Note for Part 1C: Prior adjuvant or neoadjuvant therapy is allowed as long as that therapy did not include compounds targeting PD-1, PD-L1, BRAF or MEK. Also, subjects who received prior adjuvant or neoadjuvant therapy may only participate in Part 1C if they did not discontinue therapy due to a DRAE and all related AEs have either returned to baseline or stabilized (e.g., endocrinopathies). Prior adjuvant or neoadjuvant therapy with anti-CTLA-4 will only be permitted if relapse did not occur during treatment or within 6 months of treatment discontinuation.

Protocol/Amendment No.: 029-05

5. Have measurable disease based on RECIST 1.1. Cutaneous lesions and other superficial lesions that are detectable only by physical examination are not considered measurable lesions for the purposes of this protocol, but may be considered as nontarget lesions. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

6. Must provide a tumor sample (archival or newly obtained biopsy) that is adequate for determination of PD-L1 status by IHC at a central pathology laboratory prior to enrollment. Subjects must submit the tumor sample during screening. Subjects will be eligible to participate regardless of the level of PD-L1 expression. Subjects who do not submit a sample adequate for PD-L1 determination will not be enrolled.

> Note for Part 1C: Adequacy of the tumor sample for determination of PD-L1 status by IHC at a central pathology laboratory prior to enrollment is not required.

Note: A fine needle aspirate, frozen sample, plastic embedded sample, bone, bone marrow, cell block, clot, or cytologic specimen will not be acceptable.

Subjects with an inadequate archival sample may obtain a new biopsy and subjects with non-acceptable newly obtained biopsy may undergo re-biopsy at the discretion of the investigator. Additional biopsy sample submission is encouraged but not mandatory for Part 1C when the sample is inadequate for PD-L1 testing.

- 7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
- 8. Demonstrate adequate organ function as defined in Table 3. All screening labs should be performed within 10 days of treatment initiation.

Protocol/Amendment No.: 029-05

Table 3 Adequate Organ Function Laboratory Values

| System | Laboratory Value |
|---|---|
| Hematological | • |
| Absolute neutrophil count (ANC) | $\geq 1500/\mu L$ |
| Platelets | $\geq 100~000/\mu L$ |
| Hemoglobin | $\geq$ 9.0 g/dL or $\geq$ 5.6 mmol/L <sup>a</sup> |
| Renal | |
| Creatinine <b>OR</b> | ≤1.5 × ULN <u><b>OR</b></u> |
| Measured or calculated <sup>b</sup> creatinine clearance | ≥30 mL/min for subject with creatinine levels |
| (GFR can also be used in place of creatinine or | >1.5 × institutional ULN |
| CrCl) | |
| Hepatic | |
| Total bilirubin | ≤1.5 ×ULN OR direct bilirubin ≤ULN for |
| | subjects with total bilirubin levels |
| | $>1.5 \times ULN$ (or $< 3x$ ULN in subjects with |
| | Gilbert's syndrome) |
| AST (SGOT) and ALT (SGPT) | $\leq$ 2.5 × ULN ( $\leq$ 5 × ULN for subjects with |
| | liver metastases) |
| Albumin | ≥3.0 g/dL |
| Coagulation | |
| International normalized ratio (INR) <b>OR</b> | ≤1.5 × ULN unless subject is receiving |
| prothrombin time (PT) | anticoagulant therapy as long as PT or aPTT |
| Activated partial thromboplastin time (aPTT) | is within therapeutic range of intended use of |
| | anticoagulants |

ALT (SGPT) = alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT) = aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR = glomerular filtration rate; ULN = upper limit of normal

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

- 9. Have resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia) for Part 1 A and B (Note: This sentence does not apply to Part 1C subjects as they are not permitted to have had prior chemotherapy). If subject received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
- 10. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
- 11. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the trial through 120 days after the last dose of trial drug.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

<sup>&</sup>lt;sup>a</sup> Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

<sup>&</sup>lt;sup>b</sup> Creatinine clearance (CrCl) should be calculated per institutional standard.

**Protocol/Amendment No.:** 029-05

12. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, starting with the first dose of trial therapy through 120 days after the last dose of trial therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

# 5.1.3 Subject Exclusion Criteria

07W8HB

The subject must be excluded from participating in the trial if the subject:

- 1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (ie, CTLA-4, OX-40, CD137) or has previously participated in a pembrolizumab clinical trial.
- 2. Has received prior anti-cancer therapy, monoclonal antibody, chemotherapy, or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer) before first dose of trial drug or not recovered (≤ Grade 1 or at baseline) from AEs due to previously administered agents. Exception to this rule would be use of denosumab, which is not excluded.

Note: Subjects with  $\leq$  Grade 2 neuropathy are an exception and may qualify for the trial.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting trial treatment.

Note for Part 1C: Prior chemotherapy or targeted small molecule therapy (including BRAF and MEK inhibitors) for the treatment of Stage III unresectable/Stage IV melanoma are not allowed prior to study treatment.

- 3. Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study Day 1.
- 4. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial drug.
- 5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
- 6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.

Note for Part 1C: Baseline MRI brain scan will be conducted for all subjects.

Protocol/Amendment No.: 029-05

7. Has severe hypersensitivity (≥Grade 3) to any pembrolizumab excipients (excipients are listed in the pembrolizumab IB).

- 8. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
- 9. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
- 10. Has an active infection requiring systemic therapy.
- 11. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
- 12. Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected). Note: Without known history, testing needs to be performed to determine eligibility. Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care.
- 13. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
- 14. Has received any prior therapy with IFN- $\alpha$  (in neoadjuvant, adjuvant or metastatic settings). Note: This criterion only applies to Part 1A.
- 15. Has severe cardiovascular disease, i.e. arrhythmias, requiring chronic treatment, congestive heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease.
- 16. Has hepatic decompensation (Child-Pugh score > 6 [class B and C]).
- 17. Has uncontrolled thyroid dysfunction.
- 18. Has uncontrolled diabetes mellitus.
- 19. Has received a live vaccine within 30 days prior to the first dose of trial drug. Examples of live vaccines include, but are not limited to, the following: measles. mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist<sup>®</sup>) are live attenuated vaccines and are not allowed.
- 20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 21. Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.

Protocol/Amendment No.: 029-05

Is or has an immediate family member (spouse or children) who is investigational site or sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject.

### 5.2 **Trial Treatment(s)**

The treatment(s) to be used in this trial are outlined below in Table 4. The dosing schedules for each doublet combinations are outlined in Section 6 - Trial Flow Chart.

**Trial Treatments** Table 4

| | | | Route of | |
|---|---|---|---|---|
| Drug | Dose/Potency | Dose Frequency | Administration | Use |
| pembrolizumab | 200 mg | q3w | IV infusion | Experimental |
| pembrolizumab | 2 mg/kg | q3w | IV infusion | Experimental |
| PEG-IFN | 0.5 μg/kg | Weekly | SC | Experimental |
| PEG-IFN | 1 μg/kg | Weekly | SC | Experimental |
| PEG-IFN | 2 μg/kg | Weekly | SC | Experimental |
| PEG-IFN | 3 μg/kg | Weekly | SC | Experimental |
| IPI | 1 mg/kg | q3w | IV infusion | Experimental |
| IPI | 50 mg | q6w | IV infusion | Experimental |
| IPI | 100 mg | q12w | IV infusion | Experimental |

Trial treatment for Cycle 1 should begin within 7 days of randomization.

All supplies indicated in Table 4 above will be provided centrally by the Sponsor or locally by the trial site, subsidiary or designee, depending on local country operational or regulatory requirements.

For any commercially available product that is provided by the trial site, subsidiary or designee every attempt will be made to source these supplies from a single lot/batch number. The trial site will be responsible for recording the lot number, manufacturer and expiry date of any locally purchased product.

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of trial treatments in accordance with the protocol and any applicable laws and regulations.

### 5.2.1 Dose Selection/Modification

### **5.2.1.1** Dose Selection (Preparation)

The rationale for selection of doses to be used in this trial is provided in Section 4.0.

The dose amount required to prepare study treatments (pembrolizumab, PEG-IFN, and IPI) will be based on the subject's weight in kilograms (kg). Details on the dose calculation, preparation and administration are provided in the Pharmacy Manual.

**Protocol/Amendment No.:** 029-05

With the approval of Amendment 03, subjects continuing pembrolizumab treatment on Parts 1A and 1B will switch to a fixed dose of 200mg q3w (not weight-based). The rationale for the fixed dose regimen is outlined in Section 4.2.2.

In Part 1C, subjects will receive a fixed dose of pembrolizumab 200 mg q3w. IPI will be administered as a fixed dose of 50 mg q6w (Arm 1) or 100 mg q12w (Arm 2). The rationale for fixed dose regimen is outlined in Section 4.2.2.

# **5.2.1.2** Rules for Dose Finding (Part 1A)

Dose limiting toxicities (DLTs) observed in Cycle 1 will be used to determine escalation to the next dose level. A cycle is 6 weeks. The study is using a design based on the modified TPI method [84].

The rules applied for the dose finding algorithm are as follows:

Subjects will be initially assigned between combinations (pembrolizumab + PEG-IFN or pembrolizumab + IPI). For the pembrolizumab + PEG-IFN combination, an initial cohort of 3 subjects will be enrolled. Subsequent dosing decisions will be based on the rules in Table 5. For the pembrolizumab + IPI combination, a run-in cohort of up to 18 subjects will be enrolled. If both combinations are open for enrollment, eligible subjects will be randomly assigned to a combination; otherwise, subjects will be enrolled to the combination that is open for enrollment.

## Dose Finding Rules for pembrolizumab + PEG-IFN Combination (Part 1A)

Dose finding will continue until ≤4 of 14 subjects experience a DLT at a given dose combination level. As subjects become evaluable for DLT assessment, the number of subjects who are evaluable for DLT versus the number of subjects who developed a DLT will be continuously assessed and de-escalation and re-escalation to eligible doses will occur as shown in Table 5. The decisions are generated from Ji et al. (2010) [84] using the parameters in the table with a conservative adjustment by treating 5 or more DLTs observed in any dose combinations as unacceptably toxic (denoted as DU in Table 5).

**Protocol/Amendment No.:** 029-05

Table 5 Dose Finding Rules

| | | | | Number of subjects treated at current dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| | 0 | Е | E | Е | Ε | Е | Ε | Ε | Е | Е | Е | Е | E |
| | 1 | S | S | S | Ε | Е | Ε | Ε | Е | Е | Е | Е | Ε |
| ies | 2 | D | S | S | S | S | S | S | S | Е | Е | Е | Ε |
| Number of toxicities | 3 | DU | DU | D | S | S | S | S | S | S | S | S | S |
| f to) | 4 | | DU | DU | DU | D | D | S | S | S | S | S | S |
| r of | 5 | | | DU | DU | DU | DU | DU | DU | DU | DU | DU | DU |
| mbe | 6 | | | | DU | DU | DU | DU | DU | DU | DU | DU | DU |
| S S | 7 | | | | | DU | DU | DU | DU | DU | DU | DU | DU |
| | 8 | | | | | | DU | DU | DU | DU | DU | DU | DU |
| | 9 | | | | | | | DU | DU | DU | DU | DU | DU |
| | E = Escalate to the next higher dose | | | | | | | | | | | | |
| | S = Stay at the current dose | | | | | | | | | | | | |
| | D = De-escalate to the next lower dose | | | | | | | | | | | | |
| | DU = The current dose is unacceptably toxic | | | | | | | | | | | | |
| | Target DLT rate = 30% | | | | | | | | | | | | |
| | Epsi | lon1=l | Epsilo | n2=0.0 | )5 | | | | | | | | |
| | Sour | ce: Ji | et al. ( | (2010) | [84] | | | | | | | | |

It is conceptually acceptable to de-escalate to an intermediate, not pre-defined and not previously-studied dose, if evaluation of toxicity at such a dose is desired in lieu of deescalating to a lower dose. If this approach is taken, 3 new subjects should be enrolled at the new intermediate dose, and the aforementioned rules should be used to determine further enrollment at this dose level.

The maximum number of subjects who are enrolled at a certain dose but are not yet fully evaluable for DLT assessment may not exceed the number of remaining subjects who are at risk of developing a DLT before the dose would be considered unacceptably toxic (denoted as DU in Table 5). For example, if 0/3 subjects have experienced a DLT at a given dose level, no more than an additional 5 subjects should be enrolled at this dose level until additional DLT data are available. This is because this dose level would be considered unacceptably toxic if all 5 of the additional subjects experience a DLT (i.e., 5/8 subjects with DLT in Table 5). An exception to the rule above is that a minimum of 3 subjects must be enrolled upon each dose decision.

If enrollment expands to 14 subjects for a dose level and ≤4 of the 14 subjects develop a DLT, then the dose finding is expected to stop. However, additional dose expansion to 14 subjects at a lower dose combination may be considered at the discretion of the Sponsor in consultation with the study investigators even if enrollment has expanded at a higher dose combination with ≤4 of the 14 subjects experiencing a DLT. If enrollment expands to 14 subjects for a dose level and >4/14 subjects develop a DLT, then the next lower dose may be expanded to further explore the dose-response relationship. Note that while 30% has been the target toxicity rate used to generate the guidelines in Table 5, the observed rate of

Protocol/Amendment No.: 029-05

subjects with DLT at the MTD will always be below 30% (i.e.,  $\leq 4/14$ ) due to the conservative adjustment by treating 5 or more DLTs observed in any dose combinations as unacceptably toxic.

## Safety Run-in/Dose Finding Rules for pembrolizumab + IPI Combination (Part 1A)

If  $\leq 6$  DLTs are observed in the 18 subjects enrolled in DL1 (Part 1A), this dose will be considered tolerable. If > 6 DLTs are observed in the 18 subjects enrolled, this dose level (DL1) will be proven not tolerable, and the combination with IPI will not be further developed.

If DL1 is considered tolerable, at least 90 and up to additional 150 MEL subjects will be enrolled in the expansion cohort (Part 1B) at DL1 for further evaluation of safety and tolerability.

# **5.2.1.2.1 Definition of Dose-Limiting Toxicities**

All toxicities will be graded using NCI CTCAE Version 4.0 (Appendix 12.5). Dose-limiting hematologic and non-hematologic toxicities will be defined differently. Dose-limiting toxicities (DLT) assessment will be based on events occurring during DLT assessment period, which is defined as the Cycle 1. The DLT portion of the study applies to Part 1A only. Dose-limiting toxicities include all adverse experiences that are clearly not related to disease progression or intercurrent illness if judged by the investigator to be possibly, probably or definitely related to study treatments.

# Hematological DLTs

- 1. Any Grade 3 or higher hematologic toxicity with the exception of
  - Grade 3 neutropenia
  - Grade 3 anemia

### Non-Hematological DLTs

- 1. Grade 4 non-hematologic toxicity (not laboratory).
- 2. Grade 3 non-hematologic toxicity (not laboratory) lasting >3 days despite optimal supportive care with the exception of:
  - Hypersensitivity/infusion reactions lasting ≤2 days.
- 3. Any Grade 3 or higher non-hematologic laboratory value if:
  - Medical intervention is required to treat the subject, or
  - The abnormality leads to hospitalization, or
  - The abnormality persists for >1 week

**Protocol/Amendment No.:** 029-05

4. Febrile neutropenia Grade 3 or Grade 4:

Grade 3 is defined as ANC <1000/mm<sup>3</sup> with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of ≥38 degrees C (100.4 degrees F) for more than one hour

- Grade 4 is defined as ANC <1000/mm<sup>3</sup> with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of ≥38 degrees C (100.4 degrees F) for more than one hour, with life-threatening consequences and urgent intervention indicated
- 5. Thrombocytopenia <25,000/mm<sup>3</sup> if associated with:
  - A bleeding event which does not result in hemodynamic instability but requires an elective platelet transfusion, or
  - A life-threatening bleeding event which results in urgent intervention and admission to an Intensive Care Unit.
- 6. Grade 5 toxicity (i.e., death)
- 7. Delay in the scheduled administration of any component of therapy (IPI, PEG-IFN, pembrolizumab) of >14 days
- 8. A delay of >14 days due to drug-related toxicity in initiating Cycle 2
- 9. Unable to complete at least 80% of any of the three treatments during the first course of therapy due to treatment-related toxicity (even if not meeting above DLT criteria)

## 5.2.1.2.2 Replacement of Subjects in DLT Period (Part 1A)

Replacement of subjects in DLT Period applies to Part 1A only. In order to determine safety, all subjects selected must meet the criteria for evaluability for Cycle 1. Subjects are considered non-evaluable and will be replaced if:

- they are randomized but not treated.
- they discontinue from the trial prior to completing all safety evaluations due to reasons other than DRAEs,
- they received <90% of the total pembrolizumab infusion in Cycle 1 (e.g., because the infusion had to be discontinued due to an infusion reaction) and did not experience a drug-related event.
- they received <80% of PEG-IFN or IPI intended for the trial during first Cycle 1 and did not experience a drug-related event.

Non-evaluable subjects will not be counted toward the cohort total for DLT evaluation. Subjects who experience a DLT in Cycle 1 should be discontinued from the trial. However, if it has been determined that the subject is deriving clinical benefit from the study therapy, the subject may be allowed to continue at a lower dose.

**Protocol/Amendment No.:** 029-05

### **5.2.1.3** Dose Modification (Escalation/Titration/Other)

AE Management Guidelines, including dose modification algorithms, are provided in this section for subjects treated with:

- Treatment Group A: pembrolizumab + PEG-IFN (Part 1A)
- Treatment Group B: pembrolizumab + IPI (Part 1A, 1B and 1C)

Toxicities common to PEG-IFN, IPI, and pembrolizumab include, but are not limited to rash, endocrinopathy, hepatotoxicity, diarrhea, and pneumonitis. Therefore, it is possible that these and/or other toxicities may be exacerbated when pembrolizumab is given in combination with either PEG-IFN or IPI.

The dose levels for the doublets for this trial are provided in Table 1 and Table 2.

All AEs are to be graded according to NCI CTCAE v4 (http://ctep.cancer.gov). All dose modifications and the reason for the dose modification must be documented in the eCRF.

If possible, the investigator may attribute each toxicity event to pembrolizumab, PEG-IFN, or IPI alone such that a stepwise dose reduction or increase in dosing schedule, upon resolution of the event to baseline, can be made according to Table 6, Table 8, Table 9, and Table 10.

Subjects requiring an increase in dosing schedule due to toxicity may resume pembrolizumab upon resolution of toxicity to Grade 0-1 or baseline. This dose would be considered Day 1 of the next cycle and should be in alignment with the new schedule.

For example: A subject is CURRENTLY on Cycle 3 of a pembrolizumab q3w schedule. Subject has an AE on D22 resulting in increase of dosing schedule of pembrolizumab and resolution of AE is on C3D36, drug administration should resume on D37 (now called C4D1).

Permanent discontinuation of PEG-IFN but not pembrolizumab is appropriate if in the opinion of the investigator and the Sponsor, the toxicity is clearly related to PEG-IFN. Pembrolizumab treatment may resume upon resolution of toxicity to Grade 0-1 or baseline. If in the opinion of the Investigator and the Sponsor the toxicity is related to the combination of 2 agents, both drugs should be modified according to the recommended dose modifications.

Subjects who experience an unacceptable toxicity that is attributed to IPI in the opinion of the investigator and the Sponsor, may permanently discontinue IPI, but may continue with pembrolizumab, upon resolution of toxicity to Grade 0-1 or baseline, until unacceptable toxicity or progression. Subjects who discontinue pembrolizumab due to untoward toxicities may not continue on the trial receiving only PEG-IFN or IPI.

Study treatments will be withheld for drug-related  $\geq$  Grade 3 hematologic toxicities (excluding Grade 3 neutropenia and anemia),  $\geq$  Grade 3 non-hematologic toxicity, including laboratory abnormalities; and severe or life-threatening AEs as per Table 6 and Table 8. This will also apply to subjects included in Part 1C receiving IPI + pembrolizumab combination.

**Protocol/Amendment No.:** 029-05

In Part 1C, isolated Grade 4 amylase or lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis and decrease to < Grade 4 within 7 days ±3 days of onset will not require treatment discontinuation. If not resolved to < Grade 4 within this window, trial treatment may continue with Sponsor consultation. Exceptions for restarting treatment according to the Dose Modification and Supportive Care Guidelines per Table 9 and Table 10 should be followed.

For subjects who experience a recurrence of the same AE(s) at the same grade or greater with rechallenge of study treatment(s), a consultation between the Sponsor and the investigator should occur to determine whether the subject should continue on the trial. However, for a subject who experiences a recurrence of the same SAE at the same grade or greater with rechallenge, the subject must discontinue trial treatment.

Investigators should refer to the appropriate IB/label for PEG-IFN, pembrolizumab, and IPI for additional information regarding the background of each drug and the management of other AEs or potential safety-related issues. Dosing interruptions are permitted in the case of medical/surgical events or logistical reasons not related to trial therapy (e.g., elective surgery, unrelated medical events, subject vacation, and/or holidays). Subjects should be placed back on trial therapy within 3 weeks of the scheduled interruption, unless otherwise discussed with the Sponsor. The reason for interruption should be documented in the subject's trial record.

**Protocol/Amendment No.:** 029-05

# 5.2.1.3.1 Dose Modification Guidelines for pembrolizumab + PEG-IFN or pembrolizumab + IPI Combination Therapy

# 5.2.1.3.1.1 Dose Modification Guidelines for Treatment Group A (Part 1A Only): pembrolizumab + PEG-IFN

Table 6 Dose Modification Guidelines for DRAEs for pembrolizumab + PEG-IFN

| Toxicity | Grade | Cycle<br>Number | Hold<br>Treatment<br>(Y/N) | Timing for restarting treatment | Dose/Schedule for restarting treatment | Discontinue Subject (after<br>consultation with<br>Sponsor) |
|---|---|---|---|---|---|---|
| Hematological Toxicity | Any | C1 | | | Please refer to Section 5.2.1.2.1 | |
| | 1, 2 | | No | N/A | N/A | N/A |
| | 3 Excludes Grade 3 neutropenia, and anemia | C2 and<br>Beyond | Yes | Toxicity<br>resolves to<br>Grade 0-1 or<br>baseline | Subject is dosed at DL1-DL3: May decrease PEG-IFN dose to next dose level below for each occurrence Subject is dosed at DL(-1): May discontinue PEG-IFN and increase dosing interval of pembrolizumab by 1 week° for each occurrence | Toxicity does not resolve within 12 weeks of last infusion Permanent discontinuation should be considered for any severe or life- |
| | 4 | | Yes | Toxicity<br>resolves to<br>Grade 0-1 or<br>baseline and<br>after<br>Sponsor<br>consultation | Subject is dosed at DL1-DL3: May decrease PEG-IFN dose to next dose level below Subject is dosed at DL(-1): May discontinue PEG-IFN and increase dosing interval of pembrolizumab by 1 week° | threatening event |

**Protocol/Amendment No.:** 029-05

| | | Cycle<br>Number | Hold<br>Treatment | Timing for restarting | | Discontinue Subject (after consultation with |
|---|---|---|---|---|---|---|
| Toxicity | Grade | | (Y/N) | treatment | Dose/Schedule for restarting treatment | Sponsor) |
| Non-hematological | Any | C1 | | | Please refer to Section 5.2.1.2.1. | |
| Toxicity | 1 | | No | N/A | N/A | N/A |
| Note: Exception to be treated similar to Grade 1 toxicity Grade 2 alopecia Grade 2 fatigue | 2 | | Consider withholding for persistent symptoms. | Toxicity<br>resolves to<br>Grade 0-1 or<br>baseline | Clinical AE resolves within 4 weeks: Same dose and schedule (reference Section 5.6.1 for recommendations regarding pneumonitis) Clinical AE does not resolve within 4 weeks Subject is dosed at DL1-DL3: May decrease | Toxicity does not resolve within 12 weeks of last infusion |
| PEG-IFN should be permanently discontinued if subject experiences Grade 3 liver toxicity. | | C2 and<br>Beyond | Ocular, Liver<br>and GI<br>toxicity, hold<br>both | | PEG-IFN dose to next lower dose level for each occurrence Subject is dosed at DL(-1): May discontinue PEG-IFN and increase dosing interval of pembrolizumab by 1 week° | |
| For additional information regarding irAEs, reference Section 5.6.1. | 3 | | Yes | Toxicity<br>resolves to<br>Grade 0-1 or<br>baseline | Subject is dosed at DL1-DL3:May decrease PEG-IFN dose to next dose level below Subject is dosed at DL(-1): May discontinue PEG-IFN and increase dosing interval of pembrolizumab by 1 week° | Toxicity does not resolve within 12 weeks of last infusion Permanent discontinuation should be considered for any severe or lifethreatening event |
| | 4 | | NA | NA | NA | Permanently discontinued |

<sup>°</sup> Subject may resume pembrolizumab upon resolution of toxicity to baseline. This dose would be considered Day 1 of the next cycle and should be in alignment with the new schedule. For example: A subject is CURRENLTY on Cycle 3 of a pembrolizumab q3w schedule. Subject has an AE on D22 resulting in increase of dosing schedule of pembrolizumab and resolution of AE is on C3D36, drug administration should resume on D37 (now called C4D1).

Protocol/Amendment No.: 029-05

For Part 1A, in an individual subject, following a reduction in the dose of pembrolizumab and PEG-IFN a subsequent increase in the dose will not be permitted.

### 5.2.1.3.1.2 Dose Modification Guidelines for PEG-IFN

Follow criteria listed in Table 6 for withholding study drug and dose modification for pembrolizumab + PEG-IFN. In addition,

- withhold PEG-IFN dose for the following:
  - > Grade 3 or higher thrombocytopenia
  - > Grade 3 or higher flu-like symptoms (including fever, associated tachycardia, myalgia, fatigue or chills)
  - Depressed mood/Neuropsychiatric disorder
- reduce dose of PEG-IFN to lower dose level if CrCl decreases below 50 mL/min.

Please refer to criteria for PEG-IFN dose modification, as shown in Table 7.

Table 7 Recommended Dose Reduction for PEG-IFN

| Dose Level | Dosage and Schedule |
|---|---|
| PEG-IFN Treatment at DL3 | SC 3 µg/kg/weekly |
| Dose Modification #1 | SC 2 μg/kg/weekly |
| Dose Modification #2 | SC 1 µg/kg/weekly |
| Dose Modification #3 | SC 0.5 µg/kg/weekly |
| | Permanently discontinue if unable to tolerate |
| | 0.5 μg/kg/weekly |

### 5.2.1.3.1.2.1 Dose Modification for Management of Depression

Subjects who develop mild depression during the trial may continue their study medication and should be monitored weekly (by visit or by phone) for 4 to 8 weeks. If the subject's status is stable at that time, the subject may resume the normal visit schedule with instructions to call the study center immediately if the subject feels that the depression has worsened. If the subject's condition worsens, see instructions for moderate and/or severe depression below.

Subjects who develop moderate depression during the trial should have their dose of PEG-IFN reduced (Table 7) at the discretion of the investigator. Subjects should be monitored weekly (by visit or phone for 4 to 8 weeks, depending on the subjects' status) to assure that their status is stable. These subjects may remain on reduced PEG-IFN dosing if the condition is considered stable and does not interfere with the subject's normal activities. Other clinical management intervention may be instituted as necessary. Subjects will be instructed to call the study center immediately if they feel their depression has worsened.

If the subject's condition worsens, the subject should immediately discontinue PEG-IFN, and a physician should make a priority assessment of the severity of the subject's condition. Appropriate therapeutic measures should be instituted, and the subject should be followed

MK-3475-029-05 Final Protocol

**Protocol/Amendment No.:** 029-05

weekly or biweekly (depending on the physician's clinical judgment) by visit or by phone until the subject's status has returned to baseline conditions.

## 5.2.1.3.1.2.2 Interruption or Discontinuation of PEG-IFN

Follow criteria for subject discontinuation listed in Table 6.

In addition, treatment with PEG-IFN should be permanently discontinued for any of the following reasons:

- The subject experiences new onset of ventricular arrhythmia or cardiovascular decompensation.
- The subject develops severe depression (≥ Grade 3).
- The subject experiences a persistent or worsening severe (≥ Grade 3) neuropsychiatric disorder.
- The subject experiences new or worsening retinopathy.
- The subject experiences >Grade 3 liver toxicity (AST, ALT or bilirubin) or hepatic decompensation (Child-Pugh score > 6 [class B and C]).
- The subject develops hypothyroidism, hyperthyroidism or diabetes mellitus that cannot be effectively managed.
- The subject experiences drug-related ≥ Grade 3 fever, flu-like symptoms, fatigue, or chills
- The subject experiences drug-related ≥ Grade 3 injection reactions at site of SC administration.
- The subject is unable to tolerate PEG-IFN at 0.5 µg/kg/weekly dose.

All subjects enrolled in the pembrolizumab + PEG-IFN treatment group should have a baseline ophthalmologic exam including visual acuity, visual field and color discrimination by an ophthalmologist.

Any subject complaining of ocular symptoms, including loss of visual acuity or visual field must have a prompt and complete ophthalmologic examination. In addition, because these ocular events may occur in conjunction with other disease states, periodic visual examinations during the trial are recommended, per standard of care, in subjects with disorders that may be associated with retinopathy, such as diabetes mellitus or hypertension.

If a subject's study treatment has been interrupted for more than 4 weeks for PEG-IFN and/or pembrolizumab have been withheld, the investigator must contact the Sponsor to review the subject's condition in order to resume the treatment.

Subjects being treated on combination therapy with pembrolizumab + PEG-IFN who require discontinuation of PEG-IFN for toxicity may continue treatment with pembrolizumab. The reason for discontinuation must be recorded. For subsequent management of toxicities on pembrolizumab, see Section 5.2.1.3.3.

**Protocol/Amendment No.:** 029-05

# 5.2.1.3.2 Dose Modification Guidelines for Treatment Group B: pembrolizumab + IPI

Table 8 Dose Modification Guidelines for DRAEs for pembrolizumab + IPI (Part 1A and 1B)

| Toxicity | Grade | Cycle<br>Number | Hold Treatment<br>(Y/N) | Timing for restarting treatment | Dose/Schedule for restarting treatment | Discontinue Subject (after consultation with Sponsor) |
|---|---|---|---|---|---|---|
| Any | Any | C1 | (=/=/) | *************************************** | Please refer to Section 5.2.1.2.1. | |
| | 1, 2 | C2 and<br>Beyond | No | N/A | N/A | N/A |
| | 3 Excludes Grade 3 neutropenia, and anemia | C2 | Yes | Yes $ \begin{array}{c} & Clinical \ AE \ resolves \ within \ 4^{\S} \ weeks: \ May \\ decrease \ dose \ of \ IPI \ to \ 0.3 \ mg/kg \ for \ first \\ occurrence. \ Any \ subsequent \ occurrences, \\ discontinue \ IPI \\ Clinical \ AE \ does \ not \ resolve \ within \ 4^{\S} \ weeks: \\ Discontinue \ IPI \\ \end{array} $ | | Toxicity does not resolve within 12 weeks of last infusion Permanent discontinuation should be considered for any severe or life-threatening event |
| Hematological<br>Toxicity | | C3° and beyond | Please refer to <b>Tal</b> | or DRAEs for pembrolizumab | | |
| | 4 | C2 | Yes | Toxicity resolves to Grade 0-1 or baseline and after Sponsor consultation | Clinical AE resolves within 4 <sup>§</sup> weeks: May decrease dose of IPI to 0.3 mg/kg for first occurrence. Any subsequent occurrences, discontinue IPI Clinical AE does not resolve within 4 <sup>§</sup> weeks: Discontinue IPI | Toxicity does not resolve within 12 weeks of last infusion Permanent discontinuation should be considered for any severe or life-threatening event |
| | 4 | C3° and beyond | Please refer to <b>Tal</b> | Please refer to Table 9 and Table 10 Dose Modification and Supportive Care Guidelines for DRAEs for pembrolizumab monotherapy and Part 1C | | |

Protocol/Amendment No.: 029-05

| Toxicity | Grade | Cycle<br>Number | Hold Treatment<br>(Y/N) | Timing for restarting treatment | Dose/Schedule for restarting treatment | Discontinue Subject (after consultation with Sponsor) |
|---|---|---|---|---|---|---|
| | 1 | C 2 and beyond | No | N/A | N/A | N/A |
| Non-hematological<br>Toxicity Note: Exception to<br>be treated similar | 2 | C2 | Consider withholding for persistent symptoms. For Grade 2 Ocular, Liver and GI toxicity, hold both drugs | Toxicity<br>resolves to<br>Grade 0-1 or<br>baseline | Clinical AE resolves within 4 <sup>§</sup> weeks: May resume treatment at same schedule (reference Section 5.6.1 for recommendations regarding pneumonitis) Clinical AE does not resolve within 4 <sup>§</sup> weeks: May decrease dose of IPI to 0.3 mg/kg for first occurrence. Any subsequent occurrences, discontinue IPI | Toxicity does not resolve within 12 weeks of last infusion |
| to Grade 1 toxicity: Grade 2 alopecia | 2 | C3° and beyond | Please refer to Table 9 and Table 10 Dose Modification and Supportive Care Guidelines for DRAEs for pembrolizumab monotherapy and Part 1C | | | |
| • Grade 2 fatigue For additional information regarding irAEs, Toxicity related AE. Clinical AE resolve. Grade 0-1 or baseline discontinue IPI Permanently discontinue related AE. Toxicity resolves to decrease dose of IP occurrence. Any discontinue IPI | | | | Clinical AE resolves within 4 <sup>§</sup> weeks: May decrease dose of IPI to 0.3 mg/kg for first occurrence. Any subsequent occurrences, discontinue IPI Clinical AE does not resolve within 4 <sup>§</sup> weeks: | Toxicity does not resolve within 12 weeks of last infusion Permanent discontinuation should be considered for any severe or life-threatening event | |
| | 3 | C3° and beyond | Please refer to and Table 10 Dose Modification and Supportive Care Guidelines for DRAEs for pembrolizumab monotherapy and Part 1C | | | |
| | 4 | C2 and beyond | NA | NA | NA | Permanently discontinued |

<sup>°</sup>Scheduled treatment with pembrolizumab + IPI doublet is administrated for 2 cycles (12 weeks), followed by treatment with pembrolizumab single agent.

<sup>§</sup> IPI should be permanently discontinued for subject's failure to complete full treatment course of IPI within 16 weeks from administration of first dose.

Note: Subject may resume pembrolizumab upon resolution of toxicity to baseline. This dose would be considered Day 1 of the next cycle and should be in alignment with the new schedule. For example: A subject is CURRENTLY on Cycle 3 of a pembrolizumab q3w schedule. Subject has an AE on D22 resulting in increase of dosing schedule of pembrolizumab and resolution of AE is on C3D36, drug administration should resume on D37 (now called C4D1).

**Protocol/Amendment No.:** 029-05

### 5.2.1.3.2.1 Dose Modification Guidelines for IPI

Please refer to criteria for IPI dose modification included in the approved label and described above in Table 8 for Part 1A and 1B and in Table 9 and Table 10 for pembrolizumab monotherapy and Part 1C.

### **5.2.1.3.2.1.1** Interruption or Discontinuation of IPI

In Part 1B, IPI should be permanently discontinued for subjects who fail to complete the full treatment course of IPI within 16 weeks from administration of first dose.

In Part 1C, IPI should be permanently discontinued for subjects who fail to complete the full treatment course of IPI within 30 weeks from administration of first dose for the IPI 50 mg g6w dose regimen and within 60 weeks for the IPI 100 mg g12w dose regimen.

If a subject's study treatment has been interrupted for more than 2 doses of IPI (with or without pembrolizumab being withheld), the investigator must contact the Sponsor to review the subject's condition in order to resume the treatment.

Subjects being treated on combination therapy with pembrolizumab + IPI who require discontinuation of IPI due to toxicity may continue treatment with pembrolizumab. The reason for discontinuation must be recorded.

# 5.2.1.3.3 Dose Modification and Supportive Care Guidelines for DRAEs for Pembrolizumab Monotherapy and Part 1C

# Dose modification and toxicity management for immune-related AEs associated with pembrolizumab

Adverse events associated with pembrolizumab exposure may represent an immunologic etiology. These immune-related AEs (irAEs) may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than one body system simultaneously. Therefore, early recognition and initiation of treatment is critical to reduce complications. Based on existing clinical trial data, most irAEs were reversible and could be managed with interruptions of pembrolizumab, administration of corticosteroids and/or other supportive care. For suspected irAEs, ensure adequate evaluation to confirm etiology or exclude other causes. Additional procedures or tests such as bronchoscopy, endoscopy, or skin biopsy may be included as part of the evaluation. Based on the severity of irAEs, withhold or permanently discontinue pembrolizumab and administer corticosteroids. Dose modification and toxicity management guidelines for irAEs associated with pembrolizumab are provided in Table 9.

**Protocol/Amendment No.:** 029-05

Table 9 Dose Modification and Toxicity Management Guidelines for Immune-Related AEs for Pembrolizumab Monotherapy and Part 1C

### **General instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤10 mg prednisone or equivalent per day within 12 weeks.

3. For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with<br>corticosteroid and/or other<br>therapies | Monitor and follow-up |
|---|---|---|---|---|
| Pneumonitis | Grade 2 | Withhold | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | <ul> <li>Monitor subjects for signs and symptoms of pneumonitis</li> <li>Evaluate subjects with suspected</li> </ul> |
| | Grade 3 or 4, or recurrent Grade 2 | Permanently discontinue | | <ul> <li>pneumonitis with radiographic imaging and initiate corticosteroid treatment</li> <li>Add prophylactic antibiotics for opportunistic infections</li> </ul> |
| Diarrhea / Colitis | Grade 2 or 3 | Withhold | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | <ul> <li>Monitor subjects for signs and symptoms of enterocolitis (ie, diarrhea, abdominal pain, blood or mucus in stool with or without fever) and of bowel perforation (ie, peritoneal signs and ileus)</li> <li>Subjects with ≥ Grade 2 diarrhea suspecting</li> </ul> |
| | Grade 4 | Permanently discontinue | | <ul> <li>colitis should consider GI consultation and performing endoscopy to rule out colitis.</li> <li>Subjects with diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion.</li> </ul> |

**Protocol/Amendment No.:** 029-05

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with corticosteroid and/or other therapies | Monitor and follow-up |
|---|---|---|---|---|
| AST / ALT<br>elevation or<br>Increased | Grade 2 | Withhold | Administer corticosteroids (initial<br>dose of 0.5- 1 mg/kg prednisone or<br>equivalent) followed by taper | Monitor with liver function tests (consider<br>weekly or more frequently until liver<br>enzyme value returned to baseline or is |
| bilirubin <sup>a</sup> | Grade 3 or 4 | Permanently discontinue <sup>a</sup> | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | stable |
| Type 1 diabetes<br>mellitus (T1DM)<br>or<br>Hyperglycemia <sup>b</sup> | Newly onset<br>T1DM or<br>Grade 3 or 4<br>hyperglycemia<br>associated with<br>evidence of β-cell<br>failure | Withhold | <ul> <li>Initiate insulin replacement<br/>therapy for subjects with T1DM</li> <li>Administer anti-hyperglycemic in<br/>subjects with hyperglycemia</li> </ul> | Monitor subjects for hyperglycemia or other signs and symptoms of diabetes |
| Hypophysitis | Grade 2 | Withhold | Administer corticosteroids and initiate hormonal replacements as clinically indicated | <ul> <li>Monitor for signs and symptoms of<br/>hypophysitis (including hypopituitarism and<br/>adrenal insufficiency)</li> </ul> |
| | Grade 3 or 4 <sup>b</sup> | Withhold or permanently discontinue <sup>c</sup> | Chimouny murous | |
| Hyperthyroidism <sup>b</sup> | Grade 2 | Continue | Treat with non-selective beta-<br>blockers (eg, propranolol) or<br>thionamides as appropriate | Monitor for signs and symptoms of thyroid disorders |
| | Grade 3 or 4 b | Withhold or permanently discontinue c | | |
| Hypothyroidism | Grade 2-4 | Continue | Initiate thyroid replacement<br>hormones (eg, levothyroxine or<br>liothyroinine) per standard of care | Monitor for signs and symptoms of thyroid disorders |
| Nephritis and<br>Renal | Grade 2 | Withhold | Administer corticosteroids<br>(prednisone 1-2 mg/kg or | Monitor changes of renal function |
| dysfunction | Grade 3 or 4 | Permanently discontinue | equivalent) followed by taper | |

**Protocol/Amendment No.:** 029-05

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with<br>corticosteroid and/or other<br>therapies | Monitor and follow-up |
|---|---|---|---|---|
| Myocarditis | Grade 1 or 2 | Withhold | Based on severity of AE administer corticosteroids | Ensure adequate evaluation to confirm<br>etiology and/or exclude other causes |
| | Grade 3 or 4 | Permanently discontinue | | |
| All other immune-related | Intolerable/<br>persistent Grade 2 | Withhold | Based on type and severity of AE administer corticosteroids | Ensure adequate evaluation to confirm<br>etiology and/or exclude other causes |
| AEs <sup>d</sup> | Grade 3 | Withhold or<br>discontinue based<br>on the type of<br>event. Events that<br>require<br>discontinuation<br>include and not<br>limited to:<br>Guillain-Barre<br>Syndrome,<br>encephalitis | | |
| | Grade 4 or recurrent Grade 3 | Permanently discontinue | | |

AE=adverse event; ALT=alanine aminotransferase; AST= aspartate aminotransferase; CTCAE= Common Toxicity Criteria for Adverse Events; GI=gastrointestinal; irAE=immune related adverse event; IV=intravenous; T1DM=Type 1 diabetes mellitus.

### **NOTES:**

<sup>&</sup>lt;sup>a</sup> For subjects with liver metastasis who begin treatment with Grade 2 AST or ALT, if AST or ALT increases by greater than or equal to 50% relative to baseline and lasts for at least 1 week then subject should be discontinued.

b For subjects with Grade 3 or 4 immune-related endocrinopathy where withhold of pembrolizumab is required, pembrolizumab may be resumed when AE resolves to ≤ Grade 2 and is controlled with hormonal replacement therapy, or achieved metabolic control (in case of T1DM).

<sup>&</sup>lt;sup>c</sup> Withhold or permanently discontinue pembrolizumab is at the discretion of the investigator or treating physician.

d In Part 1C, isolated Grade 4 amylase or lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis and decrease to < Grade 4 within 7 days ±3 days of onset will not require treatment discontinuation. If not resolved to < Grade 4 within this window, trial treatment may continue with Sponsor consultation.

**Protocol/Amendment No.:** 029-05

# Dose modification and toxicity management of infusion-reactions related to **pembrolizumab**

Pembrolizumab may cause severe or life threatening infusion-reactions including severe hypersensitivity or anaphylaxis. Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Dose modification and toxicity management guidelines on pembrolizumab associated infusion reaction are provided in Table 10.

**Protocol/Amendment No.:** 029-05

Pembrolizumab Infusion Reaction Dose Modification and Treatment Table 10 Guidelines

| NCI CTCAE Grade | Treatment | Premedication at Subsequent Dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |
| Grade 2 Requires therapy or infusion interruption but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDs, narcotics, IV fluids); prophylactic medications indicated for ≤24 hrs | Stop Infusion. Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines NSAIDs Acetaminophen Narcotics Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. If symptoms resolve within 1 hour of stopping drug infusion, the infusion may be restarted at 50% of the original infusion rate (eg, from 100 mL/hr to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and the subject should be premedicated for the next scheduled dose. Subjects who develop Grade 2 toxicity despite adequate premedication should be permanently discontinued from further study drug treatment. | Subject may be premedicated 1.5h (± 30 minutes) prior to infusion of pembrolizumab with: Diphenhydramine 50 mg po (or equivalent dose of antihistamine); Acetaminophen 500-1000 mg po (or equivalent dose of analgesic). |
| Grades 3 or 4 Grade 3: Prolonged (ie, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for other clinical sequelae (eg, renal impairment, pulmonary infiltrates) Grade 4: Life-threatening; pressor or ventilatory support indicated | Stop Infusion. Additional appropriate medical therapy may include but is not limited to: Epinephrine** IV fluids Antihistamines NSAIDs Acetaminophen Narcotics Oxygen Pressors Corticosteroids Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. Hospitalization may be indicated. **In cases of anaphylaxis, epinephrine should be used immediately. Subject is permanently discontinued from | No subsequent dosing |

Appropriate resuscitation equipment should be available at the bedside and a physician readily available during the period of drug administration.

For further information, please refer to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE) at http://ctep.cancer.gov

**Protocol/Amendment No.:** 029-05

In case toxicity does not resolve to Grade 0-1 within 12 weeks after last infusion of pembrolizumab, trial treatments should be discontinued after consultation with the Sponsor. With investigator and Sponsor agreement, subjects with a laboratory AE still at Grade 2 after 12 weeks may continue treatment in the trial only if asymptomatic and controlled. Refer to Table 9 for exception with regard to amylase and lipase abnormalities. For information on the management of AEs, see Section 5.6.1.

### **5.2.2** Timing of Dose Administration

Trial treatment should be administered following the schedule on Section 6 and after all procedures/assessments have been completed as detailed on the Trial Flow Chart (Section 6). Unless otherwise specified, trial treatment may be administered up to 3 days, before or after the scheduled day of each cycle due to administrative reasons.

The specific time of treatment administration (e.g., time of the week for first administration; time of the day for each administration) should take into consideration PK sampling time points and study visit procedures.

All trial treatments will be administered on an outpatient basis.

The Pharmacy Manual contains specific instructions for pembrolizumab dose calculation, reconstitution, preparation of the infusion fluid, and administration. The local product labels and institutional standards for PEG-IFN and IPI should be referenced.

## **Pembrolizumab**

Pembrolizumab will be administered as a 30 minute IV infusion q3w. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min). Pembrolizumab should always be administered first when in combination with either PEG-IFN or IPI.

### **PEG-IFN**

PEG-IFN is a once-weekly SC injection that may be self-injected. Subjects should be premedicated with acetaminophen 500 to 1000 mg orally 30 minutes prior to the first dose of PEG-IFN and as needed for subsequent doses.

The first dose of trial treatment will be administered at the trial site on Day 1. Acetaminophen [500-1000 mg orally (po)] will be given in the clinic 30 minutes prior to the first dose of PEG-IFN. Subjects should be monitored for 1-2 hours after the first dose. Acetaminophen (500-650 mg po every 4-6 hours) should be continued as needed, and should not exceed 3000 mg/day.

Subsequent dosing will be performed once weekly by the subject (i.e., unsupervised at his/her home) at approximately the same time of day. Subjects may choose to take PEG-IFN with acetaminophen at bedtime to minimize common "flu-like" symptoms (including chills, fever, muscle aches, joint pain, headaches, and tiredness).

MK-3475-029-05 Final Protocol 7-Nov-2017


**Protocol/Amendment No.:** 029-05

### IPI

In Part 1B, IPI will be administered once q3w for a total of 4 doses.

In Part 1C, IPI will be administered once q6w for a maximum of 4 doses (Arm 1) and once g12w for a maximum of 4 doses (Arm 2).

IPI will be administered as a 90 minute IV infusion. Sites should make every effort to target infusion timing to be as close to 90 minutes as possible. For additional instructions regarding dosing please refer to the IPI label.

The pharmacists will prepare IPI per the instructions in the label.

### 5.2.3 Treatment after Initial Evidence of Radiologic Disease Progression

Immunotherapeutic agents such as pembrolizumab may produce antitumor effects by potentiating endogenous cancer-specific immune responses. The response patterns seen with such an approach may extend beyond the typical time course of responses seen with cytotoxic agents, and can manifest as a clinical response after an initial increase in tumor burden or even the appearance of new lesions.

In Part 1A and 1B, tumor imaging will be assessed first at week 12 (± 3 days), then every 6 weeks ( $42 \pm 3$  days) until week 30. Subsequently, tumor imaging will be performed every 12 weeks ( $84 \pm 7$  days). In Part 1C, tumor imaging will be assessed every 6 weeks ( $\pm$  3 days) until week 24. Subsequently, tumor imaging will be performed every 12 weeks ( $84 \pm 7$  days).

If radiologic imaging shows PD, tumor assessment should be repeated ≥4 weeks later in order to confirm PD with the option of continuing treatment per below while awaiting radiologic confirmation of progression. If repeat imaging shows a reduction in the tumor burden compared to the initial scan demonstrating PD, treatment may be continued as per treatment calendar. If repeat imaging confirms PD, subjects will be discontinued from study therapy (exception noted in Section 7.1.2.8). In determining whether or not the tumor burden has increased or decreased, investigators should consider all target lesions as well as non-target lesions (please refer to the Site Imaging Manual).

When feasible, subjects should not be discontinued until progression is confirmed; however, the decision to continue study treatment after the first evidence of disease progression is at the investigator's discretion based on the clinical status of the subject as described in Table 11 below. Subjects that are deemed clinically unstable or who have biopsy proven new metastatic lesions are not required to have repeat imaging for confirmation of PD.

Note: Treatment may be continued despite modified RECIST 1.1 defined progression if the subject is clinically stable and is considered to be deriving clinical benefit by the investigator. In these cases, subjects should continue to undergo imaging as outlined in the footnote in Table 11.

Protocol/Amendment No.: 029-05

### Clinical Stability is defined as:

• Absence of signs and symptoms (including worsening of laboratory values) indicating clinically significant disease progression

- No decline in ECOG performance status
- Absence of rapid progression of disease
- Absence of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention

Table 11 Imaging and Treatment after 1st Radiologic Evidence of PD

| | Clinically Stable | | Clinically Unstable | |
|---|---|---|---|---|
| | Imaging | Treatment | Imaging | Treatment |
| 1st radiologic | Repeat imaging at | May continue | Repeat imaging | Discontinue |
| evidence of PD | $\geq$ 4 weeks to | study treatment at | at $\geq$ 4 weeks to | treatment |
| | confirm PD | the investigator's | confirm PD if | |
| | | discretion while | possible | |
| | | awaiting | | |
| | | confirmatory scan | | |
| Repeat scan | No additional | Discontinue | No additional | N/A |
| confirms PD | imaging required | treatment | imaging | |
| | | (exception noted | required | |
| | | in Section 7.1.2.8) | | |
| Repeat scan | Continue | Continue study | Continue | May restart |
| shows SD, PR or | regularly | treatment at the | regularly | study treatment |
| CR | scheduled | investigator's | scheduled | if condition has |
| | imaging | discretion | imaging | improved and/or |
| | assessments, as | | assessments, as | clinically stable |
| | per the schedule | | per the | per |
| | noted at the | | schedule noted | investigator's |
| | bottom of this | | at the bottom | discretion |
| | table. | | of this table. | |

CR = complete response; irRECIST = immune-related Response Evaluation Criteria in Solid Tumors; PD = progressive disease; PFS = progression-free survival; PR = partial response; SD = stable disease.

In Parts 1A and 1B, tumor imaging will be assessed first at week 12 (± 3 days), then every 6 weeks (42 ± 3 days) until week 30. Subsequently, tumor imaging will be performed every 12 weeks ( $84 \pm 7$  days).

In Part 1C, tumor imaging will be assessed first at week 6 ( $\pm$  3 days), then every 6 weeks ( $42 \pm 3$  days) until Week 24. Subsequently, tumor imaging will be performed every 12 weeks ( $84 \pm 7$  days).

#### 5.2.4 Trial Blinding/Masking

This is an open-label trial; therefore, the Sponsor, investigator and subject will know the treatment administered

#### 5.3 **Randomization or Treatment Allocation**

Randomization will occur centrally using an interactive voice response system / integrated web response system (IVRS/IWRS). There are two Part 1A treatment arms. Subjects will be

**Protocol/Amendment No.:** 029-05

assigned randomly in a 1:1 ratio to pembrolizumab + PEG-IFN and pembrolizumab + IPI, respectively, when both dose combination treatment groups are open for enrollment.

In Part 1B, subjects with advanced MEL will be enrolled in the pembrolizumab + IPI treatment group.

In Part 1C, subjects with advanced MEL will be randomized 1:1 to the following treatment groups:

- Arm 1: pembrolizumab 200 mg q3w + IPI 50 mg q6w
- Arm 2: pembrolizumab 200 mg q3w +IPI 100 mg q12w

### 5.4 Stratification

In Part 1A and 1C, there will be no stratification prior to randomization.

## 5.5 Concomitant Medications/Vaccinations (Allowed & Prohibited)

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for any medication or vaccination specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Sponsor Clinical Director. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician. However, the decision to continue the subject on trial therapy or vaccination schedule requires the mutual agreement of the investigator, the Sponsor and the subject.

### **5.5.1** Acceptable Concomitant Medications

All treatments that the investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the eCRF including all prescription, over-the-counter (OTC) products, herbal supplements, and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date should also be included on the eCRF.

All concomitant medications received within 28 days prior to the screening visit and up to 30 days after the last dose of trial treatment should be recorded. Concomitant medications administered 30 days after the last dose of trial treatment should be recorded for SAEs and ECIs as defined in Section 7.2.

# **5.5.2** Prohibited Concomitant Medications

07W8HB

Subjects are prohibited from receiving the following therapies during the Screening and Treatment Phase (including Second Course Phase) of this trial:

- Antineoplastic systemic chemotherapy or biological therapy
- Immunotherapy not specified in this protocol

MK-3475-029-05 Final Protocol 7-Nov-2017

**Protocol/Amendment No.:** 029-05

Chemotherapy not specified in this protocol

- Investigational agents other than pembrolizumab, PEG-IFN, or IPI
- Radiation therapy

Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be allowed at the investigator's discretion.

- Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist<sup>®</sup>) are live attenuated vaccines and are not allowed.
- Systemic glucocorticoids for any purpose other than to modulate symptoms from a drug-related AE of suspected immunologic etiology. Please note that inhaled or topical steroids are allowed, and systemic steroids at doses < 10 mg/day prednisone or equivalent are allowed, as described in Section 5.6.
- Local surgery resulting from disease progression is prohibited. However, if indicated for palliative measure and after Sponsor approval, local surgery may be permitted beyond Week 12 tumor assessment.

Subjects who, in the assessment of the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the trial. Subjects may receive other medications that the investigator deems to be medically necessary.

The Exclusion Criteria describes other medications which are prohibited in this trial.

There are no prohibited therapies during the Post-Treatment follow-up Phase.

#### 5.6 **Rescue Medications & Supportive Care**

#### 5.6.1 **Supportive Care Guidelines**

Subjects should receive appropriate supportive care measures as deemed necessary by the treating investigator. Suggested supportive care measures for the management of AEs with potential immunologic etiology are outlined along with the dose modification and supportive care guidelines in Section 5.2.1.3.3 Table 9 and Table 10 (pembrolizumab monotherapy and Part 1C). Where appropriate, these guidelines include the use of oral or IV treatment with corticosteroids, as well as additional anti-inflammatory agents if symptoms do not improve with administration of corticosteroids. Note that several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased. For each disorder, attempts should be made to rule out other causes such as metastatic disease or bacterial or viral infection, which might require additional supportive care. The treatment guidelines are intended to be applied when the investigator determines the events to be related to trial treatment

Protocol/Amendment No.: 029-05

Note: If after the evaluation of the event, it is determined not to be related to trial treatment, the investigator does not need to follow the treatment guidance. Refer to Table 6 and Table 8 in Section 5.2.1.3.1 and Section 5.2.1.3.2, respectively for guidelines regarding dose modification for DRAEs (Part 1A and 1B).

It may be necessary to perform conditional procedures such as bronchoscopy, endoscopy, or skin photography as part of evaluation of the event.

## 5.6.2 Guidelines for Pembrolizumab/PEG-IFN Combination Therapy

### **5.6.2.1 PEG-IFN Dosing Considerations**

Subjects can expect to get "flu-like" symptoms when taking PEG-IFN. Subjects may choose to take PEG-IFN with acetaminophen at bedtime to minimize common "flu-like" symptoms (including chills, fever, muscle aches, joint pain, headaches, and tiredness). Subjects should maintain hydration if experiencing "flu-like" symptoms.

### **Diet/Activity/Other Considerations** 5.7

### 5.7.1 Diet

Subjects should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea, or vomiting.

## 5.7.2 Contraception

Pembrolizumab may have adverse effects on a fetus in utero. Furthermore, it is not known if pembrolizumab has transient adverse effects on the composition of sperm.

For this trial, male subjects will be considered to be of non-reproductive potential if they have azoospermia (whether due to having had a vasectomy or due to an underlying medical condition).

Female subjects will be considered of non-reproductive potential if they meet 1 of the following criteria:

- She is postmenopausal, defined as at least 12 months with no menses without an alternative medical cause. In women < 45 years of age who are not using hormonal contraception or hormonal replacement therapy, a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
- She had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening.
- She has a congenital or an acquired condition that prevents childbearing.

**Protocol/Amendment No.:** 029-05

Female and male subjects of reproductive potential must agree to avoid becoming pregnant or impregnating a partner, respectively, while receiving trial drug and for 120 days after the last dose of trial drug by complying with 1 of the following:

• Practice abstinence from heterosexual activity.

Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and European Research Councils (ERCs)/Institutional Review Boards (IRBs). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.

• Use (or have their partner use) acceptable contraception during heterosexual activity.

Acceptable methods of contraception are::

- Single method (1 of the following is acceptable):
  - o Intrauterine device (IUD)
  - Vasectomy of a female subject's male partner
  - o Contraceptive rod implanted into the skin
- Combination method (requires use of 2 of the following):
  - o Diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide)
  - o Cervical cap with spermicide (nulliparous women only)
  - o Contraceptive sponge (nulliparous women only)
  - Male condom or female condom (cannot be used together)
  - o Hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection

<sup>‡</sup>If a contraceptive method listed above is restricted by local regulations/guidelines, then it does not qualify as an acceptable method of contraception for subjects participating at sites in this country/region.

Subjects should be informed that taking the trial medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the trial. In order to participate in the trial, subjects of childbearing potential must adhere to the contraception requirement (described above) from the day of trial medication initiation (or 14 days prior to the initiation of trial medication for oral contraception) throughout the trial period up to 120 days after the last dose of trial medication. If there is any question that a subject of childbearing potential will not reliably comply with the requirements for contraception, that subject should not be entered into the trial.

Protocol/Amendment No.: 029-05

## 5.7.3 Use in Pregnancy

If a subject inadvertently becomes pregnant while on treatment with pembrolizumab, the subject will be immediately discontinued from trial treatment. The site will contact the subject at least monthly and document the subject's status until the pregnancy has been completed or terminated. The outcome of the pregnancy will be reported to the Sponsor without delay and within 24 hours if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn). The trial investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn to the Sponsor. If a male subject impregnates his female partner, the trial personnel at the site must be informed immediately and the pregnancy must be reported to the Sponsor and followed as described in Section 7.2.

# 5.7.4 Use in Nursing Women

It is unknown whether pembrolizumab is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, subjects who are breastfeeding are not eligible for enrollment.

## 5.8 Subject Withdrawal/Discontinuation Criteria

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the discretion of the investigator should any untoward effect occur. In addition, a subject may be withdrawn by the investigator or the Sponsor if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons. Specific details regarding discontinuation or withdrawal procedures; including specific details regarding withdrawal from Future Biomedical Research, are provided in Section 7.1.4 – Other Procedures.

A subject must be discontinued from the trial for any of the following reasons:

• The subject or legal representative (such as a parent or legal guardian) withdraws consent.

A subject must be discontinued from treatment (but may continue to be monitored in the trial) for any of the following reasons:

- Confirmed radiographic disease progression outlined in Section 5.2.3 (exception if the Sponsor approves treatment continuation).
- Unacceptable adverse experiences as described in Section 7.2
- Any progression or recurrence of any malignancy, or any occurrence of another malignancy that requires systemic treatment
- Intercurrent illness other than another malignancy as noted above that prevents further administration of treatment

7-Nov-2017

• Recurrent Grade 2 pneumonitis

Protocol/Amendment No.: 029-05

A confirmed positive serum pregnancy test

- Noncompliance with trial treatment or procedure requirements
- Investigator's decision to withdraw the subject
- Completed a maximum of 24 month of treatment with pembrolizumab

Note: 24 months of pembrolizumab is calculated from the date of first dose. Subjects who stop pembrolizumab after 24 months may be eligible for a maximum of 17 doses of pembrolizumab and 4 doses of IPI if they progress after stopping study treatment provided they meet the requirements detailed in Section 7.1.5.2.1 and the study remains open.

Administrative reasons

The End of Treatment and Follow-up visit procedures are listed in Section 6 (Trial Flow Chart) and Section 7.1.5 (Visit Requirements). After the end of treatment, each subject will be followed for 30 days for AE monitoring (SAEs will be collected for 90 days after the end of treatment as described in Section 7.2.3.1). Subjects who discontinue for reasons other than PD will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent or becoming lost to follow-up. After documented disease progression, each subject will be followed by telephone for OS until death, withdrawal of consent, or the end of the study, whichever occurs first.

# 5.8.1 Discontinuation of Study Treatment after CR

Discontinuation of treatment with pembrolizumab may be considered for subjects who have attained an investigator-determined confirmed CR that have been treated for at least 24 weeks with pembrolizumab and had at least two additional doses of pembrolizumab beyond the date when the initial CR was declared. Upon Sponsor consultation, subjects who stop pembrolizumab with SD or better per modified RECIST 1.1 may be eligible for retreatment with pembrolizumab + IPI or pembrolizumab monotherapy for a maximum of 17 doses of pembrolizumab and 4 doses of IPI if they progress after stopping pembrolizumab at the discretion of the investigator according to the criteria in Section 7.1.5.2.1 as long as the trial Part to which the subject was initially enrolled remains open.

In Part 1C and upon Sponsor consultation, subjects who attain an investigator-determined CR or a VGPR per modified RECIST 1.1 may consider stopping treatment with IPI after a minimum of one dose of IPI on either Arm of treatment. Subjects who then experience radiographic disease progression may be eligible for Second Course Phase. Additional details are provided in Section 7.1.5.2.1.

#### 5.9 **Subject Replacement Strategy**

Additional subjects may be enrolled in a given treatment group to ensure that the required number of evaluable subjects in each treatment group is achieved. A subject that discontinues the trial for PD or a DRAE will not be replaced and will be counted in the evaluable population of subjects for the respective treatment group. Further details are provided in Section 8.0.

Confidential 04SGNN

07W8HB
**Protocol/Amendment No.:** 029-05

#### 5.10 Beginning and End of the Trial

The overall trial begins when the first subject signs the informed consent form. Part 1A and 1B will be considered complete when all enrolled subjects are a minimum of 24 weeks post initial trial treatment administration. At this point, a database lock may occur to allow analysis of the data. Part 1C will be considered complete for publication purposes when all enrolled subjects are a minimum of 72 weeks post initial treatment administration. At this point, database lock may occur to allow analysis of the data. Any remaining subjects may continue to receive trial treatment and be seen by the investigator per usual standard of care for this subject population. In addition, the investigator will be expected to monitor for and report any SAEs, events of clinical interest, and pregnancies as detailed in Section 7.2.3.1 (SAEs). The subject is considered on study until such time that he/she meets any of the discontinuation criteria and written notification is given to the Sponsor.

## 5.11 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

The clinical trial may be terminated early if the extent (incidence and/or severity) of emerging effects/clinical endpoints is such that the risk/benefit ratio to the trial population as a whole is unacceptable. In addition, further recruitment in the trial or at (a) particular trial site(s) may be stopped due to insufficient compliance with the protocol, Good Clinical Practice (GCP) and/or other applicable regulatory requirements, procedure-related problems, or the number of discontinuations for administrative reasons is too high.

04SGNN

Protocol/Amendment No.: 029-05

## 6.0 TRIAL FLOW CHART

## 6.1 Treatment Phase

# 6.1.1 Treatment Phase: Part 1A (MEL and RCC) and Part 1B and 1C (MEL only)

# 6.1.1.1 Treatment Group A: pembrolizumab + PEG-IFN Combination Therapy (Part 1A only)

| | pembroli | zuma | b q3 | w + 1 | PEG | -IFN | Coı | nbina | tion T | hera | рy | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | Screening | | | | | Tre | atme | nt | | | | | | Post-treatmer | ıt |
| Cycle <sup>1</sup> : | | | | 1 | | | | 2 | , | | nd<br>ond | End of<br>Treatment | Safety<br>Follow-<br>Up | Follow-Up<br>Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | -28 to -1 | 1 | 8 | 15 | 22 | 29 | 36 | 1 | 22 | 1 | 22 | At Time of<br>Discon | 30 Days<br>post<br>Discon | Every 12<br>Weeks | Every 12<br>Weeks |
| Scheduling Window Days <sup>4</sup> : | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Administrative Procedures | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | |
| Informed Consent for Future Biomedical Research 6 | X | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | | | | | | | | | |
| Demographics and Medical History | X | | | | | | | | | | | | | | |
| Prior and Concomitant Medication Review | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Treatment Randomization | | X | | | | | | | | | | | | | |
| Post-treatment Discontinuation Anti-Cancer Therapy<br>Status | | | | | | | | | | | | | | x | X |
| Survival Status | | < | | | | | | | | | | | | > | X |
| Clinical Procedures/Assessments | | | | | | | | | | | | | | | |
| Full Physical Examination | X | X | | | X | | | X | | X | | X | | | |
| Ophthalmologic Examination <sup>8</sup> | | X | | | | | | | | As | clinica | lly indicated | | | |
| Directed Physical Examination | | | X | | | X | | | X | | | | linically indi | cated | |
| ECOG Performance Status | X | X | X | | X | X | | X | X | X | | X | | | |
| 12-Lead Electrocardiogram (ECG) | X | | | | | | | | 1 | As clin | nically | indicated | | | |
| Vital Signs and Weight <sup>10</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| AE Monitoring <sup>11</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | |

07W8HB 04SGNN

| | pembroli | zuma | ıb q3 | 3w + ] | PEG | -IFN | Coı | nbina | tion T | hera | рy | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | Screening | | | | | Tre | atme | nt | | | | | | Post-treatmer | ıt |
| Cycle <sup>1</sup> : | | | | 1 | | | | 2 | 2 | | and<br>ond | End of<br>Treatment | Safety<br>Follow-<br>Up | Follow-Up<br>Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | -28 to -1 | 1 | 8 | 15 | 22 | 29 | 36 | 1 | 22 | 1 | 22 | At Time of<br>Discon | 30 Days<br>post<br>Discon | Every 12<br>Weeks | Every 12<br>Weeks |
| Scheduling Window Days <sup>4</sup> : | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Laboratory Procedures/Assessments performed by | LOCAL labo | orator | y | | | | | | | | | | | | |
| Complete Blood Count (CBC) with Differential 12,13,14 | X | X | X | X | X | X | X | X | X | X | | X | | | |
| Urinalysis 12,13,14 | X | X | X | X | X | X | X | X | | X | | X | | | |
| Comprehensive Chemistry Panel 12,13,14 | X | X | X | X | X | X | X | X | | X | | X | | | |
| Lactate Dehydrogenase (LDH) <sup>12</sup> | X | | | | | | | | | | | | | | |
| T3, FT4 and TSH <sup>12,13, 14</sup> | X | | | | | | | X | | X | | X | | | |
| PT/INR and aPTT <sup>12</sup> | X | | | | | | | | | | | | | | |
| Pregnancy Test- Urine or Serum (Beta Human<br>Chorionic Gonadotropin) β-hCG <sup>15</sup> | X | | | | | | | | | | | | | | |
| Drug Dispensation, Administration, and Associated | Analyses | | | | | | | | | | | | | | |
| Pembrolizumab Administration <sup>16</sup> | Ť | X | | | X | | | X | X | X | X | | | | |
| PEG-IFN Dosing Diaries Dispensation | | X | | | | | | X | | X | | | | | |
| PEG-IFN Administration/Dispensation <sup>17</sup> | | X | X | X | X | X | X | X | X | X | X | | | | |
| PKs of Pembrolizumab <sup>18</sup> | | • | | | | | | | | | | | • | | |
| Total IgG <sup>18</sup> | | | | | | | | | | | | 7.1.3.2 | | | |
| Anti-Pembrolizumab Antibodies (ADA) <sup>18</sup> | | | | | | | | (1 | able 1 | 3 and | 1 able | 14). | | | |
| Efficacy Measurements | | | | | | | | | | | | | | | |
| Tumor Imaging 19, 20 | X | | | | | | | | | X | | | | $\mathbf{X}^2$ | |
| Digital Photography: Cutaneous Lesions <sup>21</sup> | X | | | | | | | | | As clir | nically | Indicated | | | |
| Tissue and Blood Collections and Pharmacodynami | c Assessmen | t | | | | | | | | | | | | | |
| Tumor Tissue Collection <sup>22, 23</sup> | X | | | | | | | | | X | | X | | | |
| Correlative Blood Sample Collection 24 | X | | | | | | | | | X | | X | | | |
| Blood Sample Collection for Genetics 25 | | X | | | | | | | | | | | | | |
| Blood for Future Biomedical Research 26 | | X | | | | | | | | | | | | | _ |

**Protocol/Amendment No.:** 029-05

1. Treatment cycles are 6 weeks. Imaging should always be performed as scheduled and follow calendar days, regardless of any treatment delays.

- 2. Subjects who discontinue trial treatment due to a reason other than disease progression should continue follow-up and assessment by radiologic imaging (and digital photography if applicable) every 12 weeks (± 1 week) for the first year after discontinuation, then every 6 months (± 2 weeks) for years two through five, and every 12 months (± 4 weeks) after year five. Imaging follow-up should continue until (1) the start of new anti-cancer treatment, (2) documented disease progression, (3) death, or (4) the end of the trial, whichever occurs first.
- 3. After the start of new anti-cancer treatment or documented disease progression, the subject should be contacted by telephone approximately every 12 weeks after the last contact date to assess for survival status. In certain situations, survival data may be requested more frequently than every 12 weeks as per Section 7.1.5.3.3. Updated survival status may be requested by the Sponsor at any time during the course of the study. Upon Sponsor notification, all subjects who do not/will not have a scheduled study visit or study contact during the Sponsor-defined time period will be contacted for their survival status (excluding subjects that have a death event previously recorded).
- 4. In general, the window for each visit is  $\pm 3$  days unless otherwise noted.
- 5. Written consent must be obtained prior to performing any protocol specific procedure. Results of a test performed prior to the subject signing consent as part of routine clinical management are acceptable in lieu of a screening test if performed within the specified time frame (e.g., within 28 days prior to the first dose of trial treatment). Screening number will be assigned when the study informed consent is signed.
- 6. Informed consent for future biomedical research samples must be obtained before the DNA sample. DNA sample for analysis should be obtained predose, on Day 1 (or with the next scheduled blood draw) as the last sample drawn or at a later date as soon as the informed consent is obtained.
- 7. Prior medications All concomitant medications received within 28 days prior to the screening visit and up to 30 days after the last dose of trial treatment should be recorded.
- 8. All subjects should have a baseline ophthalmologic exam including visual acuity, visual field and color discrimination by an ophthalmologist. Fundus photography should be performed in subjects with history of clinically significant retinal disease (defined as macular degeneration, retinal detachment and moderate/severe non-proliferative diabetic retinopathy and any proliferative diabetic retinopathy). Enrollment of subjects with clinically significant retinal disease will require consultation with the sponsor on risk-benefit associated to treatment with pembrolizumab + PEG-IFN. Any subject complaining of ocular symptoms, including loss of visual acuity or visual field must have a prompt and complete ophthalmologic examination. In addition, because these ocular events may occur in conjunction with other disease states, periodic visual examinations during the trial are recommended in subjects with disorders that may be associated with retinopathy, such as diabetes mellitus or hypertension. Discontinuation of PEG-IFN should be considered in subjects who develop new or worsening ophthalmological disorders.
- 9. ECG should be performed at screening and as clinically indicated thereafter. ECGs are performed locally.
- 10. Vital signs to include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.
- 11. Record all AEs occurring within 30 days after the last dose of trial treatment and all SAEs (related and unrelated to trial treatment) / ECIs occurring up until 90 days following cessation of treatment or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier. Afterwards, report only SAEs and ECIs that are related to trial treatment.
- 12. Laboratory tests for screening are to be performed within 10 days prior to the first dose of trial treatment. See Section 7.1.3 for details regarding laboratory tests.
- 13. After Cycle 1, lab samples can be collected up to 72 hours prior to the scheduled time point. Laboratory results must be known and acceptable prior to dosing. See Section 7.1.3 for details regarding laboratory tests. After Cycle 8, lab samples should be collected every two cycles on D1 (i.e.; C8 D1, C10 D1, C12 D1, etc.)
- 14. Unresolved abnormal labs that are DRAEs should be followed until resolution.
- 15. For women of reproductive potential, a urine pregnancy test should be performed within 72 hours prior to first dose of trial treatment. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test performed by the local study site laboratory will be required. Pregnancy tests (serum and/or urine tests) should be repeated if required by local guidelines.
- 16. Pembrolizumab will be administered as a 30 minute IV infusion. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min). Pembrolizumab should always be administered first when given in combination.
- 17. The first dose of PEG-IFN will be administered at the trial site at C1D1. Subsequent dosing will be performed once weekly (±1 day) by the subject (i.e., unsupervised at his/her home) at approximately the same time of day. Directions for the self-administration of SC injections of PEG-IFN can be found in the Pharmacy Manual.

**Protocol/Amendment No.:** 029-05

PK samples should be collected during; C1D1; pre- and post-dose, at C1D8 (post-dose), C1D22 (pre-dose), C2D22 (pre-dose), C4D1 (pre-dose), C7D1 (pre-dose) and every 3 cycles thereafter and at 30 days after discontinuation of pembrolizumab treatment. Total IgG should be collected simultaneous with pre-dose pembrolizumab PK sampling. ADA (simultaneous with pre-dose PK sampling, except for the C2D22): C1D1 (pre-dose), C1D22 (pre-dose), C4D1 (pre-dose), C7D1 (pre-dose) and every 3 cycles thereafter and at 30 days after discontinuation of pembrolizumab treatment Pre-dose: within 60 minutes before infusion of pembrolizumab. Post-dose: within 30 minutes after the end of infusion of pembrolizumab C1D1 and at C1D8. A detailed PK/ADA scheme is described in Section 7.1.3.2.

- 19. A scan must be performed within 28 days prior to starting treatment with pembrolizumab. Scans performed as part of routine clinical management are acceptable for use as the screening scan if they are of diagnostic quality and performed within 28 days prior to the first dose of trial treatment. Imaging timing should follow calendar days and should not be adjusted for delays in cycle starts or extension of pembrolizumab cycle frequencies. The first imaging assessment should be performed 12 weeks (± 3 days) after the first dose of trial treatment, and continue to be performed every 6 weeks (42 ± 3 days) until week 30, regardless of any treatment delays. Following week 30, tumor imaging will be performed approximately every 12 weeks (84 ± 7 days) (or as clinically indicated) while the patient remains on trial therapy. Subjects who discontinue trial treatment for a reason other than disease progression should continue to be assessed in Follow-up Phase with the first scan occurring 12 weeks (84 +/- 7 days) from the date of the last scan on study. The same imaging technique should be used in a subject throughout the trial. Local reading (investigator assessment with site radiology reading) will be used to determine eligibility and for subject management. The Sponsor will collect radiological assessments for retrospective analysis by a central vendor unless otherwise noted by the Sponsor. The processes for image collection and transmission to the central vendor are in the Site Imaging Manual.
- 20. Per the modified RECIST 1.1 used in this protocol, if imaging shows PD, the imaging assessment should be performed no sooner than 4 weeks later in order to confirm PD as described in Section 4.2.3.2.
- 21. For subject with MEL only: Qualitative digital photography should be performed at baseline and at time of scheduled tumor assessments for cutaneous lesions. Cutaneous lesions are not considered measurable for the purposes of this protocol, but may be considered to be non-target lesions for tumor assessments by investigators. Copies of digital photographs should not be submitted to the central imaging vendor unless otherwise noted by the Sponsor.
- 22. Collection of archival tumor tissue for purpose of biomarker analysis. Written subject consent is required for collection of archival tumor tissue. Tumor sample should be adequate for biomarker analyses assessment. Subjects with an inadequate archival sample may obtain a new biopsy and subjects with an inadequate newly obtained biopsy may undergo re-biopsy at the discretion of the investigator. Specific instructions for tissue collection and shipment are provided in the Laboratory Manual.
- 23. A newly obtained biopsy of a tumor lesion is desirable but not mandatory. Written subject consent is required for newly obtained biopsies. Newly obtained biopsies should be limited to readily accessible tumor lesions (e.g., skin; peripheral lymph nodes; lung, liver or internal lymph node metastases which can be readily accessed using computed tomography (CT) guidance). If performed, a tissue cylinder should be obtained that has proper size for histological examination and biomarker analysis. Specific instructions for tissue collection and shipment are provided in the Laboratory Manual.
- 24. Blood samples should be obtained prior to Cycle 1. Cycle 3, and at discontinuation.
- 25. This sample should be drawn for planned analysis of the association between genetic variants in DNA and drug response. This sample will not be collected at that site if there is either a local law or regulation prohibiting collection, or if the IRB/IEC does not approve the collection of the sample for these purposes.
- 26. If the subject signs the Future Biomedical Research consent, any leftover samples may be stored for future biomedical research.

Protocol/Amendment No.: 029-05

# 6.1.1.2 Treatment Group B: pembrolizumab + IPI Combination Therapy (Part 1A, Part 1B and Part 1C)

| | | | | | | | peml | proliz | uma | b q3 | w + I | PI C | ombi | natio | n Th | erapy | y | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | Screening | | | | | | | | | Trea | tmen | t | | | | | | | | End | Po | st-treatm | ent |
| Cycle 1: | | | | | 1 | | | 2 | ! | 3 aı | nd 4 | : | 5 | ( | 6 | 7 | | aı | 8<br>nd<br>ond | of<br>Treatment | Safety<br>Follow-<br>Up | Follow<br>-Up<br>Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | -28 to -1 | 1 | 8 | 15 | 22 | 29 | 36 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | At<br>Time<br>of<br>Discon | 30<br>Days<br>Post-<br>Discon | Every<br>12<br>Weeks | Every<br>12<br>Weeks |
| Scheduling<br>Window Days <sup>4</sup> : | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Administrative Proc | edures | | | | | | | | | | | | | | | | | | | | | | |
| Informed Consent <sup>5</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Informed Consent<br>for Future<br>Biomedical<br>Research <sup>6</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | | | | | | | |
| Demographics and<br>Medical History | X | | | | | | | | | | | | | | | | | | | | | | |
| Prior and<br>Concomitant <sup>7</sup><br>Medication Review | x | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Treatment<br>Randomization | | X | | | | | | | | | | | | | | | | | | | | | |
| Post-Treatment Discontinuation Anti-Cancer Therapy Status | | | | | | | | | | | | | | | | | | | | | | X | x |
| Survival Status | | <- | | | | | | | | | | | | | | | | | | | | > | X |

07W8HB 04SGNN

| | | | | | | | peml | oroliz | uma | ıb q3 | w + I | PI C | ombi | natio | n Th | erap | y | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | Screening | | | | | | | | | Trea | tmen | t | | | | | | | | End | Po | st-treatm | ent |
| Cycle <sup>1</sup> : | | | | | 1 | | | 2 | 2 | 3 ar | ıd 4 | , | 5 | , | 6 | 7 | , | aı | 3<br>1d<br>ond | of<br>Treatment | Safety<br>Follow-<br>Up | Follow -Up Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | -28 to -1 | 1 | 8 | 15 | 22 | 29 | 36 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | At<br>Time<br>of<br>Discon | 30<br>Days<br>Post-<br>Discon | Every<br>12<br>Weeks | Every<br>12<br>Weeks |
| Scheduling<br>Window Days <sup>4</sup> : | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Clinical Procedures | Assessments | ; | | | | | | | | | | | | | | | | | | | | | |
| Full Physical<br>Examination | X | X | | | X | | | X | | X | | X | | X | | X | | X | | X | | | |
| Directed Physical<br>Examination | | | X | X | | X | | | | | | | | | As | clinic | ally i | indica | ited | | | | |
| ECOG Performance<br>Status | X | X | X | | X | X | | X | | X | | X | | X | | X | | X | | X | | | |
| 12-Lead<br>Electrocardiogram<br>(ECG) <sup>8</sup> | x | | | | | | | | | | | | As | elinica | lly inc | licate | d | | | | | | |
| Vital Signs and<br>Weight <sup>9</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| AE Monitoring <sup>10</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Laboratory Procedu | res/Assessm | ents | perf | orme | d by I | OC | AL lab | orato | ry | | | | | | | | | | | | | | |
| CBC with<br>Differential <sup>11, 12,13</sup> | X | X | X | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | | |
| Urinalysis 11, 12,13 | X | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | | |
| Comprehensive<br>Chemistry Panel <sup>11,</sup><br>12,13 | x | X | X | X | X | X | X | X | | х | | X | | X | | X | | X | | X | | | |
| LDH <sup>11</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| T3, FT4 and TSH <sup>11,</sup> 12,13 | X | | | | | | | X | | X | | X | | X | | X | | X | | X | | | |
| PT/INR and aPTT <sup>II</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test-<br>Urine or Serum β-<br>hCG <sup>14</sup> | X | | | | | | | | | | | | | | | | | | | | | | |

| | | | | | | | peml | oroliz | zuma | b q3 | w + I | PI C | ombi | natio | n Th | erap | y | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | Screening | | | | | | | | | Trea | tmen | t | | | | | | | | End | Po | st-treatm | ent |
| Cycle 1: | | | | | 1 | | | 2 | 2 | 3 ar | nd 4 | ; | 5 | | 6 | 7 | | aı<br>Bey | | of<br>Treatment | Safety<br>Follow-<br>Up | Follow<br>-Up<br>Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | -28 to -1 | 1 | 8 | 15 | 22 | 29 | 36 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | At<br>Time<br>of<br>Discon | 30<br>Days<br>Post-<br>Discon | Every<br>12<br>Weeks | Every<br>12<br>Weeks |
| Scheduling<br>Window Days <sup>4</sup> : | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Drug Dispensation, | Administrati | on, a | ınd A | Assoc | iated . | Anal | yses | | | | | | | | | | | | | | | | |
| Pembrolizumab<br>Administration <sup>15</sup> | | X | | | X | | | X | X | X | X | X | X | X | X | X | X | X | X | | | | |
| IPI Administration<br>Part 1B <sup>16</sup> | | X | | | X | | | X | X | | | | | | | | | | | | | | |
| IPI Administration<br>Part 1C, Arm 1 <sup>16</sup> | | X | | | | | | X | | X | | | | | | | | | | | | | |
| IPI Administration<br>Part 1C, Arm 2 <sup>16</sup> | | X | | | | | | | | X <sup>17</sup> | | X | | | | X | | | | | | | |
| PKs of Pembrolizumab <sup>18a,b</sup> Total IgG <sup>18a,b</sup> PKs of IPI <sup>18a,b</sup> Anti- Pembrolizumab Antibodies <sup>18a,b</sup> | | | | | | | | | | | | | efer to<br>e 14 ar | | | | | | | | | | |
| Efficacy Measureme | nts | | | | | | | | | | | | | | | | | | | | | | |
| Tumor Imaging Part<br>1A and 1B <sup>19,20</sup> | X | | | | | | | | | X | | X | | X | | | | X <sup>20</sup> | | | | $X^2$ | |
| Tumor Imaging Part<br>1C <sup>19,21</sup> | | | | | | | | X | | X | | X | | | | X <sup>21</sup> | | X <sup>21</sup> | | | | $X^2$ | |
| Digital<br>Photography:<br>Cutaneous Lesions <sup>22</sup> | X | As Clinically Indicated | | | | | | | | | | | | | | | | | | | | | |

| | | | | | | | peml | broliz | zuma | ıb q3 | w + 1 | PI C | ombi | natio | n Th | erapy | y | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | Screening | | | | | | | | | Trea | tmen | t | | | | | | | | End | Po | st-treatm | ent |
| Cycle 1: | | | | | 1 | | | 2 | 2 | 3 ar | nd 4 | | 5 | | 6 | 7 | 7 | aı | 3<br>nd<br>ond | of<br>Treatment | Safety<br>Follow-<br>Up | Follow -Up Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | -28 to -1 | 1 | 8 | 15 | 22 | 29 | 36 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | At<br>Time<br>of<br>Discon | 30<br>Days<br>Post-<br>Discon | Every<br>12<br>Weeks | Every<br>12<br>Weeks |
| Scheduling<br>Window Days <sup>4</sup> : | ±3 | ±3 | ±3 | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Tissue and Blood Co | ollections and | l Pha | arma | cody | nami | c Ass | essme | nt | | | | | | | | | | | | | | | |
| Tumor Tissue<br>Collection <sup>23</sup> | X | | | | | | | | | X | | | | | | | | | | X | | | |
| Correlative Blood<br>Sample Collection,<br>Part 1A and 1B <sup>24</sup> | X | | | | | | | | | X | | | | | | | | | | X | | | |
| Correlative Blood<br>Sample Collection,<br>Part 1C <sup>24</sup> | X | | | | | | | | | X | | | | X | | | | X | | X | | | |
| Blood Sample<br>Collection for<br>Genetics <sup>25</sup> | | X | | | | | | | | | | | | | | | | | | | | | |
| Blood for Future<br>Biomedical<br>Research <sup>26</sup> | | X | | | | | | | | | | | | | | | | | | | | | |
| Blood for Peripheral<br>Blood Mononuclear<br>Cells (PBMC), Part<br>1C <sup>27</sup> | | X | | | X | | | | | | | | X | 27 | | | | | | X | | | |
| Blood for Serum<br>and Plasma<br>Biomarker<br>Analyses, Part 1C <sup>27</sup> | | X | | | X | | | | | | | | X | 27 | | | | | | X | | | |
| Blood for T-Cell<br>Receptor (TCR)<br>DNA, Part 1C <sup>27</sup> | | X | | | X | | | | | | | | X | 27 | | | | | | X | | | |
| Blood for<br>Circulating Tumor<br>(ctDNA), Part 1C <sup>27</sup> | | х | | | X | | | | | | | | X | 27 | | | | | | Х | | | |

**Protocol/Amendment No.:** 029-05

1. Treatment cycles are 6 weeks. Imaging should always be performed as scheduled and follow calendar days, regardless of any treatment delays.

- 2. Subjects who discontinue trial treatment due to a reason other than disease progression should continue follow-up and assessment by radiologic imaging (and digital photography if applicable) every 12 weeks (± 1 week) for the first year after discontinuation, then every 6 months (± 2 weeks) for years two through five, and every 12 months (± 4 weeks) after year five. Imaging follow-up should continue until (1) the start of new anti-cancer treatment, (2) documented disease progression, (3) death, or (4) the end of the study, whichever occurs first.
- 3. After the start of new anti-cancer treatment or documented disease progression, the subject should be contacted by telephone approximately every 12 weeks after the last contact date to assess for survival status. In certain situations, survival data may be requested more frequently than every 12 weeks as per Section 7.1.5.3.3. Updated survival status may be requested by the Sponsor at any time during the course of the study. Upon Sponsor notification, all subjects who do not/will not have a scheduled study visit or study contact during the Sponsor-defined time period will be contacted for their survival status (excluding subjects that have a death event previously recorded).
- 4. In general, the window for each visit is  $\pm 3$  days unless otherwise noted.
- 5. Written consent must be obtained prior to performing any protocol specific procedure. Results of a test performed prior to the subject signing consent as part of routine clinical management are acceptable in lieu of a screening test if performed within the specified time frame (e.g., within 28 days prior to the first dose of trial treatment). Screening number will be assigned when the study informed consent is signed.
- 6. Informed consent for future biomedical research samples must be obtained before the DNA sample. DNA sample for analysis should be obtained predose, on Day 1 (or with the next scheduled blood draw) as the last sample drawn or at a later date as soon as the informed consent is obtained.
- 7. Prior medications All concomitant medications received within 28 days prior to the screening visit and up to 30 days after the last dose of trial treatment should be recorded.
- 8. ECG should be performed at screening and as clinically indicated thereafter. ECGs are performed locally.
- 9. Vital signs to include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.
- 10. Record all AEs occurring within 30 days after the last dose of trial treatment and all SAEs (related and unrelated to trial treatment)/ECIs occurring up until 90 days following cessation of treatment or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier. Afterwards, report only SAEs and ECIs that are related to trial treatment.
- 11. Laboratory tests for screening are to be performed within 10 days prior to the first dose of trial treatment. See Section 7.1.3 for details regarding laboratory tests.
- 12. After Cycle 1, lab samples can be collected up to 72 hours prior to the scheduled time point. Laboratory results must be known and acceptable prior to dosing. See Section 7.1.3 for details regarding laboratory tests. After Cycle 8, lab samples should be collected every two cycles on D1 (i.e.; C8 D1, C10 D1, C12 D1, etc.)
- 13. Unresolved abnormal labs that are DRAEs should be followed until resolution.
- 14. For women of reproductive potential, a urine pregnancy test should be performed within 72 hours prior to first dose of trial treatment. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test performed by the local study site laboratory will be required. Pregnancy tests (serum and/or urine tests) should be repeated if required by local guidelines.
- 15. Pembrolizumab will be administered as a 30 minute IV infusion. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min). Pembrolizumab should always be administered first when given in combination.
- 16. In Part 1A and B, IPI will be administered for a total of 4 doses. In Part 1C, IPI will be administered for a maximum of 4 doses. Subjects will be administered IPI as a 90 minute IV infusion. Sites should make every effort to target infusion timing to be as close to 90 minutes as possible. For additional instructions regarding dosing please refer to the IPI label. Subjects who initially attain clinical benefit (defined as modified RECIST 1.1 confirmed PR or SD>6 mo), and experience disease progression while receiving single agent pembrolizumab will be eligible for reinduction with 4 doses of IPI q3w as long as Part 1A or 1B remains open. Those subjects should follow the assessments detailed in Cycle 2 and beyond.

**Protocol/Amendment No.:** 029-05

17. IPI will be administered only on Cycle 3 and not on Cycle 4.

- 18. For PK samples, predose: within 60 minutes before infusion of pembrolizumab. Post-dose: within 30 minutes after the end of infusion of pembrolizumab. A detailed PK/ADA scheme is described in Section 7.1.3.2.
  - a. Parts 1A and 1B: PK samples should be collected during C1D1 (pre- and post-dose), C1D8 (post-dose), C1D22 (pre-dose), C2D22 (pre-dose), C4D1 (pre-dose), C7D1 (predose) and every 3 cycles thereafter and at 30 days after discontinuation of pembrolizumab treatment Total IgG should be collected simultaneous with pre-dose pembrolizumab PK sampling, ADA (simultaneous with pre-dose PK sampling, except for C2D22): C1D1 (pre-dose), C1D22 (pre-dose), C4D1 (pre-dose), C7D1 (pre-dose) and every 3 cycles thereafter and at 30 days after discontinuation of pembrolizumab treatment.
  - b. Part 1C: PK samples will be collected during C1D1, C2D1, C3D1, C5D1, C7D1, C9D1, and every 2 cycles thereafter until treatment discontinuation. A PK sample at 30 days after discontinuation of pembrolizumab treatment is not required for Part 1C.
- 19. A scan must be performed within 28 days prior to starting treatment with pembrolizumab. Scans performed as part of routine clinical management are acceptable for use as the screening scan if they are of diagnostic quality and performed within 28 days prior to the first dose of trial treatment. Imaging timing should follow calendar days and should not be adjusted for delays in cycle starts or extension of pembrolizumab cycle frequencies. The same imaging technique should be used in a subject throughout the trial. Local reading (investigator assessment with site radiology reading) will be used to determine eligibility and for subject management. The Sponsor will collect radiological assessments for retrospective analysis by a central vendor unless otherwise noted by the Sponsor. The processes for image collection and transmission to the central vendor are in the Site Imaging Manual. Per the modified RECIST 1.1 used in this protocol, if imaging shows PD, the imaging assessment should be performed no sooner than 4 weeks later in order to confirm PD as described in Section 4.2.3.2.
- 20. In Part 1A and B, the first imaging assessment should be performed 12 weeks (± 3 days) after the first dose of trial treatment, and continue to be performed every 6 weeks (42 ± 3 days) until week 30, regardless of any treatment delays. Following week 30, tumor imaging will be performed approximately every 12 weeks (84 ± 7 days or as clinically indicated) while the subject remains on trial therapy.
- 21. In Part 1C, the first imaging assessment should be performed 6 weeks (± 3 days) after the first dose of trial treatment, and continue to be performed every 6 weeks (42 ± 3 days) until week 24, regardless of any treatment delays. Following week 24, tumor imaging will be performed approximately every 12 weeks (84 ± 7 days or as clinically indicated) while the subject remains on trial therapy. Subjects who discontinue trial treatment for a reason other than disease progression should continue to be assessed in Follow-up Phase with the first scan occurring 12 weeks (84 ± 7 days) from the date of the last scan on study. In Part 1C, a baseline brain MRI will be performed to rule out brain metastasis.
- 22. For subject with MEL only: Qualitative digital photography should be performed at baseline and at time of scheduled tumor assessments for cutaneous lesions. Cutaneous lesions are not considered measurable for the purposes of this protocol, but may be considered to be non-target lesions for tumor assessments by investigators. Copies of digital photographs should not be submitted to the central imaging vendor unless otherwise noted by the Sponsor.
- 23. A newly obtained biopsy sample of at least one tumor lesion is preferred in all subjects and is mandatory for subjects who do not have an acceptable archival tumor tissue sample for PD-L1 evaluation. PD-L1 status must be assessed during screening, and if the tumor biopsy submitted is inadequate for determination of PD-L1 status by IHC at a central pathology laboratory, the subject will not be randomized. Subjects with an inadequate archival sample may obtain a new biopsy and subjects with an inadequate newly obtained biopsy may undergo re-biopsy at the discretion of the investigator. Confirmation of the tumor tissue sample adequacy for determination of PD-L1 status by IHC at a central pathology laboratory will not be required prior to enrollment in Part 1C. Additional biopsy sample submission is encouraged but not mandatory for Part 1C when the sample is inadequate for PD-L1 testing. Additional biopsy sample approximately at C3D1 and at disease progression are highly desirable when it is feasible. Newly obtained biopsies should be limited to readily accessible tumor lesions (e.g., skin; peripheral lymph nodes; lung, liver or internal lymph node metastases which can be readily accessed using CT guidance). If performed, a tissue cylinder should be obtained that has proper size for histological examination and biomarker analysis. Study sites should use the same biopsy techniques in this study as they routinely use for a given tumor lesion/location. Written subject consent is required for collection of tumor tissue. Specific instructions for tissue collection and shipment are provided in the Laboratory Manual.

**Protocol/Amendment No.:** 029-05

24. In Part 1A and 1B blood samples should be obtained prior to Cycle 1, Cycle 3, and at discontinuation. In Part 1C blood samples should be obtained prior to Cycle 1 Day 1, at Cycle 3 Day 1, at Cycle 4 Day 1 and then every 12 weeks (cycles 6 and beyond), and at Time of Discontinuation.

- 25. This sample should be drawn for planned analysis of the association between genetic variants in DNA and drug response. This sample will not be collected at that site if there is either a local law or regulation prohibiting collection, or if the IRB/IEC does not approve the collection of the sample for these purposes.
- 26. If the subject signs the Future Biomedical Research consent, any leftover samples may be stored for future biomedical research.
- 27. In Part 1C, blood for PBMC, serum and plasma biomarker analyses, TCR DNA and circulating tumor DNA should be collected at Cycle 1 Day 1, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 6 Day 1 and at Time of Discontinuation.

Protocol/Amendment No.: 029-05

# 6.2 Second Course Phase: All Parts - All Treatment Groups (MEL and RCC)

| | For | subje | ects er | ırolle | d in p | emb | roliz | uma | b q3 | w + I | EG-I | FN or | pembro | lizumal | b q3w | + IPI: | Second Cou | rse Phase | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | | | | | SI | ECO | ND C | OU | RSE | PHA | SE: T | reatn | nent | | | | End of<br>Treatment | I | Post-treatment | |
| Cycle <sup>1</sup> : | : | 1 | 2 | 2 | : | 3 | 4 | 4 | : | 5 | | 6 | 7 | | | and<br>yond | | Safety<br>Follow-Up | Follow-Up<br>Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | At Time of<br>Discon | 30 Days<br>post<br>Discon | Every 12<br>Weeks | Every 12<br>Weeks |
| Scheduling Window Days 4: | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Administrative Procedures | | | | | | | | | | | | | | | | | | | | |
| Eligibility Criteria <sup>5</sup> | X | | X | | X | | X | | X | | X | | X | | X | | | | | |
| Concomitant Medication<br>Review <sup>6</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Post-Treatment<br>Discontinuation Anti-Cancer<br>Therapy Status | | | | | | | | | | | | | | | | | | | X | X |
| Survival Status | <- | | | | | | | | | | | | | | | | | | > | X |
| Clinical Procedures/Assessm | ents | | | | | | | | | | | | | | | | | | | |
| Full Physical Examination | X | | X | | X | | X | | X | | X | | X | | X | | X | | | |
| Directed Physical<br>Examination | | X | | | | | | | | | | | As | linicall | y indi | cated | | | | |
| ECOG Performance Status | X | X | X | | X | | X | | X | | X | | X | | X | | X | | | |
| Vital Signs and Weight <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| AE Monitoring <sup>8</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |

| | For | subje | ects ei | nrolle | d in p | emb | roliz | uma | b q3 | w + P | EG-I | FN or | pembro | lizumal | b q3w | + IPI | Second Cou | rse Phase | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Period: | | | | | SI | ECO | ND C | OU | RSE | РНА | SE: T | reatn | nent | | | | End of<br>Treatment | I | ost-treatment | |
| Cycle <sup>1</sup> : | | 1 | | 2 | | 3 | 4 | 4 | | 5 | · | 6 | 7 | | | and<br>yond | | Safety<br>Follow-Up | Follow-Up<br>Visits <sup>2</sup> | Survival<br>Follow-<br>Up <sup>3</sup> |
| Day: | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | 1 | 22 | At Time of<br>Discon | 30 Days<br>post<br>Discon | Every 12<br>Weeks | Every 12<br>Weeks |
| Scheduling Window Days 4: | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±7 | ±7 |
| Laboratory Procedures/Asse | _ | nts | | | | | | | | | | | | | | • | | | | |
| CBC with Differential <sup>9,10,11</sup> | X | | X | | X | | X | | X | | X | | X | | $X^{10}$ | | X | | | |
| Urinalysis <sup>9,10,11</sup> | X | | X | | X | | X | | X | | X | | X | | X <sup>10</sup> | | X | | | |
| Comprehensive Chemistry<br>Panel <sup>9,10,11</sup> | X | | X | | X | | X | | X | | X | | X | | X <sup>10</sup> | | X | | | |
| LDH9 | X | | | | | | | | | | | | | | | | | | | |
| T3, FT4 and TSH <sup>9,10,11</sup> | X | | X | | X | | X | | X | | X | | X | | X <sup>10</sup> | | X | | | |
| Pregnancy Test- Urine or<br>Serum β-hCG <sup>12</sup> | х | | | | | | | | | | | | | | | | | | | |
| Drug Dispensation, Adminis | tratio | n, an | d Ass | ociate | d An | alyse | s | | | | | | | | | | | | | |
| Pembrolizumab<br>Administration <sup>13</sup> | X | X | X | X | x | X | X | х | х | х | Х | X | X | x | х | X | | | | |
| IPI Administration Part 1B <sup>14</sup> | X | X | X | X | | | | | | | | | | | | | | | | |
| IPI Administration Part 1C,<br>Arm 1 <sup>14</sup> | X | | X | | x | | х | | | | | | | | | | | | | |
| IPI Administration Part 1C,<br>Arm 2 <sup>14</sup> | X | | | | X | | | | X | | | | X | | | | | | | |
| Efficacy Measurement | | | | | | | | | | | | | | | | | | | | |
| Tumor Imaging Part 1A and 1B <sup>15,16,17</sup> | X | | | | x | | X | | X | | X | | | | X <sup>16</sup> | | | | X | |
| Tumor Imaging Part<br>1C <sup>15,17,18</sup> | X | | X | | X | | X | | X | | | | X <sup>18</sup> | | X <sup>18</sup> | | | | X | |
| Digital Photography:<br>Cutaneous Lesions <sup>19</sup> | X | X As clinically indicated | | | | | | | | | | | | | | | | | | |

**Protocol/Amendment No.:** 029-05

Treatment cycles are 6 weeks. Imaging should always be performed as scheduled and follow calendar days, regardless of any treatment delays. Subjects may receive Second Course Phase for a maximum of 17 doses of pembrolizumab and 4 doses of IPI. Subjects enrolled in Part 1A who received PEG-IFN who are eligible for Second Course Phase will only be allowed to receive pembrolizumab monotherapy.

- 2. Subjects who discontinue Second Course Phase due to reasons other than disease progression should continue follow-up and assessment by radiologic imaging (and digital photography if applicable) every 12 weeks (± 1 week) for the first year after discontinuation, then every 6 months (± 2 weeks) for year two through five, and every 12 months (± 4 weeks) after year five. Imaging follow-up should continue until (1) the start of new anti-cancer treatment, (2) documented disease progression, (3) death, or (4) the end of the study, whichever occurs first.
- 3. After the start of new anti-cancer treatment or documented disease progression, the subject should be contacted by telephone approximately every 12 weeks after last contact to assess for survival status. In certain situations, survival data may be requested more frequently than every 12 weeks as per Section 7.1.5.3.3. Updated survival status may be requested by the Sponsor at any time during the course of the study. Upon Sponsor notification, all subjects who do not/will not have a scheduled study visit or study contact during the Sponsor-defined time period will be contacted for their survival status (excluding subjects that have a death event previously recorded).
- 4. In general, the window for each visit is  $\pm 3$  days unless otherwise noted.
- 5. Subjects who either a) stopped initial treatment with pembrolizumab after attaining an investigator-determined confirmed CR according to modified RECIST 1.1 (subjects treated with at least 24 weeks of pembrolizumab before discontinuing therapy and received at least two treatments with pembrolizumab beyond the date when the initial CR was declared or b) had SD. PR or CR and stopped pembrolizumab treatment after 24 months of study therapy for reasons other than disease progression or intolerability may restart treatment if they meet the criteria specified in Section 7.1.5.2.1.
- Concomitant medications Enter new medications started during the trial through the Safety Follow-up visit.
- 7. Vital signs to include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.
- 8. Record all AEs occurring within 30 days after the last dose of trial treatment and all SAEs (related and unrelated to trial treatment) / ECIs occurring up until 90 days following cessation of treatment or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier. Afterwards, report only SAEs and ECIs that are related to trial treatment.
- 9. Laboratory tests for determining eligibility for retreatment are to be performed within 10 days prior to the first retreatment dose. See Section 7.1.3 for details regarding laboratory tests.
- 10. After Cycle 1, lab samples can be collected up to 72 hours prior to the scheduled time point. After Cycle 8, lab procedures should be collected every two cycles on D1 (i.e.; C8 D1, C10 D1, C12 D1, etc.). Laboratory results must be known and acceptable prior to dosing. See Section 7.1.3 for details regarding laboratory tests.
- 11. Unresolved abnormal labs that are DRAEs should be followed until resolution.
- 12. For women of reproductive potential, a urine pregnancy test should be performed within 72 hours prior to first dose of trial treatment. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test performed by the local study site laboratory will be required. Pregnancy tests (serum and/or urine tests) should be repeated if required by local guidelines.
- 13. Pembrolizumab will be administered as a 30 minute IV infusion. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes; -5 min/+10 min). Pembrolizumab should always be administered first when given in combination.
- 14. IPI will be administered for a total of 4 doses for subjects that were previously included in Part 1B and for up to 4 doses for subjects that were previously included in Part 1C. Subjects will be administered IPI as a 90 minute IV infusion. Sites should make every effort to target infusion timing to be as close to 90 minutes as possible. For additional instructions regarding dosing please refer to the IPI label. Subjects who initially attain clinical benefit (defined as modified RECIST 1.1 confirmed PR or SD>6 mo), and experience disease progression while receiving single agent pembrolizumab will be eligible for reinduction with up to 4 doses of IPI q3w as long as Part 1A or 1B remain open. Those subjects should follow the assessments detailed in Cycle 2 and beyond

**Protocol/Amendment No.:** 029-05

15. A scan must be performed within 28 days prior to starting treatment with pembrolizumab. Scans performed as part of routine clinical management are acceptable for use as the screening scan if they are of diagnostic quality and performed within 28 days prior to the first dose of trial treatment. Imaging timing should follow calendar days and should not be adjusted for delays in cycle starts or extension of pembrolizumab cycle frequencies.

- 16. For subjects that were previously included in Part 1A and Part 1B, the first imaging assessment should be performed 12 weeks (± 3 days) after the first dose of trial treatment, and continue to be performed every 6 weeks (42 ± 3 days) until week 30, regardless of any treatment delays. Following week 30, tumor imaging will be performed approximately every 12 weeks (84 ± 7 days) (or as clinically indicated) while the subject remains on trial therapy. For subjects that were previously included in Part 1A and 1B, a baseline brain MRI will be performed to rule out brain metastasis.
- 17. Subjects who discontinue trial treatment for a reason other than disease progression should continue to be assessed in Follow-up Phase with the first scan occurring 12 weeks (84 + 7 days) from the date of the last scan on study. The same imaging technique should be used in a subject throughout the trial. Local reading (investigator assessment with site radiology reading) will be used to determine eligibility and for subject management. The Sponsor will collect radiological assessments for retrospective analysis by a central vendor unless otherwise noted by the Sponsor. The processes for image collection and transmission to the central vendor are in the Site Imaging Manual. Per the modified RECIST 1.1 used in this protocol, if imaging shows PD, the imaging assessment should be performed no sooner than 4 weeks later in order to confirm PD as described in Section 4.2.3.2.
- 18. For subjects that were previously included in Part 1C, the first imaging assessment should be performed 6 weeks (± 3 days) after the first dose of trial treatment, and continue to be performed every 6 weeks (42 ± 3 days) until week 24, regardless of any treatment delays. Following week 24, tumor imaging will be performed approximately every 12 weeks (84 ± 7 days or as clinically indicated) while the subject remains on trial therapy. For subjects that were previously included in Part 1C, a baseline brain MRI will be performed to rule out brain metastasis.
- 19. For subject with MEL only: Qualitative digital photography should be performed at baseline and at time of scheduled tumor assessments for cutaneous lesions. Cutaneous lesions are not considered measurable for the purposes of this protocol, but may be considered to be non-target lesions for tumor assessments by investigators. Copies of digital photographs should not be submitted to the central imaging vendor unless otherwise noted by the Sponsor.

Protocol/Amendment No.: 029-05

#### 7.0 TRIAL PROCEDURES

#### 7.1 **Trial Procedures**

The Trial Flow Chart - Section 6.0 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below. It may be necessary to perform these procedures at unscheduled time points if deemed clinically necessary by the investigator.

Furthermore, additional evaluations/testing may be deemed necessary by the investigator and or the Sponsor for reasons related to subject safety. In some cases, such evaluation/testing may be potentially sensitive in nature (e.g., HIV, Hepatitis C, etc.), and thus local regulations may require that additional informed consent be obtained from the subject. In these cases, such evaluations/testing will be performed in accordance with those regulations.

#### 7.1.1 Administrative Procedures

#### 7.1.1.1 Informed Consent

The investigator or qualified designee must obtain documented consent from each potential subject or each subject's legally acceptable representative prior to participating in a clinical trial or Future Biomedical Research.

#### 7.1.1.1.1 General Informed Consent

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the subject before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB/ERC requirements, applicable laws and regulations and Sponsor requirements.

Protocol/Amendment No.: 029-05

## 7.1.1.1.2 Consent and Collection of Specimens for Future Biomedical Research

The investigator or qualified designee will explain the Future Biomedical Research consent to the subject, answer all of his/her questions, and obtain written informed consent before performing any procedure related to the Future Biomedical Research sub-trial. A copy of the informed consent will be given to the subject.

#### 7.1.1.2 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the trial.

## 7.1.1.3 Subject Identification Card

All subjects will be given a Subject Identification Card identifying them as participants in a research trial. The card will contain trial site contact information (including direct telephone numbers) to be utilized in the event of an emergency. The investigator or qualified designee will provide the subject with a Subject Identification Card immediately after the subject provides written informed consent.

#### 7.1.1.4 Medical History

A medical history will be obtained by the investigator or qualified designee. The medical history will collect all active conditions and any condition diagnosed within the prior 10 years that the investigator considers to be clinically significant. Details regarding the disease for which the subject has enrolled in this trial will be recorded separately and not listed as medical history.

#### 7.1.1.5 Prior and Concomitant Medications Review

#### 7.1.1.5.1 Prior Medications

The investigator or qualified designee will review prior medication use, including any protocol-specified washout requirement, and record prior medication taken by the subject within 28 days before starting the trial. Treatment for the disease for which the subject has enrolled in this trial will be recorded separately and not listed as a prior medication.

#### 7.1.1.5.2 Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the subject during the trial through the Safety Follow-up visit. In addition, new medications started during the Second Course Phase through the Second Course Safety Follow-up visit should be recorded.

All medications related to reportable SAEs and ECIs should be recorded as defined in Section 7.2.

04SGNN

Protocol/Amendment No.: 029-05

#### 7.1.1.5.3 Disease Details

The investigator or qualified designee will obtain prior and current details regarding disease status.

## 7.1.1.5.4 Prior Treatment Details

The investigator or qualified designee will review all prior cancer treatments including systemic treatments, radiation and surgeries.

## 7.1.1.5.5 Subsequent Anti-Cancer Therapy Status

The investigator or qualified designee will review all new anti-cancer therapy initiated after the last dose of trial treatment. If a subject initiates a new anti-cancer therapy within 30 days after the last dose of trial treatment, the 30 day Safety Follow-up visit must occur before the first dose of the new therapy. Once new anti-cancer therapy has been initiated the subject will move into SFU.

#### 7.1.1.6 Assignment of Screening Number

All consented subjects will be given a unique screening number that will be used to identify the subject for all procedures that occur prior to randomization or allocation. Each subject will be assigned only one screening number. Screening numbers must not be re-used for different subjects.

Any subject who is screened multiple times will retain the original screening number assigned at the initial screening visit.

Specific details on the screening visit requirements (screening/rescreening) are provided in Section 7.1.5.1.

#### 7.1.1.7 Assignment of Randomization Number

All eligible subjects will be randomly allocated and will receive a randomization number. The randomization number identifies the subject for all procedures occurring after randomization. Once a randomization number is assigned to a subject, it can never be reassigned to another subject.

A single subject cannot be assigned more than 1 randomization number.

Drug administration should start within 7 days from assignment of a randomization number.

#### 7.1.1.8 Trial Compliance (Medication/Diet/Activity/Other)

Interruptions from the protocol specified treatment plan for greater than 12 weeks between pembrolizumab doses for nondrug-related or administrative reasons require consultation between the investigator and the Sponsor and written documentation of the collaborative decision on subject management.

7-Nov-2017

Protocol/Amendment No.: 029-05

Administration of first dose of PEG-IFN will be witnessed by the investigator and/or trial staff on Day 1. Drug accountability will be collected during the study. Compliance with PEG-IFN administration will be measured by subjects: 1) receiving unscheduled study agent injections; 2) missing an injection. Numbers and percentages of subjects and injection visits with any deviation in these measures will be reported.

The instructions for preparing and administering trial treatments will be provided in the Study Manuals.

#### 7.1.2 Clinical Procedures/Assessments

## 7.1.2.1 Adverse Event (AE) Monitoring

The investigator or qualified designee will assess each subject to evaluate for potential new or worsening AEs as specified in the Trial Flow Chart (Section 6) and more frequently if clinically indicated. Adverse events will be graded and recorded throughout the trial and during the follow-up period according to NCI CTCAE Version 4.0 (see [Section 12.5). Toxicities will be characterized in terms including seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

All AEs of unknown etiology associated with pembrolizumab exposure should be evaluated to determine if it is possibly an event of clinical interest (ECI) of a potentially immunologic etiology (irAE). See Section 5.6.1 and the separate guidance document in the administrative binder regarding the identification, evaluation, and management of AEs of a potential immunological etiology.

Please refer to Section 7.2 for detailed information regarding the assessment and recording of AEs.

#### 7.1.2.2 Physical Exam

#### 7.1.2.2.1 Full Physical Exam

The investigator or qualified designee will perform a complete physical exam during the Screening period. Clinically significant abnormal findings should be recorded as medical history. The time points for full physical exams are described in Section 6. After the first dose of trial treatment, new clinically significant abnormal findings should be recorded as AEs.

#### 7.1.2.2.2 Directed Physical Exam

For cycles that do not require a full physical exam as defined in Section 6, the investigator or qualified designee will perform a directed physical exam as clinically indicated prior to the administration of the trial treatment. New clinically significant abnormal findings should be recorded as AEs.

**Product:** MK-3475 93

**Protocol/Amendment No.:** 029-05

#### **7.1.2.3 Vital Signs**

Vital signs include temperature, pulse, respiratory rate, weight and blood pressure. The investigator or qualified designee will take vital signs at screening, prior to the administration of each dose of trial treatment and during the follow-up period as specified in the Trial Flow Chart (Section 6). Height will be measured at Screening.

#### 7.1.2.4 Electrocardiogram (ECG)

A standard 12-lead ECG will be performed using local standard procedures at Screening. Clinically significant abnormal findings should be recorded as medical history. Additional time points for standard 12-lead ECGs must be performed as per Section 6 – Trial Flow Charts. Clinically significant abnormal findings seen on the follow-up ECGs should be recorded as adverse events.

## 7.1.2.5 Eastern Cooperative Oncology Group (ECOG) Performance Scale

The investigator or qualified designee will assess ECOG status (see Appendix 12.4) at screening, additional time points for assessment of ECOG must be performed as per Section 6 – Trial Flow Charts.

#### 7.1.2.6 Tumor Tissue Collection

Tumor tissue for biomarker analysis from formalin fixed paraffin embedded tumor tissue sample or newly obtained formalin fixed biopsy of a tumor lesion not previously irradiated must be provided in the form of a tissue block or at least ten unstained slides and received by the central vendor and tested for PD-L1 status by IHC before randomization. Subjects will be enrolled in the trial regardless of the expression. Subjects who do not submit a sample adequate for PD-L1 determination will not be enrolled. Subjects with an archival sample considered not adequate may obtain a new biopsy. Subjects with a newly obtained biopsy considered not adequate may undergo re-biopsy at the discretion of the investigator. Note for Part 1C: adequacy of the tumor sample for determination of PD-L1 status by IHC at a central pathology laboratory prior to enrollment is not required. Additional biopsy sample submission is encouraged but not mandatory for Part 1C when the sample is inadequate for PD-L1 testing.

Note: A fine needle aspirate or cytologic specimen will not be acceptable. Core needle or excisional biopsies, or resected tissue is required. Newly obtained formalin fixed specimens are encouraged.

If new scientific data emerge that indicate that an existing biopsy or surgical specimen is suboptimal for identification of subjects, then only new biopsies will be acceptable for determination of PD-L1 status.

If the subject signs the Future Biomedical Research (FBR) consent, any leftover tissue biopsies that would ordinarily be discarded at the end of the main study will be retained for FBR, again providing the subject has signed the FBR consent.

MK-3475-029-05 Final Protocol

04SGNN

**Protocol/Amendment No.:** 029-05

Detailed instructions for tissue collection, processing and shipment are provided in the Laboratory Manual.

#### 7.1.2.7 Tumor Imaging and Assessment of Disease

The process for image collection and transmission to the central imaging vendor can be found in the Site Imaging Manual (SIM). Tumor imaging is strongly preferred to be acquired by computed tomography (CT). Magnetic resonance imaging (MRI) should be used only when CT is contraindicated or for imaging of the brain. The same imaging technique regarding modality and the use of contrast should be used in a subject throughout the trial to optimize the visualization of existing and new tumor burden.

At least 1 year after the last subject has enrolled in Parts 1A, 1B and 1C, the Sponsor may elect to halt central vendor imaging collection and continue with investigator assessment only. If this switch will occur, the decision will be announced through an administrative memo from the Sponsor.

#### 7.1.2.8 Assessment of Disease

The primary measure for assessment of tumor response will be based on independent central review using RECIST 1.1 [1]. RECIST 1.1 will be used by independent central review as the primary measure for assessment of tumor response, date of disease progression, and as a basis for all protocol guidelines related to disease status (eg, discontinuation of trial therapy). Although RECIST 1.1 references a maximum of 5 target lesions in total and 2 per organ, the Sponsor allows a maximum of 10 target lesions in total and 5 per organ, if clinically relevant to enable a broader sampling of tumor burden.

Modified RECIST 1.1 will be applied by the site as the basis for all protocol guidelines related to disease status (e.g., discontinuation of study therapy).

RECIST 1.1 will be adapted as follows to account for the unique tumor response seen in this class of therapeutics.

If RECIST 1.1 defined progression has been assessed then the subject will be discontinued from trial treatment unless, in the opinion of the investigator, the subject is deriving clinical benefit from the therapy and the subject does not have any signs or symptoms of clinical instability as discussed in Table 11 Imaging and Treatment after 1st Radiologic Evidence of PD in Section 5.2.3.

Clinically stable is defined by the following criteria:

- Absence of signs and symptoms (including worsening of laboratory values) indicating clinically significant disease progression
- No decline in ECOG performance status
- Absence of rapid progression of disease
- Absence of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention

MK-3475-029-05 Final Protocol 7-Nov-2017

**Protocol/Amendment No.:** 029-05

Note: Treatment may be continued despite modified RECIST 1.1 defined progression if the subject is clinically stable and is considered to be deriving clinical benefit by the investigator. In these cases, subjects should continue to undergo imaging as outlined in the footnote in Table 11.

#### 7.1.2.9 Ophthalmologic Examination

All subjects receiving pembrolizumab + PEG-IFN should have a baseline ophthalmologic exam including visual acuity, visual field and color discrimination by an ophthalmologist. Fundus photography should be performed in subjects with history of clinically significant retinal disease (defined as macular degeneration, retinal detachment and moderate/severe non-proliferative diabetic retinopathy and any proliferative diabetic retinopathy). Enrollment of subjects with clinically significant retinal disease will require consultation with the sponsor on risk-benefit associated to treatment. Any subject randomized in the pembrolizumab + PEG-IFN treatment group complaining of ocular symptoms, including loss of visual acuity or visual field must have a prompt and complete ophthalmologic examination. In addition, because these ocular events may occur in conjunction with other disease states, periodic visual examinations during the trial are recommended in subjects with disorders that may be associated with retinopathy, such as diabetes mellitus or hypertension. Discontinuation of PEG-IFN should be considered in subjects who develop new or worsening ophthalmological disorders.

#### 7.1.3 Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below. The total amount of blood/tissue to be drawn/collected over the course of the trial (from pre-trial to post-trial visits), including approximate blood/tissue volumes drawn/collected by visit and by sample type per subject can be found in the Trial Laboratory Manual. Refer to the Trial Flow Chart (Section 6) for the timing of laboratory assessments.

## 7.1.3.1 Laboratory Safety Evaluations (Hematology, Chemistry and Urinalysis)

Laboratory tests for hematology, chemistry, and urinalysis are specified in Table 12.

**Protocol/Amendment No.:** 029-05

Table 12 Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hematocrit | Albumin | Blood | Pregnancy test (serum or urine) <sup>a</sup> |
| Hemoglobin | Alkaline phosphatase | Glucose | PT/INR |
| Platelet count | Alanine aminotransferase | Protein | aPTT |
| WBC (total and differential) <sup>d</sup> | Amylase | Specific gravity | Total T3 or free T3, FT4, and TSH <sup>b</sup> |
| RBC | Aspartate aminotransferase | Microscopic exam, if abnormal results are noted | Anti-HCV <sup>e</sup> |
| Absolute lymphocyte count <sup>d</sup> | Bicarbonate <sup>c</sup> | | HCV viral load <sup>e</sup> |
| Absolute neutrophil count <sup>d</sup> | Calcium | | HCV genotype <sup>e</sup> |
| | Chloride | | anti-HBs <sup>e</sup> |
| | Creatinine | | HBsAg <sup>e</sup> |
| | Glucose | | Anti-HBc (total and IgM) <sup>e</sup> |
| | LDH <sup>e</sup> | | HBeAg <sup>e</sup> |
| | Lipase | | anti-HBe <sup>e</sup> |
| | Magnesium | | HBV viral load <sup>e</sup> |
| | Phosphorus | | |
| | Potassium | | AFP <sup>e</sup> |
| | Sodium | | CRP <sup>e</sup> |
| | Total bilirubin | | GGT <sup>e</sup> |
| | Direct bilirubin | | |
| | Total protein | | |
| | Blood urea nitrogen | | |

<sup>&</sup>lt;sup>a</sup> Perform on women of childbearing potential only 72 hours prior to Day 1 of Cycle 1. Pregnancy tests must be repeated prior to every cycle if required or as specified per local regulatory guidance.

Note: If the local laboratory is unable to perform these tests, the site should submit the sample to the central laboratory for testing. Details are provided in the Laboratory Manual.

AFP=alpha-fetoprotein; aPTT=activated partial thrombin time; CRP=C-reactive protein; FT4=free thyroxine; GGT=gamma-glutamyl transferase; HBc=hepatitis B core; HBeAg=hepatitis B e antigen; HBe=hemoglobin E; HBs=hepatitis B surface; HBsAg=hepatitis B surface antigen; HBV=hepatitis B virus; HCV=hepatitis C virus; IgM=gamma M immunoglobulin; INR=insulin receptor; LDH=lactate dehydrogenase; PT=prothrombin time; RBC=red blood cells; T3=triothyronine; TSH=thyroid stimulating hormone (thyrotropin); WBC=white blood cells.

Laboratory tests for screening or entry into the Second Course Phase should be performed within 10 days prior to the first dose of trial treatment. An exception is hepatitis and thyroid serologies, which may be performed within 28 days prior to first dose. After Cycle 1, pre-dose laboratory procedures can be conducted up to 72 hours prior to dosing. After Cycle

04SGNN

<sup>&</sup>lt;sup>b</sup> T3 is preferred; if not available, free T3 may be tested.

<sup>&</sup>lt;sup>c</sup> If this test is not done as part of local standard of care, this test does not need to be performed.

d Report % or absolute results per standard of practice. Report the results in the same manner throughout the trial.

e These tests should be performed at screening, and then as clinically indicated, except for AFP and GGT, which should only be performed as clinically indicated. For the purpose of determining eligibility, perform HBsAg and HCV viral load. Anti-HCV is allowed for screening purposes in countries where HCV viral load is not part of standard of care. All other hepatitis tests should be performed per standard of care.

Protocol/Amendment No.: 029-05

8, lab procedures should be collected every two cycles on D1 (i.e., C8 D1, C10 D1, C12 D1, etc.).

Laboratory test results must be reviewed by the investigator or qualified designee and found to be acceptable prior to administration of each dose of trial treatment. Unresolved abnormal laboratory values that are DRAEs should be followed until resolution. Laboratory tests do not need to be repeated after the end of treatment if laboratory results are within the normal range.

#### 7.1.3.1.1 Serum/Urine β-hCG

All women who are being considered for participation in the trial, and who are not surgically sterilized or postmenopausal will be tested for pregnancy within 72 hours of receiving the first dose of study medication, and must be excluded in the event of a positive or borderline-positive test result. If a urine test is positive or not evaluable, a serum test will be required.

#### 7.1.3.2 Pharmacokinetic/Pharmacodynamic Evaluations

Blood samples for PK, ADA and total IgG analyses will be collected at the time points described in Table 13 and below. The actual date and time of each blood sample collection will be recorded in the eCRF. The timing of PK samples may be altered and/or PK samples may be obtained at additional time points to ensure thorough PK monitoring.

Table 13 Pharmacokinetic, Total IgG, and ADA Assessments

| | | | | | | | | | Trea | tmen | t | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| pembrolizumab<br>Dose Number | 1 | 2 | 3 | 4 | 5 | 7 | 9 | 13 | 17 | 19 | 21 and<br>every 4 <sup>th</sup><br>dose<br>thereafter | 25,<br>31,<br>37,<br>43,<br>49 | 30 day post-<br>pembrolizumab<br>treatment |
| Cohort A | | | | | | | | | | | | | |
| Pembrolizumab | X | X | | X | | X | | X | | X | | X | X |
| Cohort B q3w | | | | | | | | | | | | | |
| Pembrolizumab | X | X | | X | | X | | X | | X | | X | X |
| IPI | X | | | X | X | | | | | | | | |
| Cohort B q6w and q | 12w | | | | | | | | | | | | |
| Pembrolizumab | X | | X | | X | | X | X | X | X | X | | |
| IPI q6w | X | | X | | X | X | X | | | | | | |
| IPI q12w | X | | | | X | | X | X | X | | | | |
| All pembrolizumab<br>Antibody Test | X | X | | | | X | | X | | X | | X | X |
| Total IgG Assessmen | nt | | | | | | | | | | | | |
| At all pre-dose<br>pembrolizumab PK | X | X | | X | | X | | X | | X | | X | |

Table 14 Timing of PK and ADA Assessments, Parts 1A and 1B

| Drug | Study Part | Pembrolizumab Dose<br>Number | Time of PK and ADA Blood Sample Collection |
|---|---|---|---|
| IPI (PK and ADA) | Treatment Phase | Dose 1 and 4 | Predose IPI: within 60 min before the infusion of IPI Postdose IPI: within 30 min after end of infusions of IPI (only PK) |
| | | Dose 5 (q3w) | Predose pembrolizumab: within 60 min before the infusion of pembrolizumab |
| pembrolizumab<br>(total IgG <sup>a</sup> , PK<br>and ADA) | Treatment Phase | Dose 1 | Predose pembrolizumab: within 60 min before the start of the infusion and prior to a potential IPI or PEG-IFN dosing on the same day <sup>d</sup> Only for pembrolizumab ( <b>not for total IgG and ADA</b> ): Postdose pembrolizumab: within 30 min after the end of the infusion Only for pembrolizumab ( <b>not for total IgG and ADA</b> ): Postdose pembrolizumab: at Day 8 (and prior to a potential IPI or PEG-IFN dosing on that same day) |
| | | Dose 2, 4, 7, 13, etc. <sup>b</sup> | Predose pembrolizumab: within 60 min before the start of the infusion For ADA: Predose pembrolizumab within 60 min before start of the infusion EXCEPT for the 4th dose of pembrolizumab |
| | | 30 day post<br>pembrolizumab<br>treatment <sup>c</sup> | Obtain a PK blood sample at 30 days (±7 days) after the last dose of pembrolizumab and at the same time that the blood sample is obtained for anti-pembrolizumab antibody testing |

<sup>a. Total IgG should be collected simultaneous with every pre-dose pembrolizumab PK sampling.
b. After Dose #7 of pembrolizumab, obtain PK and total IgG blood samples before dosing of every 6th dose for the duration of the study (i.e., pembrolizumab dose 13, 19, 25,</sup> 31, 37, 43, and 49).

c. Post-treatment samples may not be collected if the subject has started treatment with a new anti-cancer therapy.

d. Predose pembrolizumab samples should be obtained at the same time that blood samples are drawn for total IgG and anti-pembrolizumab antibody testing (ADA).

Protocol/Amendment No.: 029-05

Table 15 Timing of PK and ADA Assessments, Part 1C

| Drug | Study Part | Pembrolizumab Dose Number | Time of PK and ADA Blood Sample Collection |
|---|---|---|---|
| IPI <sup>a</sup> (PK and ADA) | Treatment Phase | Arm 1 (50 mg q6w): dose 1, 3, 5, 7, 9<br>Arm 2 (100 mg q12w): dose 1, 5, 9,<br>13, 17 | Predose IPI: within 60 min before the infusion of IPI Postdose IPI: within 30 min after end of infusions of IPI (only PK) |
| Pembrolizumab <sup>a</sup> (total IgG <sup>b</sup> , PK, and ADA) | Treatment Phase | Dose 1, 3, 5, 9, then every 4 <sup>th</sup> dose thereafter | Predose pembrolizumab: within 60 min before the start of the infusion <sup>c</sup> |

NOTE: Only three samples will be collected at visits which require IPI and pembrolizumab PK. The predose sample will be the baseline for both pembrolizumab and IPI PK

NOTE: All PK and ADA samples should be taken at the same time.

a At time points with both pembrolizumab and IPI samples, predose IPI and predose pembrolizumab samples can be obtained from the same extraction.

b Total IgG should be collected simultaneous with every pre-dose pembrolizumab PK sampling.

c Predose pembrolizumab samples should be obtained at the same time that blood samples are drawn for total IgG and anti-pembrolizumab antibody testing (ADA).

**Protocol/Amendment No.:** 029-05

#### 7.1.3.2.1 Blood Collection for Serum MK-3475

Sample collection, storage and shipment instructions for serum samples will be provided in the Laboratory Manual.

#### 7.1.3.2.2 Blood Collection for Anti-MK-3475 Antibodies (ADA)

Sample collection, storage and shipment instructions for serum samples will be provided in the Laboratory Manual.

Every effort should be taken to collect samples at 30 days after end of pembrolizumab treatment for ADA.

Simultaneous PK sampling is required for interpretation of ADA analysis.

## 7.1.3.2.3 Blood Collection for total IgG

Endogenous IgG levels were found in internal unpublished studies to be a factor significantly affecting the exposure of pembrolizumab. Additional information about individual IgG levels is required to confirm this effect, in particular when patients do receive immune modulatory co-medications such as PEG-IFN and IPI.

Total IgG should be collected simultaneous with every pre-dose pembrolizumab PK sampling.

#### 7.1.3.3 Future Biomedical Research

The following specimens are to be obtained as part of Future Biomedical Research:

- Blood for genomics use
- Leftover correlative blood samples
- Leftover blood for genetics sample
- Leftover archival tumor tissue or leftover newly obtained biopsy samples taken throughout the study

#### 7.1.4 Other Procedures

#### 7.1.4.1 Withdrawal/Discontinuation

Subjects who discontinue/withdraw from treatment prior to completion of the treatment regimen should be encouraged to continue to be followed for all remaining study visits.

When a subject discontinues/withdraws from participation in the trial, all applicable activities scheduled for the final trial visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 - Assessing and Recording Adverse Events. In Part 1A and 1B and upon Sponsor consultation, subjects who

**Protocol/Amendment No.:** 029-05

either a) stopped initial treatment with pembrolizumab after attaining an investigatordetermined confirmed CR according to modified RECIST 1.1 (subjects treated with at least 24 weeks of pembrolizumab before discontinuing therapy and received at least two treatments with pembrolizumab beyond the date when the initial CR was declared) or b) had SD, PR or CR and stopped pembrolizumab treatment after 24 months of study therapy for reasons other than disease progression or intolerability may restart trial Second Course Phase if they meet the criteria specified in Section 7.1.5.2.1. Additionally in Part 1C and upon Sponsor consultation, subjects who a) attain an investigator-determined CR or b) a VGPR and complete treatment with at least one dose of IPI on either Arm of treatment may discontinue treatment with IPI with the option of restarting the Second Course Phase if they meet the criteria specified in Section 7.1.5.2.1. After discontinuing treatment following assessment of CR, these subjects should return to the site for a Safety Follow-up Visit (described in Section 7.1.5.3.1) and then proceed to the Follow-Up Period of the study (described in Section 7.1.5.3.2) and SFU (described in Section 7.1.5.3.3).

#### 7.1.4.1.1 Withdrawal From Future Biomedical Research

Subjects may withdraw their consent for Future Biomedical Research and have their specimens and all derivatives destroyed. Subjects may withdraw consent at any time by contacting the principal investigator for the main trial. If medical records for the main trial are still available, the investigator will contact the Sponsor using the designated mailbox (clinical specimen management@merck.com), and a form will be provided by the Sponsor to obtain appropriate information to complete specimen withdrawal. Subsequently, the subject's specimens will be removed from the biorepository and be destroyed. A letter will be sent from the Sponsor to the investigator confirming the destruction. It is the responsibility of the investigator to inform the subject of completion of destruction. Any analyses in progress at the time of request for destruction or already performed prior to the request being received by the Sponsor will continue to be used as part of the overall research trial data and results. No new analyses would be generated after the request is received.

In the event that the medical records for the main trial are no longer available (e.g., if the investigator is no longer required by regulatory authorities to retain the main trial records) or the specimens have been completely anonymized, there will no longer be a link between the subject's personal information and their specimens. In this situation, the request for specimen destruction cannot be processed.

#### 7.1.4.2 Blinding/Unblinding

This is an open label trial; there is no blinding for this trial.

#### 7.1.4.3 Calibration of Critical Equipment

The investigator or qualified designee has the responsibility to ensure that any critical device or instrument used for a clinical evaluation/test during a clinical trial that provides important information about inclusion/exclusion criteria and/or safety or efficacy parameters shall be suitably calibrated and maintained to ensure that the data obtained is reliable and/or

04SGNN

**Protocol/Amendment No.:** 029-05

reproducible. Documentation of equipment calibration must be retained with the study documentation as source documentation at the trial site.

Critical Equipment for this trial includes:

- Laboratory equipment as required for inclusion labs and trial assessments
- Imaging equipment as required for study objectives See Protocol-specific Administrative Binder and Site Imaging Manual.

## 7.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

## **7.1.5.1** Screening

Within 28 days prior to treatment randomization, potential subjects will be evaluated to determine that they fulfill the entry requirements as set forth in Section 5.1. Visit requirements are outlined in the Trial Flow Chart (Section 6). Screening procedures may be repeated.

Written consent must be obtained prior to performing any protocol-specific procedure. Results of a test performed prior to the subject signing consent as part of routine clinical management are acceptable in lieu of a screening test if performed within the specified time frame. Screening procedures are to be completed within 28 days prior to the first dose of trial treatment except for the following:

- Laboratory tests are to be performed within 10 days prior to the first dose of trial treatment.
- For women of reproductive potential, a urine pregnancy test will be performed within 72 hours prior to first dose of trial treatment. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test, performed by the local study site laboratory, will be required.
- Tumor imaging must be performed within 28 days prior to the first dose of trial treatment.

Subjects may be rescreened after initially failing to meet the inclusion/exclusion criteria. Results from assessments performed during the initial screening period are acceptable in lieu of a repeating a screening test if performed within the specified time frame and the results meet the inclusion/exclusion criteria.

#### 7.1.5.2 Treatment Period

Visit requirements are outlined in the Trial Flow Chart (Section 6). Specific procedure-related details are provided in Section 7.1.

After a screening phase of up to 28 days, eligible subject will receive assigned treatment on Day 1 of each dosing cycle and thereafter following a weekly (PEG-IFN) or every 3, 6 or

MK-3475-029-05 Final Protocol 7-Nov-2017

**Protocol/Amendment No.:** 029-05

12 weeks (IPI) schedule, depending on the part and the treatment group in which the subject is enrolled. Pembrolizumab will be given q3w. A cycle is 6 weeks. Additional information regarding the DLT assessment period can be found in Section 5.2.1.2.1.

Treatment with pembrolizumab + PEG-IFN doublet will continue until up to two years of therapy have been administered, documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.

In Parts 1A and 1B, treatment with pembrolizumab + IPI doublet will continue for 2 cycles (12 weeks), followed by treatment with pembrolizumab single agent until up to 24 months of therapy have been administered, documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.

In Part 1C, treatment with pembrolizumab + IPI doublet will continue for a maximum of 4 cycles (24 weeks) or 8 cycles (48 weeks), for Arm 1 and Arm 2, respectively, followed by treatment with pembrolizumab single agent until up to 24 months of therapy have been administered, documented disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.

#### 7.1.5.2.1 Second Course Phase

Upon Sponsor consultation, subjects who stop pembrolizumab with SD or better per modified RECIST 1.1 may be eligible for retreatment with pembrolizumab + IPI at a dose of pembrolizumab of 200 mg q3w or pembrolizumab 200 mg q3w monotherapy if they progress after stopping pembrolizumab, at the discretion of the investigator, as long as the Part to which the subject was initially enrolled remains open. This retreatment is termed the Second Course Phase of this trial. Subjects enrolled in Part 1A who received PEG-IFN and who are eligible for the Second Course Phase will only be allowed to receive pembrolizumab monotherapy. The Second Course Phase will be administered for a maximum of 17 doses of pembrolizumab and 4 doses of IPI. The Second Course Phase of this trial is only available if the subject meets the following conditions:

#### • Either

07W8HB

- Stopped initial treatment with pembrolizumab after attaining an investigatordetermined confirmed CR according to modified RECIST 1.1.
  - Was treated for at least 24 weeks with pembrolizumab before discontinuing therapy.
  - Received at least two treatments with pembrolizumab beyond the date when the initial CR was declared.

**Protocol/Amendment No.:** 029-05

#### OR

Subject had SD, PR or CR and stopped pembrolizumab treatment after 24 months of study therapy for reasons other than disease progression or intolerability.

#### **AND**

- Experienced an investigator-determined confirmed radiographic progression after stopping their initial treatment with pembrolizumab.
- Did not receive any anti-cancer treatment since the last dose of pembrolizumab.
- Have a performance status of 0 or 1 on the ECOG Performance Scale.
- Demonstrate adequate organ function as detailed in Section 5.1.2.
- o Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving retreatment with study medication.
- Female subjects of childbearing potential should be willing to adhere to the contraception requirements outlined in Section 5.7.2 for the course of the study through 120 days after the last dose of study medication. Subjects of child bearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
- Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
- o Does not have a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the trial or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Subjects in the Second Course Phase will restart retreatment with pembrolizumab + IPI at a dose of pembrolizumab of 200 mg q3w or pembrolizumab 200 mg q3w monotherapy. Subjects will not be allowed to restart the Second Course with pembrolizumab + PEG-IFN. The Second Course Phase will be administered for a maximum of 17 doses of pembrolizumab and 4 doses of IPI.

Visit requirements are outlined in Section 6.2 – Trial Flow Chart for Second Course of Treatment. Treatment beyond confirmed PD is not permitted for Second Course Phase.

#### 7.1.5.3 Post-Treatment Visits

#### 7.1.5.3.1 Safety Follow-up Visit

The mandatory Safety Follow-up Visit should be conducted approximately 30 days after the last dose of trial treatment or before the initiation of a new anticancer treatment, whichever comes first.

04SGNN

Protocol/Amendment No.: 029-05

All AEs that occur prior to the Safety Follow-Up Visit should be recorded. Subjects with an AE of Grade >1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anticancer therapy, whichever occurs first. Serious AEs that occur within 90 days of the end of treatment or 30 days following cessation of trial treatment if the subject initiates new anticancer therapy should also be followed and recorded.

Subjects who are eligible for retreatment with pembrolizumab may have up to 2 safety follow-up visits, 1 after the Initial Treatment Period and 1 after the Second Course Treatment.

#### 7.1.5.3.2 Follow-up Visits

Subjects who discontinue trial treatment for a reason other than disease progression will move into the Follow-Up Phase and should be assessed every 12 weeks (± 1 week) for the first year after discontinuation, then every 6 months (± 2 weeks) for years two through five, and every 12 months (± 4 weeks) after year five to monitor disease status. The Sponsor may request survival status to be assessed at additional time points during the course of the study (not to exceed approximately 12 weeks). Every effort should be made to collect information regarding disease status until the start of new anti-cancer therapy, disease progression, death, end of trial [or if the subject begins retreatment with pembrolizumab as detailed in Section 7.1.5.2.1]. Information regarding post-trial anticancer treatment will be collected if new treatment is initiated.

Subjects who are eligible to receive retreatment with pembrolizumab according to the criteria in Section 7.1.5.2 will move from the Follow-Up Phase to the Second Course Phase when they experience disease progression. Details are provided in the Trial Flow Chart (Section 6) for retreatment with pembrolizumab.

## 7.1.5.3.3 Survival Follow-up (SFU)

Subjects who experience confirmed disease progression or start a new anticancer therapy, will move into the SFU Phase and should be contacted by telephone approximately every 12 weeks from the last contact date to assess for survival status until death, withdrawal of consent, or the end of the trial, whichever occurs first.

#### 7.1.5.4 Survival Status

To ensure current and complete survival data are available at the time of database locks, updated survival status may be requested during the course of the study by the Sponsor. For example, updated survival status may be requested prior to but not limited to an external Data Monitoring Committee review, interim and/or final analysis. Upon Sponsor notification, all subjects who do not/will not have a scheduled study visit or study contact during the Sponsor-defined time period will be contacted for their survival status (excluding subjects that have a previously recorded death event in the collection tool).

**Protocol/Amendment No.:** 029-05

07W8HB

## 7.2 Assessing and Recording Adverse Events

An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.

Changes resulting from normal growth and development that do not vary significantly in frequency or severity from expected levels are not to be considered adverse events. Examples of this may include, but are not limited to, teething, typical crying in infants and children and onset of menses or menopause occurring at a physiologically appropriate time.

Sponsor's product includes any pharmaceutical product, biological product, device, diagnostic agent or protocol-specified procedure, whether investigational (including placebo or active comparator medication) or marketed, manufactured by, licensed by, provided by or distributed by the Sponsor for human use.

Adverse events may occur during clinical trials or as prescribed in clinical practice, from overdose (whether accidental or intentional), from abuse and from withdrawal.

Progression of the cancer under study is not considered an adverse event.

All adverse events that occur after the consent form is signed but before treatment allocation/randomization must be reported by the investigator if they cause the subject to be excluded from the trial, or are the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

From the time of treatment allocation/randomization through 30 days following cessation of treatment, all adverse events must be reported by the investigator. Such events will be recorded at each examination on the Adverse Event case report forms/worksheets. The reporting timeframe for adverse events meeting any serious criteria is described in section 7.2.3.1. The investigator will make every attempt to follow all subjects with non-serious adverse events for outcome.

Electronic reporting procedures can be found in the Electronic Data Capture (EDC) data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent).

# 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor

For purposes of this trial, an overdose is any dose higher than 20% over the prescribed dose for pembrolizumab or IPI, or any dose exceeding the prespecified dose of pembrolizumab by

MK-3475-029-05 Final Protocol 7-Nov-2017

**Protocol/Amendment No.:** 029-05

≥1000 mg (5 times the dose) for pembrolizumab 200 mg fixed dosing, or any dose exceeding the prescribed dose for PEG-IFN by 50%. No specific information is available on the treatment of overdose of pembrolizumab. In the event of overdose, PEG-IFN should be discontinued and the subject should be observed closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated.

If an adverse event(s) is associated with ("results from") the overdose of Sponsor's product or vaccine, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.

If a dose of Sponsor's product or vaccine meeting the protocol definition of overdose is taken without any associated clinical symptoms or abnormal laboratory results, the overdose is reported as a non-serious Event of Clinical Interest (ECI), using the terminology "accidental or intentional overdose without adverse effect."

All reports of overdose with and without an adverse event must be reported within 24 hours to the Sponsor either by electronic media or paper. Sponsor Contact information can be found in the Investigator Trial File Binder (or equivalent).

## 7.2.2 Reporting of Pregnancy and Lactation to the Sponsor

Although pregnancy and lactation are not considered adverse events, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject (spontaneously reported to them) that occurs during the trial.

Pregnancies and lactations that occur after the consent form is signed but before treatment allocation/randomization must be reported by the investigator if they cause the subject to be excluded from the trial, or are the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

Pregnancies and lactations that occur from the time of treatment allocation/randomization through 120 days following cessation of Sponsor's product, or 30 days following cessation of trial treatment if the subject initiates new anticancer therapy, whichever is earlier, must be All reported pregnancies must be followed to the reported by the investigator. completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

Such events must be reported within 24 hours to the Sponsor either by electronic media or paper. Sponsor Contact information can be found in the Investigator Trial File Binder (or equivalent).

04SGNN

**Protocol/Amendment No.:** 029-05

## 7.2.3 Immediate Reporting of Adverse Events to the Sponsor

#### 7.2.3.1 Serious Adverse Events

A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that:

- Results in death;
- Is life threatening;
- Results in persistent or significant disability/incapacity;
- Results in or prolongs an existing inpatient hospitalization;
- Is a congenital anomaly/birth defect;
- Is an other important medical event

<u>Note:</u> In addition to the above criteria, adverse events meeting either of the below criteria, although not serious per ICH definition, are reportable to the Sponsor in the same timeframe as SAEs to meet certain local requirements. Therefore, these events are considered serious by the Sponsor for collection purposes.

- Is a new cancer (that is not a condition of the study);
- Is associated with an overdose.

Refer to Table 16 for additional details regarding each of the above criteria.

For the time period beginning when the consent form is signed until treatment allocation/randomization, any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study (reference Section 7.2.3.3 for additional details), that occurs to any subject must be reported within 24 hours to the Sponsor if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment allocation/randomization through 90 days following cessation of trial treatment, or 30 days following cessation of trial treatment if the subject initiates new anticancer therapy, whichever is earlier, any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study (reference Section 7.2.3.3 for additional details), whether or not related to the Sponsor's product, must be reported within 24 hours to the Sponsor either by electronic media or paper. Electronic reporting procedures can be found in the EDC data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent)

Additionally, any serious adverse event, considered by an investigator who is a qualified physician to be related to the Sponsor's product that is brought to the attention of the investigator at any time following consent through the end of the specified safety follow-up period specified in the paragraph above, or at any time outside of the time period specified in the previous paragraph also must be reported immediately to the Sponsor.

All subjects with serious adverse events must be followed up for outcome.
**Protocol/Amendment No.:** 029-05

#### 7.2.3.2 Events of Clinical Interest

Selected non-serious and serious adverse events are also known as Events of Clinical Interest (ECI) and must be reported to the Sponsor.

For the time period beginning when the consent form is signed until treatment allocation/randomization, any ECI, or follow up to an ECI, that occurs to any subject must be reported within 24 hours to the Sponsor if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment allocation/randomization through 90 days following cessation of treatment, or 30 days following cessation of trial treatment if the subject initiates new anticancer therapy, whichever is earlier, any ECI or follow up to an ECI, whether or not related to the Sponsor's product, must be reported within 24 hours to the Sponsor, either by electronic media or paper. Electronic reporting procedures can be found in the EDC data entry guidelines. Paper reporting procedures can be found in the Investigator Trial File Binder (or equivalent).

Events of clinical interest for this trial include:

- 1. an overdose of Sponsor's product, as defined in Section 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor, that is not associated with clinical symptoms or abnormal laboratory results.
- 2. an elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing.\*
  - \*Note: These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology. The trial site guidance for assessment and follow up of these criteria can be found in the Investigator Trial File Binder (or equivalent).
- 3. In the event a subject develops any of the following AEs, a detailed narrative of the event should be reported as an ECI to the SPONSOR within 24 hours of the event:
  - a. Grade  $\geq 3$  diarrhea
  - b. Grade  $\geq 2$  colitis
  - c. Grade  $\geq 2$  pneumonitis
  - d. Grade  $\geq$  3 hypo- or hyperthyroidism
  - e. Grade  $\geq$  2 Depression

07W8HB

A separate guidance document has been provided entitled "Pembrolizumab Events of Clinical Interest and Immune-Related Adverse Event Guidance Document." This document

Protocol/Amendment No.: 029-05

can be found in the administrative binder and provides guidance regarding identification, evaluation and management of ECIs and irAEs. Additional ECIs are identified in this guidance document and also need to be reported to the SPONSOR within 24 hours of the event.

Subjects should be assessed for possible ECIs prior to each dose. Lab results should be evaluated and subjects should be asked for signs and symptoms suggestive of an immunerelated event. Subjects who develop an ECI thought to be immune-related should have additional testing to rule out other etiological causes. If lab results or symptoms indicated a possible immune-related ECI then additional testing should be performed to rule out other etiologic causes. If no other cause was found, then it is assumed to be immune-related.

# 7.2.3.3 Protocol-Specific Exceptions to Serious Adverse Event Reporting

Efficacy endpoints as outlined in this section will not be reported to the Sponsor as described in Section 7.2.3.

Specifically, the suspected/actual events covered in this exception include any event that is disease progression of the cancer under study.

# 7.2.4 Evaluating Adverse Events

An investigator who is a qualified physician will evaluate all adverse events according to the NCI Common Terminology for Adverse Events (CTCAE), version 4.0. Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded on the adverse event case report forms/worksheets.

All adverse events regardless of CTCAE grade must also be evaluated for seriousness.

For studies in which multiple agents are administered as part of a combination regimen, the investigator may attribute each adverse event causality to the combination regimen or to a single agent of the combination. In general, causality attribution should be assigned to the combination regimen (i.e., to all agents in the regimen). However, causality attribution may be assigned to a single agent if in the investigator's opinion, there is sufficient data to support full attribution of the adverse experience to the single agent.

**Protocol/Amendment No.:** 029-05

Table 16 **Evaluating Adverse Events** 

An investigator who is a qualified physician, will evaluate all adverse events as to:

| Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Sever or medically significant but not immediately life-threatening; hospitalization or prolongation or hospitalization indicated; disabiling; limiting self-care ADL. Grade 4 Life treatening consequences; urgent intervention indicated. Grade 5 Death related to AE As senous adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that: Results in death; or His life threatening; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an adverse event that, had it occurred in a more severe form, might have caused death;); or His life threatening; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an adverse event that, had it occurred in a more severe form, might have caused death;); or Hesults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or Hesults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or Hesults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or Hesults in or prolongs an existing inpatient hospitalization (hospitalization for an elective procedure to treat a pre-existing condition in a clinical condition that is diagnosed prior to the use of a Merck product and woversee when as one as errors adverse event (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours. Other important medical events that may not result in death, not be life threatening, or not used to diagnosed propropriate medical judgment, the event may jeopardize the | V4.0 CTCAE<br>Grading | | |
|---|---|---|---|
| Grade 4 Life threatening consequences; urgent intervention indicated. Grade 5 Death related to AE Seriousness A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that: **TResults in death; or **TResults in or proloages an existing impattent hospitalization in (so difficult and adverse event that, had it occurred in a more severe form, might have caused death); or **TResults in or proloages an existing impattent hospitalization is defined as an inpatitent admission, regardless of length of stay, even if the hospitalization is a precautionary measure for continued observation. (Note: Hospitalization for an elective procedure to treat a pre-existing condition that has not undersuced in the patient's medical history.); or **Ts a congenital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis); or **Is a new cancer (that is not a scolidated or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †) Duration | | Grade 2 | |
| Grade 4 Life threatening consequences; urgent intervention indicated. Grade 5 Death related to AE A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that: **Results in death;* or **Is life threatening;* or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an adverse event that, had it occurred in a more severe form, might have caused death), or **Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a presentation or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a presentation or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in a presentation or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or **Results in or prolongs an existing inpatient hospitalization in a nective procedure to treat a prevention of preparities of length of stant and nective procedure to the sample and prevention in the hospitalization in the sample in the patient is not a scondard and prevention of the study) (although not serious per ICH definition, is reportable to the Sponsor wi | | Grade 3 | |
| Seriousness A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that: **TResults in death, or **TResults in death, or **TResults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions), or **TResults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions), or **TResults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions), or **TResults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions), or **TResults in or prolongs an existing inpatient hospitalization (Note: Hospitalization is an inpatient admission, regardless of length of stay, even if the hospitalization is a precautionary measure for continued observation. (Note: Hospitalization for an elective procedure to treat a pre-existing condition that has not worsened is not a serious adverse event. A pre-existing condition that is diagnosed prior to the use of a Merck product and is documented in the patient's medical history.); or **TIS a congenital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis); or **Is a nowerdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. | | | |
| A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that: TResults in death; or | | | |
| Results in death; or | | | |
| Tis life threatening; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an adverse event that, had it occurred in a more severe form, might have caused death.); or TResults in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or TResults in or prolongs an existing inpatient hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay, even if the hospitalization is a precautionary measure for continued observation. (Note: Hospitalization for an elective procedure to treat a pre-existing condition that has not worsened is not a serious adverse event. A pre-existing condition is a clinical condition that is diagnosed prior to the use of a Merck product and is documented in the patient's medical history.); or Tis a none cancer (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements); or Tis an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threating, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a '1). Pouration Action taken Action taken Did the Adverse event cause the Sponsor's product to be discontinued? Relationship to Sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event | Seriousness | A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that: | |
| Action taken Acti | | 1 , . | |
| †Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or *Results in or prolongs an existing inpatient hospitalization (hospitalization is a precautionary measure for continued observation.) (Note: Hospitalization of an elective procedure to treat a pre-existing condition that has not worsened is not a serious adverse event. A pre-existing condition is a clinical condition that is diagnosed prior to the use of a Merck product and is documented in the patient's medical history.); or **Ts a congenital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis); or **Is a noverdose* (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Duration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Product | | †Is life threatening; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an | |
| Product | | | adverse event that, had it occurred in a more severe form, might have caused death.); or |
| hospitalization is a precautionary measure for continued observation. (Note: Hospitalization for an elective procedure to treat a pre-existing condition that has not worsened is not a serious adverse event. A pre-existing condition is a clinical condition that is diagnosed prior to the use of a Merck product and is documented in the patient's medical history.) or 7 Is a congenital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis);or Is a new cancer (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements); or Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Realtionship to Sponsor's product cause the Sponsor's product to be discontinued? Relationship to Both the Action taken and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to be discontinued? Did the Sponsor's product caused the adverse event will be provided by an entire to the sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be reta | | | |
| worsened is not a serious adverse event. A pre-existing condition is a clinical condition that is diagnosed prior to the use of a Merck product and is documented in the patient's medical history.); or Is a nower cancer (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements), or Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not a sociated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes itsed previously (designated above by a †). Duration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Action taken Product Belationship to Sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE for form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is the revidence that the subj | | | |
| the patient's medical history.); or Is a nongenital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis); or Is an overdose (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements); or Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Duration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to be discontinued? Product Did the Sponsor's product cause the Boponsor's product to be discontinued? Did the Sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an territable of the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measu | | | |
| Tis a congenital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis); or Is a new cancer (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements); or Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Duration Record the start and stop dates of the adverse event. If less than I day, indicate the appropriate length of time and units | | | |
| Is a new cancer (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours to meet certain local requirements); or | | | |
| requirements); or Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to be discontinued? Did the Sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event has adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product aused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Did the AE follow in a reasonable temporal sequence from administration of the Spons | | | |
| Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Duration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to be discontinued? | | | |
| overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Puration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to be discontinued? Did the Sponsor's product cause the Adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from adminis | | | |
| Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Product Relationship to Sponsor's Product Product Time Course Time Course Time Course Did the AE not reasonably explained by an a reasonably explained by an other etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). Duration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to use the Sponsor's product cause the sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure | | | |
| Suration Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units | | | |
| Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units Did the adverse event cause the Sponsor's product to be discontinued? Did the Sponsor's product cause the Adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course | | | |
| Action taken Relationship to Sponsor's Product Product Did the Sponsor's product cause the Sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | D | | |
| Relationship to Sponsor's product cause the adverse event? The determination of the likelihood that the Sponsor's product caused the adverse event will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| based upon the available information. The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | Froduct | | |
| The following components are to be used to assess the relationship between the Sponsor's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| and their respective elements (in number and/or intensity), the more likely the Sponsor's product caused the adverse event (AE): Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| Exposure Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | <b>Exposure</b> Is there evidence that the subject was actually exposed to the Sponsor's product such as: reliable history, acceptable compliance assessment ( | |
| Time Course Did the AE follow in a reasonable temporal sequence from administration of the Sponsor's product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | Time Course | |
| Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental | | | |
| | | Likely Cause | |
| | | - 3 | |

**Protocol/Amendment No.:** 029-05

| Relationship | The following components are to be used to assess the relationship between the test drug and the AE: (continued) | |
|---|---|---|
| to Sponsor's | Dechallenge | Was the Sponsor's product discontinued or dose/exposure/frequency reduced? |
| Product | | If yes, did the AE resolve or improve? |
| (continued) | | If yes, this is a positive dechallenge. If no, this is a negative dechallenge. |
| | | (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE resolved/improved despite continuation |
| | | of the Sponsor's product; or (3) the trial is a single-dose drug trial); or (4) Sponsor's product(s) is/are only used one time.) |
| | Rechallenge | Was the subject re-exposed to the Sponsor's product in this study? |
| | | If yes, did the AE recur or worsen? |
| | | If yes, this is a positive rechallenge. If no, this is a negative rechallenge. |
| | | (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) the trial is a single-dose drug trial); or |
| | | (3) Sponsor's product(s) is/are used only one time). |
| | | NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS AND WHICH MAY HAVE BEEN |
| | | CAUSED BY THE SPONSOR'S PRODUCT, OR IF REEXPOSURE TO THE SPONSOR'S PRODUCT POSES ADDITIONAL POTENTIAL |
| | | SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN ADVANCE BY THE SPONSOR |
| | C | CLINICAL DIRECTOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. |
| | Consistency | Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Sponsor's product or drug class |
| | with Trial<br>Treatment | pharmacology or toxicology? |
| | Profile | |
| The assessment of | | reported on the case report forms /worksheets by an investigator who is a qualified physician according to his/her best clinical judgment, including |
| consideration of th | | cported on the ease report forms / worksheets by an investigator who is a quantied physician according to institute best entitient judgment, including |
| Record one of the | | Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Sponsor's product relationship). |
| Trecord one or the | iono wing | ose the following scale of effectia as gardance (not an effectia must be present to be materially of a sponsor s produce relationship). |
| Yes, there is | a reasonable | There is evidence of exposure to the Sponsor's product. The temporal sequence of the AE onset relative to the administration of the Sponsor's |
| , | ponsor's product | product is reasonable. The AE is more likely explained by the Sponsor's product than by another cause. |
| relationship. | ponsor s product | product is reasonable. The File is more meety expanied by the Sponsor's product than by another cause. |
| T CHUICHSIN PV | | |
| No. there is n | ot a reasonable | Subject did not receive the Sponsor's product OR temporal sequence of the AE onset relative to administration of the Sponsor's product is not |
| , | ponsor's product | reasonable OR the AE is more likely explained by another cause than the Sponsor's product. (Also entered for a subject with overdose without |
| relationship | <u>.</u> | an associated AE.) |
| * | | |

Protocol/Amendment No.: 029-05

# 7.2.5 Sponsor Responsibility for Reporting Adverse Events

All Adverse Events will be reported to regulatory authorities, IRB/IECs and investigators in accordance with all applicable global laws and regulations.

#### 8.0 STATISTICAL ANALYSIS PLAN

This section outlines the statistical analysis strategy and procedures for the trial. If, after the trial has begun, changes are made to primary and/or key secondary hypotheses, or the statistical methods related to those hypotheses, then the protocol will be amended (consistent with ICH Guideline E-9). Changes to exploratory or other non-confirmatory analyses made after the protocol has been finalized, along with an explanation as to when and why they occurred, will be listed in the Clinical Study Report (CSR) for the trial. Post hoc exploratory analyses will be clearly identified in the CSR. No separate SAP will be issued for this trial.

#### 8.1 **Statistical Analysis Plan Summary**

This section contains a brief summary of the statistical analyses for this trial. Full detail is in the Statistical Analysis Plan (SAP) (Section 8.2).

#### 8.1.1 Part 1

The primary purpose of Part 1A of this trial is to investigate the safety and tolerability of MK-3475 in combination with PEG-IFN or IPI in adult subjects with MEL or RCC. The primary purpose of Part 1B of this trial is to further characterize the safety, tolerability and preliminary efficacy of the MK-3475 in combination with IPI in MEL subjects. Descriptive tables that summarize the number and percentage of subjects that experience adverse events as categorized in the NCI CTCAE Version 4 will be generated by dose level for the all subjects as treated population.

At the end of the Part 1A of the trial, the dose-response relationship, as the percentage of subjects experiencing at least one DLT in Cycle 1, for each dose level in the MK-3475+PEG-IFN combination will be estimated using a Bayesian pooling of adjacent violators analysis as outlined by Ji et al [84] using all DLT data from the trial with a conservative adjustment as described in Section 5.2.1.2. For the MK-3475+IPI combination, the percentage of subjects experiencing at least one DLT in Cycle 1 will be summarized for both Part 1A and 1B. The dose-response profile, along with other tolerability data, will be used to determine the recommended Phase 2 dose (RP2D) for MK-3475+PEG-IFN.

The Part 1A sample size of the trial depends primarily on clinical considerations rather than on statistical considerations. Specifically, the final number of subjects enrolled in the trial will depend on empirical safety (DLT) observations. However, it is estimated that a maximum of 25 subjects evaluable for safety and tolerability will be enrolled in Part 1A for the MK-3475+PEG-IFN combination, and a maximum of 18 subjects will be enrolled in Part 1A for the MK-3475+IPI combination.

The Part 1B sample size is driven by the expected number of PD-L1 negative subjects. Assuming that the prevalence of PD-L1 negative subjects is ~25%, then 90 subjects would be


**Protocol/Amendment No.:** 029-05

expected to provide ~22 subjects with PD-L1 negative MEL. If less than 22 PD-L1 negative MEL were enrolled in the MK-3475+IPI arm in Part 1A and 1B combined, enrollment will continue until at least 22 PD-L1 negative subjects are enrolled, up to a maximum of 150 subjects in Part 1B. Historical data has shown a response rate of 15% for PD-L1 negative MEL subjects treated with MK-3475 monotherapy. With 22 subjects with PD-L1 negative MEL, the study provides 80% power to rule out a lower bound on the ORR of 15% if the true ORR for MK-3475+IPI in PD-L1 negative subjects is 40%. If no less than 7 responses are observed, 22 PD-L1 negative subjects will allow excluding a 15% ORR lower bound of the 95% CI.

The Part 1C sample size provides adequate precision for the estimation of the ORR and the rate of grade 3-5 DRAEs for the regimens being assessed, with guidelines provided to assess whether the therapies maintain the ORR seen with pembrolizumab and standard dose ipilimumab, while substantially reducing the rate of grade 3-5 DRAEs.

# 8.2 Statistical Analysis Plan

## 8.2.1 Responsibility for Analyses/In-House Blinding

The statistical analysis of the data obtained from this trial will be the responsibility of the Clinical Biostatistics department of the SPONSOR.

This trial is open-label; the subject, the trial site personnel, and the Sponsor are not blinded to individual treatment group assignment for Part 1 of the study. The Clinical Biostatistics department will generate the randomized allocation schedule(s) for study treatment assignment. Subjects in Part 1A and 1C will be randomly assigned to treatment combination (pembrolizumab + PEG-IFN or pembrolizumab + IPI) if both combinations are open for enrollment.

#### 8.2.2 Hypotheses/Estimation

Objectives and hypotheses of the trial are stated in Section 3.

#### 8.2.3 Analysis Endpoints

Efficacy and safety endpoints that will be evaluated for within- and/or between-treatment differences are listed below, followed by the descriptions of the derivations of selected endpoints.

#### 8.2.3.1 Safety Endpoints

07W8HB

Safety measurements of interest are described in Section 4.2.3.1.

**Part 1A**: The primary Part 1A safety endpoint is the DLT rate.

<u>Part 1B and 1C</u>: For Part 1B and Part 1C, all ECIs listed in the irAE guidance as well as  $Grade \ge 2$  Depression are prespecified as events of interest (Tier-1 events).

7-Nov-2017

Protocol/Amendment No.: 029-05

# 8.2.3.2 Efficacy Endpoints

# **Primary Efficacy Endpoint**

The primary efficacy endpoint will be the **ORR** defined as the proportion of the subjects in the analysis population who have best response as CR or partial response (PR). Responses are based on central independent review using RECIST 1.1.

**Ordinal response score,** per RECIST 1.1, defined as the best overall response calculated as the following:

1=Complete Response

2=Very Good Partial Response [>60% tumor reduction]

3=Moderate Partial Response [>30% - ≤60% tumor reduction]

4=Stable Disease

5=Progressive Disease

Ordinal response scores are based on central independent review using RECIST 1.1.

Additional secondary efficacy endpoints include PFS, defined as the time from randomization to the first documented disease progression (based on central independent review using RECIST 1.1) or death due to any cause, whichever occurs first, duration of response among subjects who achieve a best response as CR or PR per RECIST 1.1 and OS. Pharmacokinetic endpoints include area under the curve (AUC), Cmax, and clearance.

# 8.2.4 Analysis Populations

#### 8.2.4.1 Efficacy Analysis Populations

ORR, DOR, PFS, and OS analyses will be restricted to those patients with measurable disease at baseline based on central independent review.

# 8.2.4.2 Safety Analysis Populations

For Part 1A safety analyses related to DLT rate, the DLT evaluable population will be used. The DLT evaluable population consists of all DLT evaluable subjects. In order to be considered evaluable, the subject must complete the first cycle of combination therapy or discontinue from the trial due to a DRAE. Subjects who discontinue prematurely due to a non drug-related cause are not included in the DLT evaluable population (refer to Section 5.2.1.2.2 for detailed DLT replacement criteria).

For all other Part 1 safety analyses, the APaT population will be used for the analysis of safety data. The APaT population consists of all randomized subjects who received at least one dose of study treatment. Subjects will be included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data using the APaT population. For most subjects, this will be the treatment group to which they are randomized. Subjects who take incorrect study treatment for the entire treatment period will be included in

**Protocol/Amendment No.:** 029-05

the treatment group corresponding to the study treatment actually received. At least one laboratory or vital sign measurement obtained subsequent to at least one dose of trial treatment is required for inclusion in the analysis of each specific parameter. To assess change from baseline, a baseline measurement is also required.

Details on the approach to handling missing data for safety analyses are provided in Section 8.2.5 Statistical Methods.

#### 8.2.5 Statistical Methods

## **8.2.5.1** Statistical Methods for Efficacy Analyses

# 8.2.5.1.1 Progression-free Survival (PFS)

The non-parametric Kaplan-Meier method will be used to estimate the PFS curve for each treatment group in the Part 1B and 1C of the trial.

# 8.2.5.1.2 Overall Survival (OS)

The Kaplan-Meier method will be used to estimate the OS curve in each treatment group.

#### 8.2.5.1.3 Objective Response Rate (ORR)

Exact 90% confidence intervals for ORR will be calculated for the true ORR for the treatments investigated in Part 1C.

#### 8.2.5.1.4 Ordinal Response Score

The frequency distribution of the ordinal response score will be estimated by calculating number of patients in each category divided by the total number of patients in the FAS population. Subjects with missing data will be considered non-responders.

#### 8.2.5.1.5 Duration of Response (DOR)

If sample size permits, duration of response will be summarized descriptively using Kaplan-Meier curves medians and quartiles. Only the subset of subjects who show a CR or PR will be included in this analysis.

#### **8.2.5.1.6** Pharmacokinetic Parameters

Pharmacokinetic parameters will be summarized using descriptive statistics.

Table 17 summarizes the analysis strategy for primary and secondary efficacy endpoints.

**Protocol/Amendment No.:** 029-05

Table 17 Summary of Analysis Strategy for Key Efficacy Endpoints

| Endpoint/Variable<br>(Description, Time Point) | Primary vs.<br>Supportive<br>Approach <sup>†</sup> | Statistical Method | Analysis<br>Population | Missing Data<br>Approach |
|---|---|---|---|---|
| Primary Hypothesis: | | | | |
| ORR (Part 1C) | P | Exact 90% confidence intervals for true ORR | FAS | Subjects with<br>missing data are<br>considered as<br>non-responders |
| Secondary Objectives: | | | | |
| DOR | P | Summary statistics<br>using Kaplan-Meier<br>method | All responders | Non-responders<br>are excluded in<br>analysis |
| ORR (Part 1B) | P | Exact test of binomial parameter | FAS | Subjects with<br>missing data are<br>considered as<br>non-responders |
| PFS | P | Estimation: Kaplan-Meier method for PFS curve estimation in each treatment group | ITT | Censored at last disease assessment |
| OS | P | Summary statistics<br>using Kaplan-Meier<br>method | ITT | Censored at last date known alive |
| PK | P | Descriptive Statistics | All treated subjects | Missing data excluded from analysis |
| Ordinal Response Score (Part 1B and 1C) | P | Descriptive Statistics | FAS | Subjects with<br>missing data are<br>considered as<br>non-responders |

# **8.2.5.2** Statistical Methods for Safety Analyses

Safety and tolerability will be assessed by clinical review of all relevant parameters including AEs, SAEs, laboratory tests, vital signs, ECG measurements and physical examinations.

#### Part 1A

DLTs will be listed. Adverse experiences will be summarized as counts and frequencies for each dose level. Laboratory assessments, vital signs, and other safety endpoints will be summarized as appropriate.

ECIs of a potential immunologic etiology may be defined as an adverse event of unknown etiology, associated with drug exposure and is consistent with an immune phenomenon. irAEs may be predicted based on the nature of pembrolizumab and IPI, their mechanism of action, and reported experience with immunotherapies that have a similar mechanism of

**Protocol/Amendment No.:** 029-05

action. Special attention should be paid to AEs that may be suggestive of potential irAEs. An irAE can occur shortly after the first dose or several months after the last dose of treatment.

# Part 1B and Part 1C

All ECIs listed in irAE guidance and Tier 2 or 3 safety parameters listed in Table 18 will be described via inferential and descriptive statistics.

Table 18 Analysis Strategy for Safety Parameters

| Safety<br>Tier | Safety Endpoint <sup>†</sup> | p-Value | 95% CI for<br>Treatment<br>Comparison | Descriptive<br>Statistics |
|---|---|---|---|---|
| m: 1 | | 77 | *** | 77 |
| Tier 1 | All ECIs in irAE guidance | X | X | X |
| | Grade $\geq 2$ depression | X | X | X |
| | Any AE | | X | X |
| Tier 2 | Any Serious AE | | X | X |
| | Any Grade 3-5 AE | | X | X |
| | Onset and Duration of First Grade 3-5 AE | | X | X |
| | Any Drug-Related AE | | X | X |
| | Any Serious and Drug-Related AE | | X | X |
| | Any Grade3-5 and Drug-Related AE | | X | X |
| | Dose Modification due to AE | | X | X |
| | Discontinuation due to AE | | X | X |
| | Death | | X | X |
| | Specific AEs, SOCs, or PDLCs‡ (incidence ≥4/1% of subjects in one of the treatment groups) | | X | X |
| Tier 3 | Specific AEs, SOCs or PDLCs‡ (incidence <4/1% of subjects in all of the treatment groups) | | | X |
| _ | Change from Baseline Results (Labs, ECGs, Vital Signs) | | | X |

Adverse Experience references refer to both Clinical and Laboratory AEs.

For all subjects enrolled at the RP2D for pembrolizumab + PEG-IFN and Phase 2 Dose for pembrolizumab + IPI in Part 1B, the incidence of Grade 3-5 adverse experiences will be compared between pembrolizumab + IPI and pembrolizumab + PEG-IFN using the Miettinen and Nurminen method [85].

#### 8.2.5.3 Summaries of Baseline Characteristics, Demographics, and Other Analyses

Demographic variables (e.g., age, gender), baseline characteristics, primary and secondary diagnoses, and prior and concomitant therapies will be summarized by descriptive statistics

Includes only those endpoints not pre-specified as Tier 1 or not already pre-specified as Tier-2 endpoints. Note: SOC=System Organ Class; PDLC=Pre-Defined Limit of Change; X = results will be provided.

Protocol/Amendment No.: 029-05

or categorical tables. The number and percentage of subjects screened, randomized, the primary reasons for screening failure, and the primary reason for discontinuation will be displayed.

For Part 1A RCC subjects, individual efficacy listing and/or descriptive statistics (as data permits) will be summarized to evaluate the efficacy for pembrolizumab + IPI and pembrolizumab + PEG-IFN using the same efficacy endpoints as described in Section 8.2.5.1.

# 8.2.6 Multiplicity

No adjustment will be made for multiplicity in Part 1.

# **8.2.7** Sample Size and Power Calculations

#### 8.2.7.1 Part 1

The Part 1A sample size of the trial depends primarily on clinical considerations rather than on statistical considerations. Specifically, the final number of subjects enrolled in the trial will depend on empirical safety (DLT) observations. However, it is estimated that a maximum of 25 subjects evaluable for safety and tolerability will be enrolled in Part 1A for the pembrolizumab + PEG-IFN combination, and a maximum of 18 subjects will be enrolled in Part 1A for the pembrolizumab + IPI combination.

The Part 1B sample size is driven by the expected number of PD-L1 negative subjects. Assuming that the prevalence of PD-L1 negative subjects is ~25%, then 90 subjects would be expected to provide ~22 subjects with PD-L1 negative MEL. If less than 22 PD-L1 negative MEL were enrolled in the pembrolizumab + IPI arm in Part 1A and 1B combined, enrollment will continue until at least 22 PD-L1 negative subjects are enrolled, up to a maximum of 150 subjects in Part 1B. Historical data has shown a response rate of 15% for PD-L1 negative MEL subjects treated with pembrolizumab monotherapy. With 22 subjects with PD-L1 negative MEL, the study provides 80% power to rule out a lower bound on the ORR of 15% if the true ORR for pembrolizumab + IPI in PD-L1 negative subjects is 40%. With 7 or more responses out of 22 PD-L1 negative patients, a 95% CI would exclude a 15% or lower ORR.

The Part 1C sample size is designed to provide adequate precision for the estimation of the true rate of Grade 3-5 DRAEs and the ORR for the treatments evaluated. The sample size for part 1C will be 100 patients (50 patients per treatment arm).

With 50 patients per treatment arm, a 95% upper bound for the true rate of Grade 3-5 DRAE would be:

**Protocol/Amendment No.:** 029-05

| Observed number of | 95% upper bound for true |
|-----------------------|--------------------------|
| patients experiencing | rate of |
| Grade 3-5 DRAEs | Grade 3-5 DRAEs |
| 10 (20%) | 32% |
| 12 (24%) | 36% |
| 13 (26%) | 38% |

With 50 patients per treatment group, an observed rate of Grade 3-5 DRAEs of 26% or less would suggest a meaningful reduction in the rate of DRAEs compared to other combinations of IPI and anti-PD-1 inhibitors (pembrolizumab or nivolumab), as the 90% upper bound for the true rate of Grade 3-5 DRAEs excludes 40%.

With 50 patients per treatment, a 95% upper bound for the true ORR would be:

| Observed number of patients experiencing an objective response | 95% lower<br>bound for true<br>ORR | 95% upper bound for true ORR |
|---|---|---|
| 20 (40%) | 28% | 53% |
| 22 (44%) | 32% | 57% |
| 24 (48%) | 36% | 60% |

With 50 patients per treatment group, an observed ORR of 48% or more would suggest that the combination ORR was consistent with that of other combinations of IPI and anti-PD-1 inhibitors (pembrolizumab or nivolumab) (as the 90% CI excludes 35%).

# 8.2.8 Interim Analyses

Part 1A and 1B will be considered complete when all enrolled subjects are a minimum of 24 weeks post initial trial treatment administration. At this point a database lock may occur to allow analysis of the data. Part 1C will be considered complete for publication purposes when all enrolled subjects are a minimum of 72 weeks post initial treatment administration. At this point database lock may occur to allow analysis of the data. If the study remains open, additional analyses of the data can occur to monitor the study and report on later subject follow-up.

# **8.2.9** Compliance (Medication Adherence)

Drug accountability data for trial treatment will be collected during the trial. Percent compliance with drug administration will be calculated for each subject for pembrolizumab, IPI, and IFN separately.

Protocol/Amendment No.: 029-05

Percent compliance will be calculated as following:

For IFN administered once a week, "Number of Doses that Should be Taken" will be calculated as 1 plus the number (integer) of 1-week intervals that fit between the date of the first dose and the date of the last dose. For pembrolizumab and IPI administered q3w "Number of Doses Should be Taken" will be calculated as 1 plus the number (integer) of 3-week intervals that fit between the date of the first dose and the date of the last dose. For IPI administered g6w and g12w "Number of Doses Should be Taken" will be calculated as 1 plus the number (integer) of 6-week or 12-week intervals, respectively, that fit between the date of the first dose and the date of the last dose.

# 8.2.10 Extent of Exposure

For a pembrolizumab regimen, a subject's extent of exposure to pembrolizumab is defined as the total number of doses of pembrolizumab the subject received. A subject's exposure to a dose of IPI or IFN is defined as the total number of days on therapy for that dose.

Summary statistics may be provided on Extent of Exposure for the APaT population in Parts 1B and 1C.

# 9.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL **SUPPLIES**

# 9.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Clinical Supplies utilized in the trial are:

**Product Descriptions** Table 19

| Product Name & Potency | |
|---|---|
| | Dosage Form |
| pembrolizumab 100 mg/4 mL | Solution for Infusion |
| Pegylated Interferon alfa-2b 300 mcg | Lyophilized Powder for Injection |
| Ipilimumab 50 mg and 200 mg Solution for Infusion | |
| NOTE: The investigator will be responsible for providing the following items: syringes, alcohol swabs, and sterile water for injection, USP (vial or ampule). | |

**Protocol/Amendment No.:** 029-05

Pegylated Interferon alfa-2b and IPI will be provided centrally by the Sponsor or locally by the trial site, subsidiary or designee, depending on local country operational or regulatory requirements.

For any commercially available product that is provided by the trial site, subsidiary or designee, every attempt will be made to source these supplies from a single lot/batch number. The trial site will be responsible for recording the lot number, manufacturer and expiry date of any locally purchased product. The trial site is responsible to record the lot number, manufacturer and expiry date for any locally purchased product as per local guidelines unless otherwise instructed by the Sponsor. However, as any locally sourced combination therapies specified in Table 19 of the protocol are approved drugs in the US, investigational sites participating in this trial that are located in the US are not required to collect information regarding the source (manufacturer/lot/expiry date) on trial documentation. Drug accountability and manufacturer information will be retained with the hospital pharmacy at the clinical site.

#### 9.2 **Packaging and Labeling Information**

Clinical supplies will be affixed with a clinical label in accordance with regulatory requirements.

Subjects will receive open-label pembrolizumab 100 mg/ 4mL vials, Pegylated Interferon alfa-2b 300 mcg kits, and IPI 50 mg and 200 mg kits for dosing Parts 1A, 1B, and 1C subjects.

#### 9.3 **Clinical Supplies Disclosure**

This trial is open-label; therefore, the subject, the trial site personnel, the Sponsor and/or designee are not blinded. Treatment (name, strength or potency) is included in the label text; random code/disclosure envelopes or lists are not provided.

#### 9.4 **Storage and Handling Requirements**

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

#### 9.5 **Returns and Reconciliation**

The investigator is responsible for keeping accurate records of the clinical supplies received from the Sponsor or designee, the amount dispensed to and returned by the subjects and the amount remaining at the conclusion of the trial.

For all trial sites, the local country Sponsor personnel or designee will provide appropriate documentation that must be completed for drug accountability and return.


**Protocol/Amendment No.:** 029-05

#### **Standard Policies**

Trial site personnel will have access to a central electronic randomization system (IVRS/IWRS system) to allocate subjects, to assign treatment to subjects and to manage the distribution of clinical supplies. Each person accessing the IVRS system must be assigned an individual unique PIN. They must use only their assigned PIN to access the system, and they must not share their assigned PIN with anyone.

### 10.0 ADMINISTRATIVE AND REGULATORY DETAILS

## **10.1** Confidentiality

# 10.1.1 Confidentiality of Data

By signing this protocol, the investigator affirms to the Sponsor that information furnished to the investigator by the Sponsor will be maintained in confidence, and such information will be divulged to the institutional review board, ethics review committee (IRB/ERC) or similar or expert committee; affiliated institution and employees, only under an appropriate understanding of confidentiality with such board or committee, affiliated institution and employees. Data generated by this trial will be considered confidential by the investigator, except to the extent that it is included in a publication as provided in the Publications section of this protocol.

# 10.1.2 Confidentiality of Subject Records

By signing this protocol, the investigator agrees that the Sponsor (or Sponsor representative), IRB/ERC, or regulatory authority representatives may consult and/or copy trial documents in order to verify worksheet/case report form data. By signing the consent form, the subject agrees to this process. If trial documents will be photocopied during the process of verifying worksheet/case report form information, the subject will be identified by unique code only; full names/initials will be masked prior to transmission to the Sponsor.

By signing this protocol, the investigator agrees to treat all subject data used and disclosed in connection with this trial in accordance with all applicable privacy laws, rules and regulations.

#### **10.1.3** Confidentiality of Investigator Information

By signing this protocol, the investigator recognizes that certain personal identifying information with respect to the investigator, and all subinvestigators and trial site personnel, may be used and disclosed for trial management purposes, as part of a regulatory submissions, and as required by law. This information may include:

- 1. name, address, telephone number and e-mail address;
- 2. hospital or clinic address and telephone number;
- 3. curriculum vitae or other summary of qualifications and credentials; and
- 4. other professional documentation.


**Protocol/Amendment No.:** 029-05

Consistent with the purposes described above, this information may be transmitted to the Sponsor, and subsidiaries, affiliates and agents of the Sponsor, in your country and other countries, including countries that do not have laws protecting such information. Additionally, the investigator's name and business contact information may be included when reporting certain serious adverse events to regulatory authorities or to other investigators. By signing this protocol, the investigator expressly consents to these uses and disclosures.

If this is a multicenter trial, in order to facilitate contact between investigators, the Sponsor may share an investigator's name and contact information with other participating investigators upon request.

# 10.1.4 Confidentiality of IRB/IEC Information

The Sponsor is required to record the name and address of each IRB/IEC member that reviews and approves this trial. The Sponsor is also required to document that each IRB/IEC meets regulatory and ICH GCP requirements by requesting and maintaining records of the names and qualifications of the IRB/IEC members and to make these records available for regulatory agency review upon request by those agencies.

#### 10.2 Compliance with Financial Disclosure Requirements

Financial Disclosure requirements are outlined in the US Food and Drug Administration Regulations, Financial Disclosure by Clinical Investigators (21 CFR Part 54). It is the Sponsor's responsibility to determine, based on these regulations, whether a request for Financial Disclosure information is required. It is the investigator's/subinvestigator's responsibility to comply with any such request.

The investigator/subinvestigator(s) agree, if requested by the Sponsor in accordance with 21 CFR Part 54, to provide his/her financial interests in and/or arrangements with the Sponsor to allow for the submission of complete and accurate certification and disclosure statements. The investigator/subinvestigator(s) further agree to provide this information on a Certification/Disclosure Form, commonly known as a financial disclosure form, provided by the Sponsor or through a secure password-protected electronic portal provided by the Sponsor. The investigator/subinvestigator(s) also consent to the transmission of this information to the Sponsor in the United States for these purposes. This may involve the transmission of information to countries that do not have laws protecting personal data.

#### 10.3 Compliance with Law, Audit and Debarment

By signing this protocol, the investigator agrees to conduct the trial in an efficient and diligent manner and in conformance with this protocol; generally accepted standards of Good Clinical Practice (e.g., International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice: Consolidated Guideline and other generally accepted standards of good clinical practice); and all applicable federal, state and local laws, rules and regulations relating to the conduct of the clinical trial.

MK-3475-029-05 Final Protocol 7-Nov-2017

Protocol/Amendment No.: 029-05

The Code of Conduct, a collection of goals and considerations that govern the ethical and scientific conduct of clinical investigations sponsored by Merck, is provided in Section 12.1 -Merck Code of Conduct for Clinical Trials.

The investigator also agrees to allow monitoring, audits, IRB/ERC review and regulatory authority inspection of trial-related documents and procedures and provide for direct access to all trial-related source data and documents.

The investigator agrees not to seek reimbursement from subjects, their insurance providers or from government programs for procedures included as part of the trial reimbursed to the investigator by the Sponsor.

The investigator shall prepare and maintain complete and accurate trial documentation in compliance with Good Clinical Practice standards and applicable federal, state and local laws, rules and regulations; and, for each subject participating in the trial, provide all data, and, upon completion or termination of the clinical trial, submit any other reports to the Sponsor as required by this protocol or as otherwise required pursuant to any agreement with the Sponsor.

Trial documentation will be promptly and fully disclosed to the Sponsor by the investigator upon request and also shall be made available at the trial site upon request for inspection. copying, review and audit at reasonable times by representatives of the Sponsor or any regulatory authorities. The investigator agrees to promptly take any reasonable steps that are requested by the Sponsor as a result of an audit to cure deficiencies in the trial documentation and worksheets/case report forms.

The investigator must maintain copies of all documentation and records relating to the conduct of the trial in compliance with all applicable legal and regulatory requirements. This documentation includes, but is not limited to, the protocol, worksheets/case report forms, advertising for subject participation, adverse event reports, subject source data, correspondence with regulatory authorities and IRBs/ERCs, consent forms, investigator's curricula vitae, monitor visit logs, laboratory reference ranges, laboratory certification or quality control procedures and laboratory director curriculum vitae. By signing this protocol, the investigator agrees that documentation shall be retained until at least 2 years after the last approval of a marketing application in an ICH region or until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. Because the clinical development and marketing application process is variable, it is anticipated that the retention period can be up to 15 years or longer after protocol database lock. The Sponsor will determine the minimum retention period and notify the investigator when documents may be destroyed. The sponsor also recognizes that documents may need to be retained for a longer period if required by local regulatory requirements. All trial documents shall be made available if required by relevant regulatory authorities. The investigator must consult with and obtain written approval by the Sponsor prior to discarding trial and/or subject files.

**Protocol/Amendment No.:** 029-05

ICH Good Clinical Practice guidelines recommend that the investigator inform the subject's primary physician about the subject's participation in the trial if the subject has a primary physician and if the subject agrees to the primary physician being informed.

The investigator will promptly inform the Sponsor of any regulatory authority inspection conducted for this trial.

Persons debarred from conducting or working on clinical trials by any court or regulatory authority will not be allowed to conduct or work on this Sponsor's trials. The investigator will immediately disclose in writing to the Sponsor if any person who is involved in conducting the trial is debarred or if any proceeding for debarment is pending or, to the best of the investigator's knowledge, threatened.

In the event the Sponsor prematurely terminates a particular trial site, the Sponsor will promptly notify that trial site's IRB/IEC.

According to European legislation, a Sponsor must designate an overall coordinating investigator for a multi-center trial (including multinational). When more than one trial site is open in an EU country, Merck, as the Sponsor, will designate, per country, a national principal coordinator (Protocol CI), responsible for coordinating the work of the principal investigators at the different trial sites in that Member State, according to national regulations. For a single-center trial, the Protocol CI is the principal investigator. In addition, the Sponsor must designate a principal or coordinating investigator to review the trial report that summarizes the trial results and confirm that, to the best of his/her knowledge, the report accurately describes the conduct and results of the trial [Clinical Study Report (CSR) CI]. The Sponsor may consider one or more factors in the selection of the individual to serve as the Protocol CI and or CSR CI (e.g., availability of the CI during the anticipated review process, thorough understanding of clinical trial methods, appropriate enrollment of subject cohort, timely achievement of trial milestones). The Protocol CI must be a participating trial investigator.

#### 10.4 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to the Clinical Trials Data Bank, http://www.clinicaltrials.gov. Merck, as Sponsor of this trial, will review this protocol and submit the information necessary to fulfill these requirements. Merck entries are not limited to FDAMA/FDAAA mandated trials. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

By signing this protocol, the investigator acknowledges that the statutory obligations under FDAMA/FDAAA are that of the Sponsor and agrees not to submit any information about this trial or its results to the Clinical Trials Data Bank.

MK-3475-029-05 Final Protocol

**Protocol/Amendment No.:** 029-05

# 10.5 Quality Management System

By signing this protocol, the Sponsor agrees to be responsible for implementing and maintaining a quality management system with written development procedures and functional area standard operating procedures (SOPs) to ensure that trials are conducted and data are generated, documented, and reported in compliance with the protocol, accepted standards of Good Clinical Practice, and all applicable federal, state, and local laws, rules and regulations relating to the conduct of the clinical trial.

#### 10.6 Data Management

The investigator or qualified designee is responsible for recording and verifying the accuracy of subject data. By signing this protocol, the investigator acknowledges that his/her electronic signature is the legally binding equivalent of a written signature. By entering his/her electronic signature, the investigator confirms that all recorded data have been verified as accurate.

Detailed information regarding Data Management procedures for this protocol will be provided separately.

#### 10.7 Publications

This trial is intended for publication, even if terminated prematurely. Publication may include any or all of the following: posting of a synopsis online, abstract and/or presentation at a scientific conference, or publication of a full manuscript. The Sponsor will work with the authors to submit a manuscript describing trial results within 12 months after the last data become available, which may take up to several months after the last subject visit in some cases such as vaccine trials. However, manuscript submission timelines may be extended on OTC trials. For trials intended for pediatric-related regulatory filings, the investigator agrees to delay publication of the trial results until the Sponsor notifies the investigator that all relevant regulatory authority decisions on the trial drug have been made with regard to pediatric-related regulatory filings. Merck will post a synopsis of trial results for approved products on www.clinicaltrials.gov by 12 months after the last subject's last visit for the primary outcome, 12 months after the decision to discontinue development, or product marketing (dispensed, administered, delivered or promoted), whichever is later.

These timelines may be extended for products that are not yet marketed, if additional time is needed for analysis, to protect intellectual property, or to comply with confidentiality agreements with other parties. Authors of the primary results manuscript will be provided the complete results from the Clinical Study Report, subject to the confidentiality agreement. When a manuscript is submitted to a biomedical journal, the Sponsor's policy is to also include the protocol and statistical analysis plan to facilitate the peer and editorial review of the manuscript. If the manuscript is subsequently accepted for publication, the Sponsor will allow the journal, if it so desires, to post on its website the key sections of the protocol that are relevant to evaluating the trial, specifically those sections describing the trial objectives and hypotheses, the subject inclusion and exclusion criteria, the trial design and procedures,

**Protocol/Amendment No.:** 029-05

the efficacy and safety measures, the statistical analysis plan, and any amendments relating to those sections. The Sponsor reserves the right to redact proprietary information.

For multicenter trials, subsequent to the multicenter publication (or after public disclosure of the results online at www.clinicaltrials.gov if a multicenter manuscript is not planned), an investigator and his/her colleagues may publish their data independently. In most cases, publication of individual trial site data does not add value to complete multicenter results, due to statistical concerns. In rare cases, publication of single trial site data prior to the main paper may be of value. Limitations of single trial site observations in a multicenter trial should always be described in such a manuscript.

Authorship credit should be based on 1) substantial contributions to conception and design, or acquisition of data, or analysis and interpretation of data; 2) drafting the article or revising it critically for important intellectual content; and 3) final approval of the version to be published. Authors must meet conditions 1, 2 and 3. Significant contributions to trial execution may also be taken into account to determine authorship, provided that contributions have also been made to all three of the preceding authorship criteria. Although publication planning may begin before conducting the trial, final decisions on authorship and the order of authors' names will be made based on participation and actual contributions to the trial and writing, as discussed above. The first author is responsible for defending the integrity of the data, method(s) of data analysis and the scientific content of the manuscript.

The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

#### 11.0 LIST OF REFERENCES

- [1] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer 2009;45:228-47.
- [2] Disis ML. Immune regulation of cancer. J Clin Oncol 2010;28(29):4531-8.
- [3] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, et al. Tumorassociated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med 2002;8(8):793-800.
- [4] Sharpe AH, Freeman GJ. The B7-CD28 superfamily. Nat Rev Immunol 2002;2(2):116-26.
- [5] Brown JA, Dorfman DM, Ma F-R, Sullivan EL, Munoz O, Wood CR, et al. Blockade of programmed death-1 ligands on dendritic cells enhances T cell activation and cytokine production. J Immunol 2003;170(3):1257-66.

**Protocol/Amendment No.:** 029-05

[6] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev 2010;236:219-42.

- [7] Thompson RH, Dong H, Lohse CM, Leibovich BC, Blute ML, Cheville JC, et al. PD-1 is expressed by tumor-infiltrating immune cells and is associated with poor outcome for patients with renal cell carcinoma. Clin Cancer Res 2007;13(6):1757-61.
- [8] Sasaki A, Tanaka F, Mimori K, Inoue H, Kai S, Shibata K, et al. Prognostic value of tumor-infiltrating FOXP3+ regulatory T cells in patients with hepatocellular carcinoma. EJSO 2008;34:173-9.
- [9] Shen Z, Zhou S, Wang Y, Li R, Zhong C, Liang C, et al. Higher intratumoral infiltrated Foxp3+ Treg numbers and Foxp3+/CD8+ ratio are associated with adverse prognosis in resectable gastric cancer. J Cancer Res Clin Oncol 2010;136:1585-95.
- [10] Talmadge JE, Donkor M, Scholar E. Inflammatory cell infiltration of tumors: Jekyll or Hyde. Cancer Metastasis Rev 2007;26(3-4):373-400.
- [11] Usubütün A, Ayhan A, Uygur MC, Özen H, Toklu C, Ruacan S. Prognostic factors in renal cell carcinoma. J Exp Clin Cancer Res 1998;17(1):77-81.
- [12] Al-Shibli KI, Donnem T, Al-Saad S, Persson M, Bremnes RM, Busund L-T. Prognostic effect of epithelial and stromal lymphocyte infiltration in non-small cell lung cancer. Clin Cancer Res 2008;14(16):5220-7.
- [13] Deschoolmeester V, Baay M, Van Marck E, Weyler J, Vermeulen P, Lardon F, et al. Tumor infiltrating lymphocytes: an intriguing player in the survival of colorectal cancer patients. BMC Immunol 2010;11:19.
- [14] Diez M, Pollán M, Enriquez JM, Dominguez P, Santana A, Tobaruela E, et al. Histopathologic prognostic score in colorectal adenocarcinomas. Anticancer Res 1998;18(1B):689-94.
- [15] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pagès C, et al. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science 2006;313(5795):1960-4.
- [16] Hiraoka N. Tumor-infiltrating lymphocytes and hepatocellular carcinoma: molecular biology. Int J Clin Oncol 2010;15(6):544-51.
- [17] Nobili C, Degrate L, Caprotti R, Franciosi C, Leone BE, Trezzi R, et al. Prolonged survival of a patient affected by pancreatic adenocarcinoma with massive lymphocyte and dendritic cell infiltration after interleukin-2 immunotherapy. Report of a case. Tumori 2008;94(3):426-30.

Protocol/Amendment No.: 029-05

[18] Hodi FS. Dranoff G. The biologic importance of tumor-infiltrating lymphocytes. J Cutan Pathol 2010;37(Suppl 1):48-53.

- [19] Kloor M. Lymphocyte infiltration and prognosis in colorectal cancer. Lancet Oncol. 2009 Sep;10(9):840-1.
- [20] Hillen F, Baeten CIM, van de Winkel A, Creytens D, van der Schaft DWJ, Winnepenninckx V, et al. Leukocyte infiltration and tumor cell plasticity are parameters of aggressiveness in primary cutaneous melanoma. Cancer Immunol Immunother 2008;57(1):97-106.
- [21] Lee HE, Chae SW, Lee YJ, Kim MA, Lee HS, Lee BL, et al. Prognostic implications of type and density of tumour-infiltrating lymphocytes in gastric cancer. Br J Cancer 2008;99(10):1704-11.
- [22] Leffers N, Gooden MJM, de Jong RA, Hoogeboom B-N, ten Hoor KA, Hollema H, et al. Prognostic significance of tumor-infiltrating T-lymphocytes in primary and metastatic lesions of advanced stage ovarian cancer. Cancer Immunol Immunother 2009;58(3):449-59.
- [23] Nishimura H, Honjo T, Minato N. Facilitation of beta selection and modification of positive selection in the thymus of PD-1-deficient mice. J Exp Med. 2000 Mar 6;191(5):891-8.
- [24] Oble DA, Loewe R, Yu P, Mihm MC Jr. Focus on TILs: prognostic significance of tumor infiltrating lymphocytes in human melanoma. Cancer Immun. 2009 Apr 2;9:3.
- [25] Pölcher M, Braun M, Friedrichs N, Rudlowski C, Bercht E, Fimmers R, et al. Foxp3(+) cell infiltration and granzyme B(+)/Foxp3(+) cell ratio are associated with outcome in neoadjuvant chemotherapy-treated ovarian carcinoma. Cancer Immunol Immunother 2010;59(6):909-19.
- Suzuki H, Chikazawa N, Tasaka T, Wada J, Yamasaki A, Kitaura Y, et al. [26] Intratumoral CD8+ T/FOXP3+ cell ratio is a predictive marker for survival in patients with colorectal cancer. Cancer Immunol Immunother 2010;59:653-61.
- [27] Chew V, Tow C, Teo M, Wong HL, Chan J, Gehring A, et al. Inflammatory tumor microenvironment is associated with superior survival in hepatocellular carcinoma patients. J Hepatol 2010;52:370-9.
- [28] Liotta F, Gacci M, Frosali F, Querci V, Vittori G, Lapini A, et al. Frequency of regulatory T cells in peripheral blood and in tumour-infiltrating lymphocytes correlates with poor prognosis in renal cell carcinoma. BJU Int 2011;107(9):1500-6.

**Protocol/Amendment No.:** 029-05

[29] Hamid O, Puzanov I, Dummer R, Schachter J, Daud A, Schadendorf D, et al. Melanoma and other skin tumours: Final overall survival for KEYNOTE-002: pembrolizumab (pembro) versus investigator-choice chemotherapy (chemo) for ipilimumab (ipi)-refractory melanoma [abstract]. Ann Oncol. 2016;27 Suppl 6. Abstract no. 11070.

- [30] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, et al. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32.
- [31] U.S. Prescribing Information: KEYTRUDA (Pembrolizumab) Injection, for intravenous use: 2014.
- [32] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, et al. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28.
- [33] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, et al. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18.
- [34] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol 2005;23:515-48.
- [35] Eggermont AMM, Suciu S, Santinami M, Testori A, Kruit WH, Marsden J, et al. Adjuvant therapy with pegylated interferon alfa-2b versus observation alone in resected stage III melanoma: final results of EORTC 18991, a randomised phase III trial. Lancet 2008;372:117-26.
- [36] Dummer R, Garbe C, Thompson JA, Eggermont AM, Yoo K, Maier T, Bergstrom B. Randomized dose-escalation study evaluating peginterferon alfa-2a in patients with metastatic malignant melanoma. J Clin Oncol. 2006 Mar 1;24(7):1188-94.
- [37] Eggermont AMM, Suciu S, Testori A, Kruit WH, Marsden J, Punt CJ, et al. Ulceration and stage are predictive of interferon efficacy in melanoma: results of the phase III adjuvant trials EORTC 18952 and EORTC 18991. Eur J Cancer 2012;48:218-25.
- [38] Escudier B, Szczylik C, Hutson TE, Demkow T, Staehler M, Rolland F, et al. Randomized phase II trial of first-line treatment with sorafenib versus interferon alfa-2a in patients with metastatic renal cell carcinoma (including Errata). J Clin On 2009;27(8):1280-9.
- [39] Choueiri TK, Hutson TE, Bukowski RM. Evolving role of pegylated interferons in metastatic renal cell carcinoma. Expert Rev Anticancer Ther. 2003 Dec;3(6):823-9.

Protocol/Amendment No.: 029-05

[40] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, et al. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med 2011;364(26):2517-26.

- [41] Yang JC, Hughes M, Kammula U, Royal R, Sherry RM, Topalia SL. Ipilimumab (anti-CTLA4 antibody) causes regression of metastatic renal cell cancer associated with enteritis and hypophysitis. J Immunother 2007;30(8):825-30.
- [42] Ropponen KM, Eskelinen MJ, Lipponen PK, Alhava E, Kosma V-M. Prognostic value of tumour-infiltrating lymphocytes (TILs) in colorectal cancer. J Pathol 1997;182(3):318-24.
- [43] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, et al. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol 2005;23(10):2346-57.
- [44] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, et al. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med 2008;358(25):2698-703.
- [45] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domaincontaining tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A 2001;98(24):13866-71.
- [46] Chapman PB, Hauschild A, Robert C, Larkin JMG, Haanen JBAG, Ribas A, et al. Updated overall survival (OS) results for BRIM-3, a phase III randomized, openlabel, multicenter trial comparing BRAF inhibitor vemurafenib (vem) with dacarbazine (DTIC) in previously untreated patients with BRAFV600E mutated melanoma [Abstract]. J Clin Oncol 2012;30:abstract 8502.
- [47] Flaherty KT, Robert C, Hersey P, Nathan P, Garbe C, Milhem M, et al. Improved survival with MEK inhibition in BRAF-mutated melanoma. N Engl J Med 2012:1-8.
- [48] Hauschild A, Grob JJ, Demidov LV, Jouary T, Gutzmer R, Millward M, et al. Dabrafenib in BRAF-mutated metastatic melanoma: a multicentre, open-label, phase 3 randomised controlled trial. Lancet 2012;380:358-65.
- [49] Hauschild A, Grobb J, Demidov LV, Jouary T, Gutzmer R, Millward M, et al. An update on Overall Survival (OS) and follow-on therapies in BREAK-3, a Phase III, randomized trial: dabrafenib (D) vs. dacarbazine (DTIC) in Patients (pts) with BRAF V600E mutation-positive metastatic melanoma (MM). Poster session presented at: ESMO Annual Meeting; 2014 Sep 29; Madrid.

Protocol/Amendment No.: 029-05

[50] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, et al. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2014 Nov 16. [Epub ahead of print]

- Postow MA, Chesney J, Pavlick AC, Robert C, Grossmann K, McDermott D, et al. [51] Nivolumab and ipilimumab versus ipilimumab in untreated melanoma. N Engl J Med. 2015 May 21;372(21):2006-17.
- [52] Postow M, Chesney J, Pavlick A, Robert C, Grossmann K, McDermott D, et al. Initial report of overall survival rates from a randomized phase II trial evaluating the combination of nivolumab (NIVO) and ipilimumab (IPI) in patients with advanced melanoma (MEL) [abstract]. Abstracts of the 2016 AACR Annual Meeting; 2016 Apr 16-20; New Orleans, LA; AACR; 2016. p. 1.
- [53] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, et al. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34.
- [54] Escudier B, Bellmunt J, Negrier S, Bajetta E, Melichar B, Bracarda S, et al. Phase III trial of bevacizumab plus interferon alfa-2a in patients with metastatic renal cell carcinoma (AVOREN): Final analysis of overall survival. J Clin Oncol 2010;28(13):2144-50.
- [55] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, et al. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81.
- [56] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, et al. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24.
- [57] Sternberg CN, Davis ID, Mardiak J, Szczylik C, Lee E, Wagstaff J, et al. Pazopanib in locally advanced or metastatic renal cell carcinoma: results of a randomized phase III trial. J Clin Oncol. 2010 Feb 20;28(6):1061-8.
- [58] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, et al. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13.
- [59] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, et al. Safety and Tumor Responses with Lambrolizumab (AntiΓÇôPD-1) in Melanoma. N Engl J Med 2013;369(2):134-44.

**Protocol/Amendment No.:** 029-05

[60] Drake CG, McDermott DF, Sznol M, Choueiri TK, Kluger HM; Powderly JD, et al. Survival, safety, and response duration results of nivolumab (Anti-PD-1; BMS-936558; ONO-4538) in a phase I trial in patients with previously treated metastatic renal cell carcinoma (mRCC): Long-term patient follow-up. [Abstract 4514]. 2013 ASCO Annual Meeting, Oral Abstract Session, Poster Discussion Session, Genitourinary (Nonprostate) Cancer; 2013.

- [61] Cho DC, Sosman JA, Sznol M, Gordon MS, Hollebecque A, Hamid O, et al. Clinical activity, safety, and biomarkers of MPDL3280A, an engineered PD-L1 antibody in patients with metastatic renal cell carcinoma (mRCC). [Abstract 4505]. 2013 ASCO Annual Meeting, Oral Abstract Session, Genitourinary (Nonprostate) Cancer; 2013.
- [62] Kirkwood JM, Ernstoff MS. Interferons in the treatment of human cancer. J Clin Oncol 1984;2(4):336-52.
- [63] Legha SS, Ring S, Eton O, Bedikian A, Buzaid AC, Plager C, et al. Development of a biochemotherapy regimen with concurrent administration of cisplatin, vinblastine, dacarbazine, interferon alfa, and interleukin-2 for patients with metastatic melanoma. J Clin Oncol 1998;16:1752-9.
- [64] Atkins MB, Hsu J, Lee S, Cohen GI, Flaherty LE, Sosma JA, et al. Phase III trial comparing concurrent biochemotherapy with cisplatin, vinblastine, dacarbazine, interleukin-2, and interferon alfa-2b with cisplatin, vinblastine, and dacarbazine alone in patients with metastatic malignant melanoma (E3695): A trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol 2008;26(35):5748-54.
- [65] Terawaki S, Chikuma S, Shibayama S, Hayashi T, Yoshida T, Okazaki T, et al. IFN-a directly promotes programmed cell death-1 transcription and limits the duration of T cell-mediated immunity. J Immunol 2011;186:2772-9.
- [66] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, et al. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med 2010;363(8):711-23.
- [67] Selby M, Engelhardt J, Lu LS, Quigley M, Wang C, Chen B, et al. Antitumor activity of concurrent blockade of immune checkpoint molecules CTLA-4 and PD-1 in preclinical models. [Abstract 3061]. 2013 ASCO Annual Meeting, General Poster Session, Developmental Theraputics Immunotherapy; 2013 May 31 Jun 3. Chicago, IL, 2013.
- [68] Sznol M, Callahan MK, Kluger H, Postow MA, Burke M, Hong Q, et al. Combined nivolumab (anti-PD-1, BMS-936558, ONO-4538) and ipilimumab in the treatment of advanced melanoma patients: Safety and clinical activity. [Abstract 3734]. European Society for Medical Onocology 2013 Annual Meeting; 2013 Sep 27-Oct 1; Amsterdam, Netherlands, 2013.

**Protocol/Amendment No.:** 029-05

[69] Topalian SL, Sznol M, Brahmer JR, McDermott DF, Smith DC, Gettinger SN, et al. Nivolumab (anti-PD-1; BMS-936558; ONO-4538) in patients with advanced solid tumors: Survival and longterm safety in a phase I trial [Abstract 3002]. 2013 ASCO Annual Meeting; 2013 May 31 - Jun 4. Chicago, IL, 2013.

- [70] Bukowski R, Ernstoff MS, Gore ME, Nemunaitis JJ, Amato A, Gupta SK, et al. Pegylated interferon alfa-2b treatment for patients with solid tumors: A phase I/II study. J Clin Oncol 2002;20(18):3841-49.
- [71] Talpaz M, O'Brien S, Rose E, Gupta S, Shan J, Cortes J, et al. Phase 1 study of polyethylene glycol formulation of interferon alpha-2B (Schering 54031) in Philadelphia chromosome-positive chronic myelogenous leukemia. Blood. 2001 Sep 15;98(6):1708-13.
- Tannir NM, Cohen L, Wang X, Thall P, Mathew PF, Jonasch E, et al. Improved [72] tolerability and quality of life with maintained efficacy using twice-daily low-dose interferon-a-2b. Cancer 2006;107:2254-61.
- [73] George S, Hutson TE, Mekhail T, Wood L, Finke J, Elson P, et al. Phase I trial of PEG-interferon and recombinant IL-2 in patients with metastatic renal cell carcinoma. Cancer Chemother Pharmacol 2008;62:347-54.
- [74] Kudchadkar RR, Gibney GT, Weber J, Chen A, Smith K, Merek S, et al. A phase IB study of ipilimumab with peginterferon alfa-2b in patients with unresectable melanoma. [Abstract 9079]. 2013 ASCO Annual Meeting, Oral Abstract Session, General Poster Session, Melanoma/Skin Cancers; 2013.
- [75] Lyrdal D, Stienrner U, Lundstam S. Metastatic renal cell carcinoma treated with peg-interferon alfa-2b. Acta Oncol 2009;48:901-8.
- [76] Escudier B, Pluzanska A, Koralewski P, Ravaud A, Bracarda S, Szczylik C, et al. Bevacizumab plus interferon alfa-2a for treatment of metastatic renal cell carcinoma: a randomised, double-blind phase III trial. Lancet 2007;370:2103-11.
- [77] Rini BI, Halabi S, Rosenberg JE, Stadler WM, Vaena DA, Ou SS, et al. Bevacizumab plus interferon alfa compared with interferon alfa monotherapy in patients with metastatic renal cell carcinoma: CALGB 90206. J Clin Oncol. 2008 Nov 20;26(33):5422-8.
- [78] Melichar B, Bracarda S, Matveev V, Alekseev B, Ivanov S, Zyryanov A, et al. A multinational phase II trial of bevacizumab with low-dose interferon-α2a as firstline treatment of metastatic renal cell carcinoma: BEVLiN. Ann Oncol. "in press" 2013.

Protocol/Amendment No.: 029-05

[79] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med 2013;369:122-33.

- [80] Hodi FS, Chesney J, Pavlick AC, Robert C, Grossmann KF, McDermott DF, et al. Combined nivolumab and ipilimumab versus ipilimumab alone in patients with advanced melanoma: 2-year overall survival outcomes in a multicentre, randomised, controlled, phase 2 trial. Lancet Oncol. 2016 Nov;17(11):1558-1568.
- [81] Agrawal S, Feng Y, Roy A, Kollia G, Lestini B. Nivolumab dose selection: challenges, opportunities and lessons learned for cancer immunotherapy. J Immunother Cancer. 2015 Nov 4;3(2): P141.
- [82] Feng Y, Masson E, Dai D, Parker SM, Berman D, Roy A. Model-based clinical pharmacology profiling of ipilimumab in patients with advanced melanoma. Br J Clin Pharmacol. 2014 Jul;78(1):106-17.
- [83] Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body sizebased dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009;49:1012-1024.
- [84] Ji Y, Liu P, Li Y, Bekele BN. A modified toxicity probability interval method for dose-finding trials. Clin Trials 2010;7:653-63.
- [85] Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med 1985;4:213-26.

Protocol/Amendment No.: 029-05

#### 12.0 APPENDICES

#### 12.1 Merck Code of Conduct for Clinical Trials

#### Merck\* **Code of Conduct for Clinical Trials**

#### I. Introduction

#### A. Purpose

Merck, through its subsidiaries, conducts clinical trials worldwide to evaluate the safety and effectiveness of our products. As such, we are committed to designing, implementing, conducting, analyzing and reporting these trials in compliance with the highest ethical and scientific standards. Protection of subject safety is the overriding concern in the design of clinical trials. In all cases, Merck clinical trials will be conducted in compliance with local and/or national regulations and in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

Such standards shall be endorsed for all clinical interventional investigations sponsored by Merck irrespective of the party (parties) employed for their execution (e.g., contract research organizations, collaborative research efforts). This Code is not intended to apply to trials which are observational in nature, or which are retrospective. Further, this Code does not apply to investigator-initiated trials which are not under the control of Merck.

#### II. Scientific Issues

#### A. Trial Conduct

#### Trial Design

Except for pilot or estimation trials, clinical trial protocols will be hypothesis-driven to assess safety, efficacy and/or pharmacokinetic or pharmacodynamic indices of Merck or comparator products. Alternatively, Merck may conduct outcomes research trials, trials to assess or validate various endpoint measures, or trials to determine subject preferences, etc.

The design (i.e., subject population, duration, statistical power) must be adequate to address the specific purpose of the trial. Research subjects must meet protocol entry criteria to be enrolled in the trial.

Merck selects investigative sites based on medical expertise, access to appropriate subjects, adequacy of facilities and staff, previous performance in Merck trials, as well as budgetary considerations. Prior to trial initiation, sites are evaluated by Merck personnel to assess the ability to successfully conduct the trial.

### 3. Site Monitoring/Scientific Integrity

Trial sites are monitored to assess compliance with the trial protocol and general principles of Good Clinical Practice. Merck reviews clinical data for accuracy, completeness and consistency. Data are verified versus source documentation according to standard operating procedures. Per Merck policies and procedures, if fraud, misconduct or serious GCP-non-Compliance are suspected, the issues are promptly investigated. When necessary, the clinical site will be closed, the responsible regulatory authorities and ethics review committees notified and data disclosed accordingly.

#### B. Publication and Authorship

To the extent scientifically appropriate, Merck seeks to publish the results of trials it conducts. Some early phase or pilot trials are intended to be hypothesis-generating rather than hypothesis testing. In such cases, publication of results may not be appropriate since the trial may be underpowered and the analyses complicated by statistical issues of multiplicity.

Merck's policy on authorship is consistent with the requirements outlined in the ICH-Good Clinical Practice guidelines. In summary, authorship should reflect significant contribution to the design and conduct of the trial, performance or interpretation of the analysis, and/or writing of the manuscript. All named authors must be able to defend the trial results and conclusions. Merck funding of a trial will be acknowledged in publications.

7-Nov-2017 Confidential 04SGNN

07W8HB

**Protocol/Amendment No.:** 029-05

#### **III. Subject Protection**

#### A. IRB/ERC review

All clinical trials will be reviewed and approved by an independent IRB/ERC before being initiated at each site. Significant changes or revisions to the protocol will be approved by the IRB/ERC prior to implementation, except that changes required urgently to protect subject safety and well-being may be enacted in anticipation of IRB/ERC approval. For each site, the IRB/ERC and Merck will approve the subject informed consent form.

#### B. Safety

The guiding principle in decision-making in clinical trials is that subject welfare is of primary importance. Potential subjects will be informed of the risks and benefits of, as well as alternatives to, trial participation. At a minimum, trial designs will take into account the local standard of care. Subjects are never denied access to appropriate medical care based on participation in a Merck clinical trial.

All participation in Merck clinical trials is voluntary. Subjects are enrolled only after providing informed consent for participation. Subjects may withdraw from a Merck trial at any time, without any influence on their access to, or receipt of, medical care that may otherwise be available to them.

#### C. Confidentiality

Merck is committed to safeguarding subject confidentiality, to the greatest extent possible. Unless required by law, only the investigator, sponsor (or representative) and/or regulatory authorities will have access to confidential medical records that might identify the research subject by name.

#### D. Genomic Research

Genomic Research will only be conducted in accordance with informed consent and/or as specifically authorized by an Ethics Committee.

#### IV. Financial Considerations

#### A. Payments to Investigators

Clinical trials are time- and labor-intensive. It is Merck's policy to compensate investigators (or the sponsoring institution) in a fair manner for the work performed in support of Merck trials. Merck does not pay incentives to enroll subjects in its trials. However, when enrollment is particularly challenging, additional payments may be made to compensate for the time spent in extra recruiting efforts.

Merck does not pay for subject referrals. However, Merck may compensate referring physicians for time spent on chart review to identify potentially eligible subjects.

#### **B.** Clinical Research Funding

Informed consent forms will disclose that the trial is sponsored by Merck, and that the investigator or sponsoring institution is being paid or provided a grant for performing the trial. However, the local IRB/ERC may wish to alter the wording of the disclosure statement to be consistent with financial practices at that institution. As noted above, publications resulting from Merck trials will indicate Merck as a source of funding.

#### C. Funding for Travel and Other Requests

Funding of travel by investigators and support staff (e.g., to scientific meetings, investigator meetings, etc.) will be consistent with local guidelines and practices including, in the U.S., those established by the American Medical Association (AMA).

#### V. Investigator Commitment

Investigators will be expected to review Merck's Code of Conduct as an appendix to the trial protocol, and in signing the protocol, agree to support these ethical and scientific standards.

\* In this document, "Merck" refers to Merck Sharp & Dohme Corp. and Schering Corporation, each of which is a subsidiary of Merck & Co., Inc. Merck is known as MSD outside of the United States and Canada. As warranted by context, Merck also includes affiliates and subsidiaries of Merck & Co., Inc."

MK-3475-029-05 Final Protocol
Confidential

**Protocol/Amendment No.:** 029-05

# 12.2 Collection and Management of Specimens for Future Biomedical Research

#### 1. Definitions

a. Biomarker: A biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition. <sup>1</sup>

- b. Pharmacogenomics: The investigation of variations of DNA and RNA characteristics as related to drug/vaccine response.2
- c. Pharmacogenetics: A subset of pharmacogenomics, pharmacogenetics is the influence of variations in DNA sequence on drug/vaccine response.2
- d. DNA: Deoxyribonucleic acid.
- e. RNA: Ribonucleic acid.

# 2. Scope of Future Biomedical Research

The DNA, leftover tumor tissue and leftover blood specimen(s) collected in the current trial will be used to study various causes for how subjects may respond to a drug/vaccine. The DNA, leftover tumor tissue and leftover blood specimen(s) will be stored to provide a resource for future trials conducted by Merck focused on the study of biomarkers responsible for how a drug/vaccine enters and is removed by the body, how a drug/vaccine works, other pathways a drug/vaccine may interact with, or other aspects of disease. The specimen(s) may be used for future assay development and/or drug/vaccine development.

It is now well recognized that information obtained from studying and testing clinical specimens offers unique opportunities to enhance our understanding of how individuals respond to drugs/vaccines, enhance our understanding of human disease and ultimately improve public health through development of novel treatments targeted to populations with the greatest need. All specimens will be used by Merck or designees and research will be monitored and reviewed by a committee of our scientists and clinicians.

# 3. Summary of Procedures for Future Biomedical Research

a. Subjects for Enrollment

All subjects enrolled in the clinical trial will be considered for enrollment in the Future Biomedical Research sub-trial.

#### b. Informed Consent

07W8HB

Informed consent for specimens (i.e., DNA, RNA, protein, etc.) will be obtained during screening for protocol enrollment from all subjects or legal guardians, at a trial visit by the investigator or his or her designate. Informed consent for Future Biomedical Research should be presented to the subjects on Visit 1. If delayed, present consent at next possible Subject Visit. Informed consent must be obtained prior to collection of all Future Biomedical Research specimens. Consent forms signed by the subject will be kept at the clinical trial site under secure storage for regulatory reasons. Information contained on the consent form alone cannot be traced

MK-3475-029-05 Final Protocol
O4SGNN
Confidential
7-Nov-2017

Protocol/Amendment No.: 029-05

to any specimens, test results, or medical information once the specimens have been rendered de-identified.

Subjects are not required to participate in the Future Biomedical Research sub-trial in order to participate in the main trial. Subjects who decline to sign the Future Biomedical Research informed consent will not have the specimen collected nor will they be discontinued from the main trial.

A template of each trial site's approved informed consent will be stored in the Sponsor's clinical document repository. Each consent will be assessed for appropriate specimen permissions.

Each informed consent approved by an ethics committee is assigned a unique tracking number. The tracking number on this document will be used to assign specimen permissions for each specimen into the Entrusted Keyholder's Specimen Database.

# c. eCRF Documentation for Future Biomedical Research Specimens

Documentation of both consent and acquisition of Future Biomedical Research specimens will be captured in the electronic Case Report Forms (eCRFs). Reconciliation of both forms will be performed to assure that only appropriatelyconsented specimens are used for this sub-trial's research purposes. Any specimens for which such an informed consent cannot be verified will be destroyed.

# d. Future Biomedical Research Specimen Collections

Blood specimens for DNA or RNA isolation will usually be obtained at a time when the subject is having blood drawn for other trial purposes. Specimens like tissue and bone marrow will usually be obtained at a time when the subject is having such a procedure for clinical purposes.

Specimens will be collected and sent to the laboratory designated for the trial where they will be processed (e.g., DNA or RNA extraction, etc) following the Merck approved policies and procedures for specimen handling and preparation.

If specimens are collected for a specific genotype or expression analysis as an objective to the main trial, this analysis is detailed in the main body of this protocol (Section 8.0 - Statistical Analysis Plan). These specimens will be processed. analyzed, and the remainder of the specimen will be destroyed. The results of these analyses will be reported along with the other trial results. A separate specimen will be obtained from properly-consented subjects in this protocol for storage in the biorepository for Future Biomedical Research.

#### 4. Confidential Subject Information for Future Biomedical Research

In order to optimize the research that can be conducted with Future Biomedical Research specimens, it is critical to link subject' clinical information with future test results. In fact little or no research can be conducted without connecting the clinical trial data to the specimen. The clinical data allow specific analyses to be conducted. Knowing subject characteristics like gender, age, medical history and treatment outcomes are critical to understanding clinical context of analytical results.

Confidential 04SGNN

07W8HB

**Protocol/Amendment No.:** 029-05

To maintain privacy of information collected from specimens obtained for Future Biomedical Research, Merck has developed secure policies and procedures. All specimens will be de-identified as described below.

At the clinical trial site, unique codes will be placed on the Future Biomedical Research specimens for transfer to the storage facility. This first code is a random number which does not contain any personally identifying information embedded within it. The link (or key) between subject identifiers and this first unique code will be held at the trial site. No personal identifiers will appear on the specimen tube.

This first code will be replaced with a second code at a Merck designated storage/lab facility. The second code is linked to the first code via a second key. The specimen is now double coded. Specimens with the second code are sometimes referred to as deidentified specimens. The use of the second code provides additional confidentiality and privacy protection for subjects over the use of a single code. Access to both keys would be needed to link any data or specimens back to the subject's identification.

The second code is stored separately from the first code and all associated personal specimen identifiers. A secure link, the second key, will be utilized to match the second code to the first code to allow clinical information collected during the course of the trial to be associated with the specimen. This second key will be transferred under secure procedures by the Merck designated facility to an Entrusted Keyholder at Merck. The second code will be logged into the primary biorepository database at Merck and, in this database, this identifier will not have identifying demographic data or identifying clinical information (i.e., race, sex, age, diagnosis, lab values) associated with it. The specimen will be stored in a designated biorepository site with secure policies and procedures for specimen storage and usage.

The second key can be utilized to reconstruct the link between the results of future biomedical research and the clinical information, at the time of analysis. This linkage would not be possible for the scientist conducting the analysis, but can only be done by the Merck Entrusted Keyholder under strict security policies and procedures. The Merck Entrusted Keyholder will link the information and then issue a de-identified data set for analysis. The only other circumstance by which future biomedical research data would be directly linked to the full clinical data set would be those situations mandated by regulatory authorities (e.g., EMEA, FDA), whereby this information would be directly transferred to the regulatory authority.

#### 5. Biorepository Specimen Usage

07W8HB

Specimens obtained for the Merck Biorepository will be used for analyses using good scientific practices. However, exploratory analyses will not be conducted under the highly validated conditions usually associated with regulatory approval of diagnostics. The scope of research performed on these specimens is limited to the investigation of the variability in biomarkers that may correlate with a clinical phenotype in subjects.

Analyses utilizing the Future Biomedical Research specimens may be performed by Merck, or an additional third party (e.g., a university investigator) designated by Merck. The investigator conducting the analysis will be provided with double coded specimens. Re-association of analysis results with corresponding clinical data will only be conducted

**Protocol/Amendment No.:** 029-05

by the Merck Entrusted Keyholder. Any contracted third party analyses will conform to the specific scope of analysis outlined in this sub-trial. Future Biomedical Research specimens remaining with the third party after the specific analysis is performed will be returned to the sponsor or destroyed and documentation of destruction will be reported to Merck

#### 6. Withdrawal From Future Biomedical Research

Subjects may withdraw their consent for Future Biomedical Research and have their specimens and all derivatives destroyed. Subjects may withdraw consent at any time by contacting the principal investigator for the main trial. If medical records for the main trial are still available, the investigator will contact Merck using the designated mailbox (clinical specimen management@merck.com) and a form will be provided by Merck to obtain appropriate information to complete specimen withdrawal. Subsequently, the subject's specimens will be removed from the biorepository and be destroyed. A letter will be sent from Merck to the investigator confirming the destruction. It is the responsibility of the investigator to inform the subject of completion of destruction. Any analyses in progress at the time of request for destruction or already performed prior to the request being received by the Sponsor will continue to be used as part of the overall research trial data and results. No new analyses would be generated after the request is received.

In the event that the medical records for the main trial are no longer available (e.g., if the investigator is no longer required by regulatory authorities to retain the main trial records) or the specimens have been completely anonymized, there will no longer be a link between the subject's personal information and their specimens. In this situation, the request for specimen destruction can not be processed.

# 7. Retention of Specimens

Future Biomedical Research specimens will be stored in the biorepository for potential analysis for up to 20 years from acquisition. Specimens may be stored for longer if a regulatory or governmental authority has active questions that are being answered. In this special circumstance, specimens will be stored until these questions have been adequately addressed.

Specimens from the trial site will be shipped to a central laboratory and then shipped to the Merck designated biorepository. The specimens will be stored under strict supervision in a limited access facility which operates to assure the integrity of the specimens. Specimens will be destroyed according to Merck policies and procedures and this destruction will be documented in the biorepository database.

#### 8. Data Security

Separate databases for specimen information and for results from the Future Biomedical Research sub-trial will be maintained by Merck. This is done to separate the future exploratory test results (which include genetic data) from the clinical trial database thereby maintaining a separation of subject number and these results. The separate databases are accessible only to the authorized Sponsor and the designated trial administrator research personnel and/or collaborators. Database user authentication is highly secure, and is accomplished using network security policies and practices based in

MK-3475-029-05 Final Protocol 7-Nov-2017

**Protocol/Amendment No.:** 029-05

international standards (e.g., ISO17799) to protect against unauthorized access. The Merck Entrusted Keyholder maintains control over access to all specimen data. These data are collected for future biomedical research purposes only as specified in this subtrial will not be used for any other purpose.

# 9. Reporting of Future Biomedical Research Data to Subjects

There is no definitive requirement in either authoritative ethical guidelines or in relevant laws/regulations globally that research results have to be, in all circumstances, returned to the trial participant. Some guidelines advocate a proactive return of data in certain instances. No information obtained from exploratory laboratory studies will be reported to the subject or family, and this information will not be entered into the clinical database maintained by Merck on subjects. Principle reasons not to inform or return results to the subject include: lack of relevance to subject health, limitations of predictive capability, concerns of misinterpretation and absence of good clinical practice standards in exploratory research typically used for diagnostic testing.

If any exploratory results are definitively associated with clinical significance for subjects while the clinical trial is still ongoing, investigators will be contacted with information as to how to offer clinical diagnostic testing (paid for by Merck) to subjects enrolled and will be advised that counseling should be made available for all who choose to participate in this diagnostic testing.

If any exploratory results are definitively associated with clinical significance after completion of a clinical trial, Merck will publish the results without revealing specific subject information, inform all trial sites who participated in the Merck clinical trial and post anonymized results on our website or other accredited website(s) that allow for public access (e.g., disease societies who have primary interest in the results) in order that physicians and patients may pursue clinical diagnostic testing if they wish to do so.

#### 10. Gender, Ethnicity and Minorities

Although many diagnoses differ in terms of frequency by ethnic population and gender, every effort will be made to recruit all subjects diagnosed and treated on Merck clinical trials for future biomedical research. When trials with specimens are conducted and subjects identified to serve as controls, every effort will be made to group specimens from subjects and controls to represent the ethnic and gender population representative of the disease under current investigation.

#### 11. Risks Versus Benefits of Future Biomedical Research

For future biomedical research, risks to the subject have been minimized. Risks include those associated with venipuncture to obtain the whole blood specimen. This specimen will be obtained at the time of routine blood specimens drawn in the main trial.

Merck has developed strict security, policies and procedures to address subject data privacy concerns. Data privacy risks are largely limited to rare situations involving possible breach of confidentiality. In this highly unlikely situation there is risk that the information, like all medical information, may be misused.

It is necessary for subject-related data (i.e., ethnicity, diagnosis, drug therapy and dosage, age, toxicities, etc.) to be re-associated to double coded specimens at the time of data

MK-3475-029-05 Final Protocol 7-Nov-2017

**Protocol/Amendment No.:** 029-05

analysis. These subject data will be kept in a separate, secure Merck database, and all specimens will be stripped of subject identifiers. No information concerning results obtained from future biomedical research will be entered into clinical records, nor will it be released to outside persons or agencies, in any way that could be tied to an individual subject.

# 12. Self-Reported Ethnicity

Subjects who participate in future biomedical research will be asked to provide selfreported ethnicity. Subjects who do not wish to provide this data may still participate in future biomedical research.

### 13. Questions

Any questions related to the future biomedical research should be e-mailed directly to clinical.specimen.management@merck.com.

#### 14. References

- 1. National Cancer Institute: http://www.cancer.gov/dictionary/?searchTxt=biomarker
- 2. International Conference on Harmonization: DEFINITIONS FOR GENOMIC BIOMARKERS, PHARMACOGENOMICS, PHARMACOGENETICS, GENOMIC DATA AND **SAMPLE** CODING **CATEGORIES** E15; http://www.ich.org/LOB/media/MEDIA3383.pdf
Protocol/Amendment No.: 029-05

12.3 Understanding the Intent, Scope and Public Health Benefits of Exploratory Biomarker Research: A Guide for IRBs/IECs and Investigational Site Staff



Protocol/Amendment No.: 029-05

This informational brochure is intended for IRBs/IECs and Investigational Site Staff. The brochure addresses issues relevant to specimen collection for biomarker research in the context of pharmaceutical drug and vaccine development.

Developed by The Industry Pharmacogenomics Working Group (I-PWG) www.i-pwg.org

#### What is a Biomarker and What is Biomarker Research?

A biomarker is a "characteristic that is objectively measured and evaluated as an indicator of normal biological processes. pathogenic processes, or pharmacologic responses to a therapeutic intervention".

Biomarker research, including research on pharmacogenomic biomarkers, is a tool used to improve the development of pharmaceuticals and understanding of disease. It involves the analysis of biomolecules (such as DNA, RNA, proteins, and lipids), or other measurements (such as blood pressure or brain images) in relation to clinical endpoints of interest. Biomarker research can be influential across all phases of drug development, from drug discovery and preclinical evaluations to clinical development and post-marketing studies. This brochure focuses on biomarker research involving analysis of biomolecules from biological samples collected in clinical trials. Please refer to I-PWG Pharmacogenomic Informational Brochure<sup>2</sup> and ICH Guidance E153 for additional information specific to pharmacogenomic biomarkers.

#### 2. Why is Biomarker Research Important?

#### Importance to Patients and Public Health

Biomarker research is helping to improve our ability to predict, detect, and monitor diseases and improve our understanding of how individuals respond to drugs. This research underlies personalized medicine: a tailored approach to patient treatment based on the molecular analysis of genes, proteins, and metabolites.4 The goal of biomarker research is to aid clinical decision-making toward safer and more efficacious courses of treatment. improved patient outcomes, and overall cost-savings. It also allows for the continued development and availability of drugs that are effective in certain sub-populations when they otherwise might not have been developed due to insufficient efficacy in the broader population.

Recent advances in biomedical technology, including genetic and molecular medicine, have greatly increased the power and precision of analytical tools used in health research and have accelerated the drive toward personalized medicine. In some countries, highly focused initiatives have been created to promote biomarker research (e.g., in the US: www.fda.gov/oc/initiatives/criticalpath/; in the EU: www.imi.europa.eu/index\_en.html).

#### Importance to Drug Development

Biomarker research is being used by the pharmaceutical industry to streamline the drug development process. Some biomarkers are used as substitutes or "surrogates" for safety or efficacy endpoints in clinical trials particularly where clinical outcomes or events cannot practically or ethically be measured (e.g., cholesterol as a surrogate for cardiovascular disease).5 By using biomarkers to assess patient response, ineffective drug candidates may be terminated earlier in the development process in favor of more promising drug candidates. Biomarkers are being used to optimize clinical trial designs and outcomes by identifying patient populations that are more likely to respond to a drug therapy or to avoid specific adverse events.

I-PWG

Protocol/Amendment No.: 029-05

Biomarker research is also being used to enhance scientific understanding of the mechanisms of both treatment response and disease processes, which can help to identify future targets for drug development. Depending on the clinical endpoints in a clinical trial, biomarker sample collection may either be a required or optional component of the trial. However, both mandatory and optional sample collections are important for drug development.

## 3. Importance of Biomarkers to Regulatory Authorities

Regulatory health authorities are increasingly aware of the benefits of biomarkers and how they may be used for drug approval, clinical trial design, and clinical care. Biomarkers have been used to establish risk:benefit profiles. For example, the FDA has modified the US warfarin (Coumadin®) label to include the analysis of CYP2C9 and VKORC1 genes to guide dosing regimens. Health authorities such as the FDA (USA), EMEA (European Union), MHLW (Japan), and ICH (International) are playing a key role in advancing this scientific field as it applies to pharmaceutical development by creating the regulatory infrastructure to facilitate this research. Numerous regulatory guidances and concept papers have already been issued, many of which are available through www.i-pwg.org. Global regulatory authorities have highlighted the importance of biomarker research and the need for the pharmaceutical industry to take the lead in this arena. 3, 6-24

## 4. How are Biomarkers Being Used in Drug/Vaccine Development?

Biomarker research is currently being used in drug/vaccine development to:

- · Explain variability in response among participants in clinical trials
- · Better understand the mechanism of action or metabolism of investigational drugs
- · Obtain evidence of pharmacodynamic activity (i.e., how the drug affects the body) at the molecular level
- Address emerging clinical issues such as unexpected adverse events
- Determine eligibility for clinical trials to optimize trial design
- Optimize dosing regimens to minimize adverse reactions and maximize efficacy
- Develop drug-linked diagnostic tests to identify patients who are more likely or less likely to benefit from treatment or who may be at risk of experiencing adverse events
- Provide better understanding of mechanisms of disease
- Monitor clinical trial participant response to medical interventions

Biomarker research, including research on banked samples, should be recognized as an important public health endeavor for the overall benefit of society, whether by means of advancement of medical science or by development of safer and more effective therapies.7 Since the value of collected samples may increase over time as scientific discoveries are made, investment in long-term sample repositories is a key component of biomarker research.



Protocol/Amendment No.: 029-05

#### Biomarkers are Already a Reality in Health Care

A number of drugs now have biomarker information included in their labels.26 Biomarker tests are already being used in clinical practice to serve various purposes:

Predictive biomarkers (efficacy) - In clinical practice, predictive efficacy biomarkers are used to predict which patients are most likely to respond, or not respond, to a particular drug. Examples include: i) Her2/neu overexpression analysis required for prescribing trastuzumab (Herceptin®) to breast cancer patients, ii) c-kit expression analysis prior to prescribing imatinib mesylate (Gleevec®) to gastrointestinal stromal tumor patients, and iii) KRAS mutational status testing prior to prescribing panitumumab (Vectibix®) or cetuximab (Erbitux®) to metastatic colorectal cancer patients.

Predictive biomarkers (safety) - In clinical practice, predictive safety biomarkers are used to select the proper drug dose or to evaluate the appropriateness of continued therapy in the event of a safety concern. Examples include: i) monitoring of blood potassium levels in patients receiving drospirenone and ethinyl estradiol (Yasmin®) together with daily long-term drug regimens that may increase serum potassium, and ii) prospective HLA-B\*5701 screening to identify those at increased risk for hypersensitivity to abacavir (Ziagen®).

Surrogate biomarkers - In clinical practice, surrogate biomarkers may be used as alternatives to measures such as survival or irreversible morbidity. Surrogate biomarkers are measures that are reasonably likely, based on epidemiologic, therapeutic, pathophysiologic, or other evidence, to predict clinical benefit. Examples include: i) LDL level as a surrogate for risk of cardiovascular diseases in patients taking lipid-lowering agents such as atorvastatin calcium (Lipitor®), ii) blood glucose as a surrogate for clinical outcomes in patients taking anti-diabetic agents, and iii) HIV plasma viral load and CD4 cell counts as sur-

rogates for time-to-clinical-events and overall survival in patients receiving antiretroviral therapy for HIV disease.

Prognostic biomarkers - Biomarkers can also help predict clinical outcomes independent of any treatment modality. Examples of prognostic biomarkers used in clinical practice include: i) CellSearch™ to predict progressionfree survival in breast cancer, ii) anti-CCP (cyclic citrullinated protein) for the severity of rheumatoid arthritis, iii) estrogen receptor status for breast cancer, and iv) antidsDNA for the severity of systemic lupus erythematosus.

#### 6. Biomarker Samples from Clinical Trials: An Invaluable Resource

Adequate sample sizes and high-quality data from controlled clinical trials are key to advancements in biomarker research. Samples collected in clinical trials create the opportunity for investigation of biomarkers related to specific drugs, drug classes, and disease areas. Clinical drug development programs are therefore an invaluable resource and a unique opportunity for highly productive biomarker research. In addition to conducting independent research, pharmaceutical companies are increasingly contributing to consortia efforts by pooling samples, data, and expertise in an effort to conduct rigorous and efficient biomarker research and to maximize the probability of success. 26-27

## Informed Consent for Collection & Banking of Biomarker Samples

Collection of biological samples in clinical trials must be undertaken with voluntary informed consent of the participant (or legally-acceptable representative). Policies

1-PWG

3

Protocol/Amendment No.: 029-05

and regulations for legally-appropriate informed consent vary on national, state, and local levels, but are generally based on internationally recognized pillars of ethical conduct for research on human subjects.28-31

Optional vs. Required Subject Participation Depending on the relevance of biomarker research to a clinical development program at the time of protocol development, the biomarker research may be a core required component of a trial (e.g., key to elucidating the drug mechanism of action or confirming that the drug is interacting with the target) or may be optional (e.g., to gain valuable knowledge that enhances the understanding of diseases and drugs). Informed consent for the collection of biomarker samples may be presented either in the main clinical informed consent form or as a separate informed consent form, with approaches varying somewhat across pharmaceutical companies. The relevance of biomarker research to a clinical development program may change over time as the science evolves. The samples may therefore increase in value after a protocol is developed.

Consent for Future Research Use While it can be a challenge to specify the details of the research that will be conducted in the future, the I-PWG holds the view that future use of samples collected for exploratory biomarker research in clinical trials should be permissible when i) the research is scientifically sound, ii) participants are informed of the scope of the intended future research, even if this is broadly defined (see potential uses in Section 4 above), iii) autonomy is respected by providing the option to consent separately to future use of samples or by providing the option to terminate further use of samples upon request (consent withdrawal / sample destruction), and iv) industry standards for confidentiality protection per Good Clinical Practice guidelines are met.3, 31 Importantly, any research using banked samples should be consistent with the original informed consent, except where otherwise permitted by local law or regulation.

Important elements of informed consent for future use of samples include, but are not limited to:39

The scope of research - Where the scope of the potential future research is broad, participants should be informed of the boundaries of the research. While it may not be possible to describe the exact analytical techniques that will be used, or specific molecules that will be analyzed, it is possible to clearly articulate in reasonable detail the type of research to be conducted and its purpose. Information regarding whether stored samples may be shared with other parties or utilized for commercialization purposes should also be addressed.

Withdrawal of consent / sample destruction - The informed consent form should inform participants of their right to withdraw their consent / request destruction of their samples. This should include the mechanisms for exercising that right and any limitations to exercising that right. For example, participants should be informed that it is not possible to destroy samples that have been anonymized.3 In addition, according to industry standards and regulatory guidance, participants should be informed that data already generated prior to a consent withdrawal request are to be maintained as part of the study data.36

The duration of storage - The permissible duration of storage may vary according to the nature and uses of the samples and may also vary on national, state, and local levels. The intended duration of storage, including indefinite storage, should be specified.

I-PWG



Protocol/Amendment No.: 029-05

#### 8. Biomarker Sample Collection in Different Countries

Collection of biological samples for biomarker research is straightforward in most jurisdictions. Some countries have specific laws and regulations regarding collection, labeling, storage, export, and/or use of exploratory samples. In addition, some regulations distinguish between DNA and non-DNA samples or between samples used for diagnostic purposes and samples collected for scientific research. Processes for the collection, labeling, storage. export, and/or use of biomarker samples should always adhere to the laws and regulations of the country/region in which those samples are collected.

#### 9. Return of Research Results to Study **Participants**

Policies for the return of biomarker research results to study participants who request them vary among pharmaceutical companies. There are many considerations that pharmaceutical companies weigh when determining their policy regarding the return of biomarker research results to study participants. These include:

- i) the conditions under which biomarker research results were generated (i.e., exploratory research laboratory versus accredited diagnostic laboratory)
- ii) whether the results will have an impact on the medical care of the participant or on a related person, if applicable
- iii) whether genetic counseling is recommended (for genetic results)
- iv) the ability to accurately link the result to the individual from whom the sample was collected
- v) international, national, and local guidelines, policies, legislation, and regulations regarding participants' rights to access data generated on them

Renegar et al. 2006 and Article 29 Data Protection Working Party (an advisory committee to the European Commission on the European Data Protection Directive) have addressed these considerations in detail in relation to pharmacogenomic research data and provided a list of documents addressing the general issue of return of research results. 34-36

#### Benefits and Risks Associated with Biomarker Research

#### **Benefits**

While it may not always directly benefit the study participant who is providing the samples, biomarker research can improve overall understanding of disease and treatment of future patients receiving therapies developed from such research. Patients are now benefiting from retrospective biomarker research conducted on samples collected from clinical trials and stored for exploratory research. One example is the recent label update to the EGFR antibody drugs cetuximab (Erbitux®) and panitumumab (Vectibix®) which highlights the value of KRAS status as a predictive biomarker for treatment of metastatic colorectal cancer with this class of drug.

The humanitarian benefit of human research is recognized by the Nuremberg Code. 28,33 Provided that the degree of risk does not exceed that determined by the humanitarian importance of the problem to be solved, research participants should not be denied the right to contribute to the greater common good.28,32

Risks associated with biomarker research are primarily related to the physical aspects of obtaining the sample and to patient privacy concerns.

Physical risks associated with biomarker sample collection in clinical trials can be characterized in two ways: i) negligible additional risk when the biomarker sample is collected as part of a procedure conducted to support

-PWG

Protocol/Amendment No.: 029-05

other core trial objectives, and ii) some added risk where the sampling procedure would otherwise have not been performed as a core component of a trial. Risks are also determined by the invasiveness of the sample collection

Privacy risks are generally those associated with the inappropriate disclosure and misuse of data. Pharmaceutical companies have policies and procedures for confidentiality protection to minimize this risk for all data collected and generated in clinical trials. These may vary across companies, but are based on industry standards of confidentiality and privacy protection highlighted in the following section. Importantly, privacy risks inherent to biomarker data are no greater than other data collected in a clinical trial.

### 11. Privacy, Confidentiality, and Patient Rights

Maintaining the privacy of study participants and the confidentiality of information relating to them is of paramount concern to industry researchers, regulators, and patients. Good Clinical Practice (GCP), the standard adhered to in pharmaceutical clinical research, is a standard that

"... provides assurance that the data and reported results are credible and accurate, and that the rights, integrity, and confidentiality of trial subjects are protected",

where confidentiality is defined as, "The prevention of disclosure, to other than authorized individuals, of a sponsor's proprietary information or of a subject's identity."

This standard dictates that "the confidentiality of records that could identify subjects should be protected, respecting the privacy and confidentiality rules in accordance with applicable regulatory requirements."

Exploratory biomarker research in pharmaceutical development is commonly conducted in research laboratories that are not accredited to perform diagnostic tests used for healthcare decision-making. Therefore, results from exploratory biomarker research usually are not appropriate for use in making decisions about a trial participant's health. In addition, exploratory research data should not be included as part of a participant's medical record accessible for use by insurance companies. Legislation and policies to protect individuals against discrimination based on genetic information continually evolve based on social, ethical, and legal considerations. Examples of such legislation include the Human Tissue Act 2004 (UK) and the Genetic Information Nondiscrimination Act (GINA) 2008 (USA).36-3

#### 12. Where to Get More Information?

Educational resources related to biomarker and pharmacogenomic research that caters to health care professionals, IRBs/IECs, scientists, and patients are continually being created and are publicly available. Links to many of these resources are available through the I-PWG website: www.i-pwg.org.

#### 13. What is I-PWG?

The Industry Pharmacogenomics Working Group (I-PWG) (formerly the Pharmacogenetics Working Group) is a voluntary association of pharmaceutical companies engaged in pharmacogenomic research. The Group's activities focus on non-competitive educational, informational, ethical, legal, and regulatory topics. The Group provides information and expert opinions on these topics and sponsors educational/ informational programs to promote better understanding of pharmacogenomic and other biomarker research for key stakeholders. The I-PWG interacts with regulatory author-

I-PWG

Protocol/Amendment No.: 029-05

ities and policy groups to ensure alignment. More information about the I-PWG is available at: www.i-pwg.org.

#### 14. Contributing authors

Monique A. Franc, Teresa Hesley, Feng Hong, Ronenn Roubenoff, Jasjit Sarang, Andrea Tyukody Renninger, Amelia Warner

#### 15. References

- Atkinson AJ, Colbum WA, DeGruttola VG, et al. Blomarkers and surrogate enopoints: Preferred definitions and conceptual framework. Clinical Pharmacology & Therapeutics 2001; 69(3): 89-95. (Accessed at: www.ncbt.nim.nih.gov/pubmed/11240971)
- I PWG Pharmacogenomics Informational Brochure, 2008. (Accessed at: http://www.l-pwg.org/cms/index.php?option=com\_docman&task=doc\_domioad&gid=77&itemid=118)
- ICH E15 Definitions for Genomic Biomarkers, Pharmacogenomics, Pharmacogenetics, Genomic Data and Sample Coding Categories. April 2008. (Accessed at: www.fda.gov/OHRMs/DOCKETS/98ft/FDA-2008-D-0199-gdl.pdf and at: http://www.lch.org/LOB/media/MEDIA3383.pdf)
- Davis JC, Furstenthal L, Desal AA, et al. The microeconomics of personalized medicine: today's challenge and tomorrow's promise. Nature Reviews Drug Discovery, 2009; 8: 279. (Accessed at:http: www.nature.com/nrd/ournal/v8/hd/abs/hrd/2825.html)
- Bems B, Démolis P, Scheufen ME. How can blomarkers become surrogate endpoints? European Journal of Canoer Supplements 2007; S: 37-40.
   Accessed at: www.journals.elsevlerhealth.com/periodicals/ejcsup/issues/ contents/rissue\_kev=S1359-6349%2907%29079031-4)
- Lesko LJ, Woodcock J. Translation of pharmacogenomics and pharmacogenetics: a regulatory perspective. Nature Reviews Drug Discovery, 2004; 3: 763-769. (Accessed al: www.nature.com/ind/journal/v3/in5/abs/ind/1499.html)
- Lesko LJ, Woodcock J. Pharmacogenomic-guided drug development: regulatory perspective. The Pharmacogenomics Journal, 2002; 2: 20-24. (Accessed at www.ncbi.nim.nih.gov/pubmed/11990376)
- Petricoin EF, Hackett JL, Lesko LJ, et al. Medical applications of microarray technologies: a regulatory science perspective. Nat Genet., 2002; 32: 474-479.

(Accessed at: www.nature.com/ng/journal/v32/n4s/abs/ng1029.html)

- Lesko LJ, Salemo RA, Spear BB, et al. Pharmacogenetics and pharmacogenomics in drug development and regulatory decision making: report of the first FDA-PWG-PhRMA-DruSafe Workshop. J Clin Pharmacol., 2003; 43: 342-358. (Accessed at: http://jop.sagepub.com/og/content/abstract/43/4/342)
- Salemo RA, Lesko LJ. Pharmacogenomics in Drug Development and Regulatory Decision-making: the Genomic Data Submission (GDS) Proposal. Pharmacogenomics, 2004; 5: 28-30. (Accessed at: www.futuremedicine.com/doi/pdf/10/2217/14622416.5.1.25)
- Frueh PW, Goodsald F, Rudman A, et al. The need for education in pharmacogenomics: a regulatory perspective. The Pharmacogenomics Journal, 2005; 5: 218-220. (Accessed at: www.nature.com/tpi/journal/v5/n4/ abs/i550316a.html)
- Genomic Biomarkers Related to Drug Response: Context, Structure and Format of Qualification Submissions. ICH E16 Step 3 draft. (Accessed at: www.emea.europa.europtis.human/ich/38063609endraft.pdf)
- Guiding principles Processing Joint FDA EMEA Voluntary Genomic Data Submissions (VGDSs) within the framework of the Confidentiality Arrangement. May 19, 2006. (Accessed at:
- www.file.gov/forwebself/Drugs/folence/Research/Research/Vessa/Pharmacogeretics/cor065578.pdf)
  14. Guldanoe for Industry Pharmacogenomic Data Submissions. FDA. March 2005. (Accessed at:
- www.tls.govstoverbeathCingstCuttineoComplianceRegulator/informationCuttineosAccre77648.pdf)

  5. Pharmacogenomic Data Submissions Companion Guldanoe. FDA Draft Guldanoe. August 2007. (Accessed at:
- www.ta.gov/conseads/Drugs/Outbroot/conprisons/Regulatory/reformation/Outbrooss/ucm078665.pdf)
  16. Reflection Paper on Pharmacogenomics in Oncology. EMEA 2008.

  (Accessor)

www.emea.europa.eu/pdfs/human/pharmacogenetics/12843505endraft.pdf)

- Position paper on Terminology in Pharmacogenetics. EMEA. 2002. (Accessed at: www.emea.europa.eu/pdfs/human/press/pp/307001en.pdf)
- Concept paper on the development of a Guideline on the use of pharmacogenomic methodologies in the pharmacokinetic evaluation of medicinal products. EMEA. 2009. (Accessed at:

www.emea.europa.eu/pdfs/human/pharmacogenetics/6327009en.pdf)

 Reflection paper on Pharmacogenomic samples, testing and data handling. EMEA. 2007. (Accessed at:

www.emea.europa.eu/pdfs/human/pharmacogenetics/20191406en.pdf)

- Ishiguro A, Toyoshima S, Uyama Y. Current Japanese regulatory situations of pharmacogenomics in drug administration. Expert Review of Clinical Pharmacology, 2008;1: 505-514. (Accessed at: www.ingentaconnect.com/ content/tid/ecp/2008/00000001/00000004/art00007)
- 21. Amur S, Frueh FW, Lesko LJ, et al. Integration and use of

I-PWG

8

Protocol/Amendment No.: 029-05

blomarkers in drug development, regulation and clinical practice: A US regulatory practice. Biomarkers Med. 2008; 2, 305-311. (Accessed at: www.ingentaconnect.com/content/fm/bmm/2008/00000002/00000003/ art00010?crawler-true)

22. Mendrick DL, Brazell C, Mansfield EA, et al. Pharmacogenomics and regulatory decision making: an international perspective. The Pharmacogenomics Journal, 2006; 6(3), 154-157. (Accessed at:

www.nature.com/tp)/journal/v6/n3/abs/6500364a.html)

23. Pendergast MK. Regulatory agency consideration of pharmacogenomics. Exp Biol Med (Maywood), 2008; 233:1498-503. (Accessed at: www.ebmonline.org/ogl/content/abstract/233/12/1496)

24. Goodsald F, Frueh F. Process map proposal for the validation of genomic biomarkers. Pharmacogenomics., 2006; 7(5):773-82 (Accessed at: www.futuremedicine.com/dol/abs/10.2217/14622416.7.5.773)

25. FDA Table of Valid Genomic Biomarkers in the Context of Approved Drug Labels. (Accessed at:

www.fda.gov/Drugs/ScienceResearch/ResearchAreas/Pharmacogenetics/ ucmD83378.htm)

26. International Serious Adverse Event Consortium. (Accessed at: www.saeconsortlum.org)

27. Predictive Safety Testing Consortium. (Accessed www.o-path.org/pstc.cfm)

28. Nuremberg code. (Accessed at:

http://ohsr.od.nlh.gov/guldellnes/nuremberg.html)

29. Declaration of Heisinki. (Accessed at: http://ohsr.od.nih.gov/guldelines/heisinki.html)

30. Belmont report. (Accessed at: http://ohsr.od.nth.gov/guldelines/belmont.html) 31. ICH E5(R1) - Guideline for Good Clinical Practice. June 1995. (Accessed at:

www.lch.org/LOB/media/MEDIA482.pdf)

32. Barnes M, Heffernan K. The "Future Uses" Dilemma: Secondary Uses of Data and Materials by Researchers for Commercial Research Sponsors. Medical Research Law & Policy, 2004; 3: 440-450.

33. Eriksson S, Helgesson G. Potential harms, anonymization, and the right to withdraw consent to blobank research. Eur J Hum Genet., 2005; 13:1071-1076. (Accessed at: www.nature.com/ejhg/journal/v13/n9/pdf/5201458a.pdf)

34. Renegar G, Webster CJ, Stuerzebecher S, et al. Returning genetic research results to individuals: points-to-consider, Bioethics 2006; 20: 24-36. (Accessed at: http://www3.interscience.wiley.com/ogi-bin/fulltext/118562753/PDFSTART)

35. Article 29 Data Protection Working Party. (Accessed at: www.ec.europa.eu/justice\_home/fsj/privacy/workinggroup/index\_en.htm)

36. Human Tissue Act 2004 (UK). (Accessed at:

www.opsl.gov.uk/acts/acts2004/en/ukpgaen\_20040030\_en\_1) 37. Genetic Information Nondiscrimination Act. (Accessed at:

http:///webgate.access.goo.gov/cgi-kin/gebloc.og/?dbname=110\_cong\_public\_lewat-locid=fpubl/253.110.pdf) 38. Guidance for Sponsors, Clinical Investigators, and IRBs Data Retention When Subjects Withdraw from FDA-Regulated Clinical Trials. FDA October 2008. www.fda.gov/OHRMS/DOCKETS/98ft/FDA-2008-D-0576-gdl.pdf

39. Anderson C. Gomez-Mandilla B. Spear BB, Barnes DM, Cheeseman K, Shaw P, Friedman J, McCarthy A, Brazell C, Ray SC, McHale D, Hashimoto L, Sanobrink R, Watson ML, Salerno RA, on behalf of The Pharmacogenetics Working Group. Elements of Informed Consent for Pharmacogenetic Research; Perspective of the Pharmacogenetics Working Group, Pharmacogenomics Journal 2002;2:284-92, (Accessed at: www.nature.com/tpl/journal/v2/n5/abs/6500131a.html)





Protocol/Amendment No.: 029-05

## 12.4 ECOG Performance Status

| GRADE | ECOG PERFORMANCE STATUS |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care; confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled; cannot carry on any self-care; totally confined to bed or chair |
| 5 | Dead |

<sup>\*</sup>Oken M, Creech R, Tormey D, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. *Am J Clin Oncol*. 1982;5:649-655

**Protocol/Amendment No.:** 029-05

# 12.5 Common Terminology Criteria for Adverse Events V4.0 (CTCAE)

The descriptions and grading scales found in the revised NCI CTCAE Version 4.0 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html)

**Protocol/Amendment No.:** 029-05

# 12.6 Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

RECIST 1.1\* will be used in this study for assessment of tumor response. While either CT or MRI may be utilized, as per RECIST 1.1, CT is the preferred imaging technique in this study.

\* As published in the European Journal of Cancer [1]

04SGNN

**Protocol/Amendment No.:** 029-05

# 12.7 List of Abbreviations

| Abbreviation/Term | Definition |
|---|---|
| ACAR | Aggregate Clinical Activity Rate |
| AE | Adverse event |
| ADA | Anti-Drug Antibodies |
| ADCC | Antibody-Dependent Cell-Mediated Cytotoxicity |
| ALT | Alanine aminotransferase |
| ANC | Absolute neutrophil count |
| APC | Antigen Presenting Cells |
| APaT | All-Patients-as-Treated |
| aPTT | Activated partial thromboplastin time |
| AUC | Area Under Curve |
| AST | Aspartate aminotransferase |
| β-hCG | Beta human chorionic gonadotropin |
| BORR | Best objective response rate |
| CBC | Complete blood count |
| CI | Confidence interval |
| CNS | Central nervous system |
| CR | Complete response |
| CrCl | Calculated creatinine clearance |
| CRF | Case report form |
| CSR | Clinical study report |
| CT | Computed tomography |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| ctDNA | Circulating tumor DNA |
| CTL | Cytotoxic T Lymphocytes |
| CTLA-4 | Cytotoxic T-lymphocyte-associated antigen-4 |
| DL | Dose Level |
| DLT | Dose Limiting Toxicity |
| DNA | Deoxyribonucleic acid |
| DOR | Duration of Response |
| DRAE | Drug-related Adverse Event |
| ECI | Events of clinical interest |
| ECI-ie | Events of clinical interest with a potential immunologic etiology |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EMA | European Medicines Agency |
| ERC | Ethics review committee |

04SGNN

| Abbreviation/Term | Definition |
|-------------------|------------------------------------------------|
| FAS | Full analysis set |
| FBR | Future Biomedical Research |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Amendments Act |
| FDAMA | Food and Drug Administration Modernization Act |
| FLC | Free Light Chain |
| FT4 | Free T4 |
| GCP | Good Clinical Practice |
| Hb | Hemoglobin |
| HBV | Hepatitis B |
| HCV | Hepatitis C |
| HIV | Human immunodeficiency virus |
| HR | Hazard ratio |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| ICH | International Conference on Harmonization |
| IgG | Immunoglobulin G |
| IHC | Immunohistochemistry |
| IMiD | Immunomodulatory |
| INR | International normalized ratio |
| IPI | Ipilimumab |
| irAEs | Immune-related adverse events |
| IRB | Institutional Review Board |
| ISS | International Staging System |
| ITSM | Immunoreceptor Tyrosine-based Switch Motif |
| ITT | Intent-To-Treat |
| IV | Intravenous |
| Kg | Kilogram |
| LDH | Lactate dehydrogenase |
| LMWH | Low molecular weight heparin |
| mAb | Monoclonal antibody |
| MAD | Maximum administered dose |
| MC38 | Mouse Colorectal Model 38 |
| mcL | Millimeters |
| MEL | Melanoma |
| MG | Milligram |
| mg/kg | Milligram per kilogram |
| mL | Milliliter |
| Mg | Microgram |
| μg/kg | Microgram per kilogram |

| Abbreviation/Term | Definition |
|---|---|
| MRI | Magnetic resonance imaging |
| MPR | Moderate Partial Response |
| MSD | Merck Sharp & Dohme Corp., a subsidiary of Merck & Co., Inc. |
| MTD | Maximum tolerated dose |
| mRNA | Messenger Ribonucleic acid |
| mTOR | Mammalian target of rapamycin |
| NA or N/A | Not Applicable |
| NCCN | National Comprehensive Cancer Network |
| NCI | National Cancer Institute |
| NK | Natural Killer |
| NSAID | Non-steroidal anti-inflammatory drug |
| NSCLC | Non-small cell lung cancer |
| ORR | Objective I response rate |
| OS | Overall survival |
| OTC | Over-the-counter |
| PBMC | Peripheral blood mononuclear cells |
| PBMC | Peripheral blood mononuclear cells |
| PD | Progressive disease |
| PD-1 | Programmed-death receptor-1 |
| PD-L1 | Programmed-death receptor-ligand 1 |
| PD-L2 | Programmed-death receptor-ligand 2 |
| PEG-IFN | Pegylated Interferon Alfa-2b |
| PET | Positron emission tomography |
| PFS | Progression-free survival |
| PGt | Pharmacogenetic |
| PK | Pharmacokinetic |
| PK-PD | Pharmacokinetic-Pharmacodynamic |
| po | orally |
| PR | Partial response |
| PT | Prothrombin time |
| RCC | Renal Cell Carcinoma |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RNA | Ribonucleic acid |
| RP2D | Recommended Phase 2 Dose |
| RR | Response rate |
| q2w | Every 2 weeks |
| q3w | Every 3 weeks |
| q6w | Every 6 weeks |
| q12w | Every 2 weeks |

| Abbreviation/Term | Definition |
|-------------------|-----------------------------------------|
| SAE | Serious adverse events |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| sCR | Stringent Complete Response |
| SFU | Survival follow-up |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SoC | Standard of Care |
| SJS | Stevens-Johnson Syndrome |
| SOP | Standard Operating Procedures |
| SPEP | Serum protein electrophoresis |
| TCR | T cell receptor |
| T1DM | Type 1 Diabetes Mellitus |
| TIL | Tumor-infiltrating lymphocytes |
| TPI | Toxicity Probability Interval |
| TSH | Thyroid stimulating hormone |
| TTP | Time To Progression |
| VEGF | Vascular endothelial growth factor |
| VGPR | Very Good Partial Response |
| ULN | Upper limit of normal |
| US | United States |

**Protocol/Amendment No.:** 029-05

#### 13.0 SIGNATURES

## 13.1 Sponsor's Representative

| TYPED NAME |
|-------------|
| TITLE |
| SIGNATURE |
| DATE SIGNED |

## 13.2 Investigator

I agree to conduct this clinical trial in accordance with the design outlined in this protocol and to abide by all provisions of this protocol (including other manuals and documents referenced from this protocol). I agree to conduct the trial in accordance with generally accepted standards of Good Clinical Practice. I also agree to report all information or data in accordance with the protocol and, in particular, I agree to report any serious adverse events as defined in Section 7.0 – Assessing and Recording Adverse Events. I also agree to handle all clinical supplies provided by the Sponsor and collect and handle all clinical specimens in accordance with the protocol. I understand that information that identifies me will be used and disclosed as described in the protocol, and that such information may be transferred to countries that do not have laws protecting such information. Since the information in this protocol and the referenced Investigator's Brochure is confidential, I understand that its disclosure to any third parties, other than those involved in approval, supervision, or conduct of the trial is prohibited. I will ensure that the necessary precautions are taken to protect such information from loss, inadvertent disclosure or access by third parties.

| TYPED NAME |
|-------------|
| TITLE |
| SIGNATURE |
| DATE SIGNED |

04SGNN